# PRS COVER PAGE for PROTOCOL

**TITLE**: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of VT-1161 Oral Capsules in the Treatment of Subjects with Recurrent Vulvovaginal Candidiasis (VMT-VT-1161-CL-012)

DATE: 01 October 2019

**CLINICALTRIALS.GOV ID: NCT**03561701



A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of VT-1161 Oral Capsules in the Treatment of Subjects with Recurrent Vulvovaginal Candidiasis

Study Number: VMT-VT-1161-CL-012

EudraCT Number: 2018-001270-26

**Version: 6 (Amendment 5)** 

Country-Specific Amendment: U.S. Only

Date of Issue: 01 October 2019

Mycovia Pharmaceuticals, Inc 4505 Emperor Boulevard, Suite 300 Durham, NC USA 27703

#### **Confidentiality Statement**

This document and the information it contains are confidential and the proprietary property of Mycovia Pharmaceuticals, Inc. The information is not to be disclosed or transmitted to any party without the written approval of Mycovia Pharmaceuticals, Inc. or its agents, and any such unauthorized use or disclosure is expressly prohibited.

# PROTOCOL SIGNATURE PAGE

A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of VT-1161 Oral Capsules in the Treatment of Subjects with Recurrent Vulvovaginal Candidiasis

Study Number: VMT-VT-1161-CL-012

EudraCT Number: 2018-001270-26

**Version: 6 (Amendment 5)** 

Country-Specific Amendment: U.S. Only

Date of Issue: 01 October 2019

Signatures of approval for protocol:

| Name | Signature | Date |
|------------------|-----------|------------|
| STEPHEN R. BRAND | Sall | 1 OCT 2019 |

# PROTOCOL SIGNATURE PAGE

A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of VT-1161 Oral Capsules in the Treatment of Subjects with Recurrent Vulvovaginal Candidiasis

Study Number: VMT-VT-1161-CL-012

EudraCT Number: 2018-001270-26

**Version: 6 (Amendment 5)** 

**Country-Specific Amendment: U.S. Only** 

Date of Issue: 01 October 2019

## Signatures of approval for protocol:

| Name | Signature | Date |
|------|-----------|------|

This study is to be performed in accordance with Good Clinical Practice, the ethical principles that have their origin in the Declaration of Helsinki, Title 21 of the Code of Federal Regulations, Parts 11 (Electronic Records; Electronic Signatures), 50 (Protection of Human Subjects), 54 (Financial Disclosure by Clinical Investigators), 56 (Institutional Review Boards), and 312 (Investigational New Drug Application), and International Conference on Harmonisation E6 (Guideline for Good Clinical Practice). Regulatory authorities, if required by national law, must give a favorable opinion/approval of the study protocol and amendments, informed consent and assent (for those ages 12 to 17) documents, and investigational brochure.

Study Sponsor:

Mycovia Pharmaceuticals, Inc.

4505 Emperor Boulevard, Suite 300, Durham, NC USA 27703

Sponsor Contact:

Stephen Brand, Ph.D.

Senior VP of Clinical Development

4505 Emperor Boulevard, Suite 300, Durham, NC USA 27703

Claude Hughes, M.D., Ph.D.

Medical Consultant

Medical Responsible: 4505 Emperor Boulevard, Suite 300, Durham, NC USA 27703

## **Investigator's Statement**

I have reviewed the protocol VMT-VT-1161-CL-012 entitled "A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of VT-1161 Oral Capsules in the Treatment of Subjects with Recurrent Vulvovaginal Candidiasis" and agree that it contains all the information necessary to conduct the study as required. I will conduct the study in accordance with the principles of International Conference on Harmonisation, Good Clinical Practice, and the Declaration of Helsinki.

I will maintain as confidential all written and verbal information provided to me by the Sponsor, including but not limited to, the protocol, case report forms, Investigational Brochure, material supplied at investigator meetings, minutes of teleconferences, etc. I agree that such material will only be provided as necessary to site personnel involved in the conduct of the study, the Institutional Review Board (IRB)/Independent Ethics Committee (IEC), regulatory authorities, or agencies as required by local law.

I will obtain written informed consent or assent (for those ages 12 to 17) from each prospective study subject or each prospective study subject's legal representative prior to conducting any protocol-specified procedures. The consent and assent forms used will have the approval of the IRB/IEC.

I will maintain adequate source documents and record all observations, treatments, and procedures pertinent to study subjects in their medical records. I will accurately complete the case report forms supplied by the Sponsor in a timely manner. I will ensure that my facilities and records are available for inspection by representatives of the Sponsor, the IRB/IEC, or other applicable regulatory authorities. I will ensure that my staff and I are available to resolve queries and meet with representatives of the Sponsor during regularly scheduled monitoring visits.

I will notify the Sponsor within 24 hours of any serious adverse events. Following this notification, a written report describing the serious adverse event will be provided to the Sponsor within 1 business day following the initial notification.

I acknowledge that I am responsible for the overall study conduct, and I agree to personally conduct and/or supervise the study. I will ensure that all associates, colleagues, and employees assisting in the conduct of the study, are informed and trained as necessary about their obligations and that there are adequate mechanisms in place for the site staff to receive the appropriate information throughout the study.

| Name | |
|-----------|------|
| Signature | Date |

Protocol VMT-VT-1161-CL-012

# PROTOCOL SYNOPSIS

**Title of Study:** A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of VT-1161 Oral Capsules in the Treatment of Subjects with Recurrent Vulvovaginal Candidiasis

**Protocol Number:** VMT-VT-1161-CL-012

**Interim Analysis:** No

**Investigational Medicinal Product:** VT-1161 capsules

Non-Investigational Medicinal Product: Fluconazole tablets or capsules

**Planned Number of Sites:** 60 to 80

Planned Number of Subjects: 600 screened; 300 randomized

Phase of Development: 3

#### **Introduction:**

VT-1161 is an orally-available inhibitor of fungal CYP51 that has shown high potency and selectivity in *in vitro* studies. VT-1161 blocks the production of ergosterol, an essential component of the fungal cell membrane, which is critical to fungal growth. *In vitro* and *in vivo* pharmacology studies have demonstrated that VT-1161 is highly active against *Candida albicans*, including fluconazole-resistant *C. albicans*, and non-albicans *Candida* species that cause vulvovaginal candidiasis (VVC). VT-1161 is highly selective for fungal CYP51 relative to off-target human CYP enzymes, and data to date suggest that it may avoid the side-effect profile that limits the use of commonly prescribed azole antifungal agents.

Oral VT-1161 has been evaluated in Phase 1 and 2 studies and shown to be safe, well tolerated, and highly effective in the treatment of vulvovaginal infections caused by *Candida* species. For example, in a Phase 2b study in subjects with recurrent VVC (RVVC), subjects in the 12-week VT-1161 treatment group (150 mg VT-1161 once daily for 7 days followed by 150 mg VT-1161 once weekly for 11 weeks) showed a 4.8% recurrence rate through Week 48 compared with a 52% recurrence rate in the placebo group in the intent-to-treat analysis.

RVVC, defined as 3 or more acute VVC episodes over a 12-month period, is experienced by 5 to 7 million women each year in the US. *Candida albicans* is the leading cause of recurrent vulvovaginal yeast infections in the United States. However, there has been an increasing trend in the number of vaginal yeast infections attributable to non-albicans species such as C. *glabrata* and C. *tropicalis*. In addition to the use of topical products to treat VVC, the majority of the women visiting healthcare professionals receive fluconazole for the treatment of each acute episode. A smaller percentage are prescribed a fluconazole maintenance regimen although fluconazole is not currently approved for the treatment of RVVC. Since some of the C. *albicans* and the majority of non-albicans isolates are resistant to fluconazole, the management of RVVC has become even more challenging.

In both nonclinical studies and clinical trials conducted to date, VT-1161 has demonstrated a favorable safety and tolerability profile, with no discernable adverse effect on liver function. In reproductive toxicity studies in pregnant rats or rabbits, VT-1161 was not teratogenic at any exposure studied. In a recent CYP3A4 drug-drug interaction study utilizing midazolam as the substrate, no clinically significant inhibition and only weak induction of midazolam metabolism was observed. These data are favorable when compared to other oral antifungal agents such as fluconazole.

Protocol VMT-VT-1161-CL-012

# **Objectives:**

#### Primary:

To evaluate the efficacy of oral VT-1161 in the treatment of RVVC through Week 48.

## Secondary:

- To evaluate the safety and tolerability of oral VT-1161 in the treatment of RVVC through Week 48.
- To evaluate the impact of oral VT-1161 treatment on patient reported outcomes through Week 48.

## Methodology:

#### Study Design:

This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled, parallel-group study. The study will evaluate the efficacy and safety of oral VT-1161 capsules in the treatment of subjects with RVVC. The impact of oral VT-1161 treatment will also be evaluated using data collected from patient reported outcome assessments.

Subjects must have a history of RVVC, defined as at least 3 episodes of acute VVC in the past 12 months, as described below:

- Subjects must have an acute VVC episode at the time of Screening, with a documented positive potassium hydroxide (KOH) or Gram stain performed at the investigative site
- Subjects must also have had 2 or more additional episodes of acute VVC in the past 12 months, with at least 1 of the episodes documented by a positive confirmatory laboratory test (i.e., culture, PCR, Affirm test, KOH test, Gram stain, a documented Papanicolaou (Pap) test, or other approved diagnostic tests)

The study consists of two Phases: 1) an open-label Induction Phase for the treatment of the acute VVC episode with 3 sequential 150 mg oral doses (every 72 hours) of fluconazole, and 2) a Maintenance Phase in which subjects will be randomly assigned to receive VT-1161 or placebo for 7 daily doses followed by 11 weekly doses and will then enter a 36-week follow-up period.

Once subjects have provided informed consent or assent (for those ages 12 to 17), the investigational site will evaluate all subjects by completing a review of pertinent medical history, obtaining vital signs, weight and height, electrocardiogram (ECG) and laboratory tests, reviewing clinical signs and symptoms of vulvovaginitis, performing a complete physical examination including speculum examination of the vagina, performing a KOH wet mount test or Gram stain from a vaginal smear to confirm the presence of yeast, and collecting vaginal swabs to establish a baseline culture for identification of fungal species. Patient reported outcome surveys (SF-36, EO-5D-3L or EO-5D-Y (for ages 12 to 17), WPAI:SHP, PHQ-9) for all regions and questions regarding their RVVC history (US only) will also be administered. Eligible subjects must have an acute VVC episode at Screening, defined as a total signs and symptoms score of ≥3 and a positive local KOH wet mount preparation or Gram stain from a vaginal smear revealing filamentous hyphae/pseudohyphae and/or budding yeast cells, and must meet other initial entry criteria. Once eligibility is confirmed, subjects will enter the Induction Phase. During the Induction Phase, the presenting acute VVC infection will be treated with 3 sequential 150 mg oral doses (every 72 hours) of fluconazole. Subjects will return approximately 14 days after the first dose of fluconazole

for evaluation. If the clinical signs and symptoms of the acute VVC infection have resolved (defined by a signs and symptoms score of <3), they will be randomized in a 2:1 ratio to receive either VT-1161 or a matching placebo regimen. Day 1 (Baseline) is defined as the first day of investigational medicinal product (IMP) administration and subsequent study days are defined by the number of consecutive days thereafter. If the acute VVC has not resolved (defined by a signs and symptoms score of  $\ge$ 3), the subject will be considered a screen failure and encouraged to see their physician for follow-up care.

#### Study Duration:

The planned study duration is expected to be approximately 26 months from screening of the first subject until last follow-up of the last subject.

## **Subject Participation:**

The duration of individual subject participation will be approximately 50 weeks, including the 2-week Induction Phase. See Table 1 for the Schedule of Assessments and Procedures which will be performed. After Screening, subjects will return to the clinic on Day 1 (Baseline), the start of the Maintenance Phase. Subjects will then have visits on Day 14 (±2 days), Weeks 6 (±7 days), 12 (±14 days), 18 (±14 days), 24 (±14 days), 30 (±14 days), 36 (±14 days), 42 (±14 days) and 48 (±14 days) (end of study [EOS]). Subjects who return to the clinic with a recurrent acute VVC episode should be evaluated as per the unscheduled visit noted in the Schedule of Assessment and Procedures.

## Scoring of Vulvovaginal Signs and Symptoms:

Vulvovaginal signs and symptoms will be evaluated at Screening and at each subsequent study visit. Each of the following vulvovaginal signs and symptoms will be scored and the individual scores combined, for a maximum score of 18 using the following scale:

- a. Signs: erythema, edema, and excoriation
- b. Symptoms: itching, burning, and irritation

Scoring Scale: Each score should be graded on a scale of 0 to 3 as follows:

- 0 = none (complete absence of any sign or symptom)
- 1 = mild (slight)
- 2 = moderate (present)
- 3 = severe (marked, intense)

## Mycology Assessment:

A local mycological assessment using KOH wet mount followed by microscopy or Gram stain will be evaluated at the Screening and at any study visit where a recurrent acute VVC episode is suspected. The investigative site is to use the same local mycology test (KOH or Gram stain) consistently for all subjects throughout the study. In addition, a vaginal swab for culture testing will be obtained and sent to the central mycology laboratory at the Screening and each subsequent study visit.

#### Plasma Pharmacokinetics:

Blood samples for assay of VT-1161 plasma concentrations will be collected from subjects at Baseline, Day 14, and Weeks 12, 24, 36, 48 and unscheduled visits.

## Safety:

Subject safety will be monitored by collection of adverse events (AEs), changes in vital signs, physical and vaginal exam parameters, ECGs, and safety laboratory parameters, including pregnancy tests for women of childbearing potential (WOCBP).

#### **Concomitant Medications:**

The following prescription and over-the-counter drug products are prohibited during the study and will be considered a protocol deviation:

- Topical or oral antifungal drugs (with the exception of fluconazole when prescribed by the Investigator to treat a subject with a recurrent VVC episode; refer to Section 8.1.12 on treatment options if fluconazole is ineffective).
- Topical products applied to the vulva or vagina (e.g. antibiotic, antitrichomonal, corticosteroids, or anti-inflammatory agents).
- 3. Oral antibacterial or antitrichomonal agents for the treatment of bacterial vaginosis, trichomonas, or other concomitant (urogenital) infection unless prescribed by the Investigator.
- Oral or injectable corticosteroid or immunosuppressive drugs for the duration of the study. Use of topical (no vulvar or vaginal steroids), inhaled, ophthalmic, collunarium/nasal, or intraarticular and intralesional steroids is permitted.
- 5. Drugs with a narrow therapeutic index that are metabolized by CYP3A4 and sensitive to induction of CYP3A4 (carbamazepine, cyclosporine, fentanyl, quinidine, sirolimus and tacrolimus).
- Vaginal douches or benzalkonium chloride disinfectant during the study.

#### **Number of Subjects (Planned):**

Approximately 600 screened and 300 randomized subjects are planned for this study. Assuming a 20% discontinuation rate for the duration of the study, approximately 240 subjects are expected to complete the study.

#### **Criteria for Inclusion and Exclusion:**

#### Criteria for Inclusion:

- 1) Subjects must be generally healthy, post-menarchal, non-pregnant females 12 years of age and older as of Screening. In Hungary, Romania, Ukraine, and Czech Republic only, subjects must be generally healthy, post-menarchal, non-pregnant females 18 years of age and older as of Screening.
- 2) Subjects must have a history of recurrent VVC as defined by three (3) or more episodes of acute VVC in the past 12 months, including the episode confirmed at Screening, with at least one episode (not including the current episode) documented by a positive culture, PCR, Affirm test, KOH test, Gram stain or a documented Pap test in the prior 12 months revealing filamentous hyphae/pseudohyphae and/or budding yeast cells, or other approved diagnostic tests.
- 3) Subjects must have an acute VVC episode at Screening, defined as:
  - a. a total signs and symptoms score of  $\geq 3$  and
  - b. a positive KOH wet mount preparation or Gram stain from a vaginal smear revealing filamentous hyphae/pseudohyphae and/or budding yeast cells.
- Subjects must have a composite vulvovaginal signs and symptoms score of <3 at the Baseline (Day 1) Visit.

- 5) Subjects must have a documented Pap test at Screening or within the timeline per current standard of care guidelines for the appropriate age requirement. Results must be either "negative for intraepithelial lesion or malignancy" or "ASCUS-atypical squamous cells of undetermined significance" (not applicable to subjects with a history of total hysterectomy).
- 6) Subjects must be suitable candidates for oral therapy and be able to swallow capsules intact.
- 7) Subjects must be willing and able to provide written informed consent or assent (for those ages 12 to 17) and authorization for use of protected health information.
- 8) Subjects must be willing and able to comply with protocol requirements, instructions, and protocol-stated restrictions and be likely to complete the study as planned.
- 9) Subjects of non-childbearing potential must meet the requirements defined below:
  - a. Pre-menopausal with documentation of surgical sterilization (i.e., hysterectomy, bilateral tubal ligation, bilateral oophorectomy, or bilateral salpingectomy) at least 3 months prior to Screening.
  - b. Post-menopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments at Screening.
- 10) Subjects of childbearing potential (includes ages 12-17) must use 1 of the following methods of contraception during the study through Week 48:

**OPTION 1** – Highly effective methods that can be used alone:

- i. Copper intrauterine device
- ii. Levonorgestrel-releasing intrauterine system
- iii. Progestin implant
- iv. Monogamous with a vasectomized male partner
- v. Abstinence<sup>a</sup>

**OPTION 2** – Acceptable first and second barrier methods to be used in combination:

FIRST (Hormonal Contraception)<sup>b</sup>

- 1. Estrogen & progestin oral contraceptives, transdermal patch or vaginal ring.
- 2. Progestin only oral contraceptives or injection

SECOND (Barrier Method)

- 1. Diaphragm (with spermicide)
- 2. Cervical cap (with spermicide)
- 3. Male condom (with or without spermicide)

In addition to OPTIONS 1 and 2, subjects of childbearing potential (includes ages 12-17) may also use 1 of the following methods of contraception after completing the Induction Phase on Study Day 1 through Week 48:

**OPTION 3 (Day 1 – Week 48)**<sup>c</sup> – Acceptable first and second barrier methods to be used in combination:

FIRST (Barrier Method)

- 1. Diaphragm (with spermicide)
- 2. Cervical cap (with spermicide)

SECOND (Barrier Method)

1. Male condom (with or without spermicide)

<sup>a</sup> Sexual abstinence is defined as refraining from heterosexual intercourse during the entire study period and where this is the usual life style of the subject. Periodic abstinence (calendar, symptothermal, postovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not considered to be acceptable methods of contraception.

Protocol Synopsis Protocol VMT-VT-1161-CL-012

<sup>b</sup> Subjects who started taking a hormonal contraceptive less than 3 months prior to the first dose of fluconazole must agree to use a double-barrier method (i.e. diaphragm plus spermicide or condom) through 3 months after starting the hormonal contraceptive.

<sup>c</sup>Because of the teratogenic risk associated with repeat dosing of fluconazole, OPTION 3 contraceptive methods cannot be used during Screening and the Induction Phase of the study [from Screening (Day 1) until Day 14 of the study].

#### Criteria for Exclusion:

- 1) Subjects must not have the presence of concomitant vulvovaginitis caused by other pathogens (e.g., bacterial vaginosis, *Trichomonas vaginalis*, *Chlamydia trachomatis*, or *Neisseria gonorrhoeae*) at Screening visit and at the Day 1 visit if an infection is suspected.
- 2) Subjects must not have an active HPV infection as evidenced by visible condylomas on vulvovaginal examination at Screening and Day 1 visits.
- 3) Subjects must not have the presence or a history of another vaginal or vulvar condition(s) that in the Investigator's opinion would confound the interpretation of clinical response.
- 4) Subjects must not have a history of cervical cancer.
- 5) Subjects must not use any systemic (e.g., oral or injectable) corticosteroid therapy during the study or within 30 days prior to Screening, nor use of topical vulvar or vaginal steroids during the study or within 7 days prior to Screening. However, use of topical (no vulvar or vaginal steroids), inhaled, ophthalmic, collunarium/nasal, intraarticular and intralesional steroids is permitted.
- 6) Subjects must not use any systemic (e.g., oral or injectable) or topical (applied to the vulva or vaginal area) antifungal, antibacterial, or antitrichomonal drugs or vaginal douches during the study (unless prescribed by the Investigator) or within 7 days prior to Screening.
- 7) Subjects must not be using drugs with a narrow therapeutic index that are metabolized by CYP3A4 and sensitive to induction of CYP3A4 during the study (carbamazepine, cyclosporine, fentanyl, quinidine, sirolimus and tacrolimus).
- 8) Subjects must not use any vaginal estrogen replacement therapy, ospemifene, Vitamin E gel capsules (vaginally) or lubricants within 7 days prior to Screening.
- 9) Subjects must not have a condition that would require treatment during the study with concomitant topical (applied to vulva and vagina) or systemic antimicrobial therapy for any reason.
- 10) Subjects must not have received an immunosuppressive medication (e.g. cyclosporine, tacrolimus, methotrexate, 6-mercaptopurine, mycophenolate, etc.), or radiation therapy within 3 months prior to Screening or have a medical condition where it would be likely that the subject may need to use these therapies during the study.
- 11) Subjects must not have evidence of any clinically significant major organ disease or current clinically significant infection or any other conditions (with the exception of acute VVC) that may affect the clinical assessment of RVVC per investigator judgment.
- 12) Subjects must not have any comorbid condition that in the opinion of the Investigator would preclude the safe participation of the subject in the study or would prevent the subject from meeting the study requirements.
- 13) Subjects must not have any condition that in the opinion of the investigator could impact drug absorption (e.g. gastrectomy, Roux-en-Y gastric bypass surgery, gastric bands or staples, etc.), distribution, or elimination.
- 14) Subjects must not have poorly controlled diabetes mellitus (HbA1c  $\geq 8.5\%$  at Screening).
- 15) Subjects must not have moderate or severe hepatic and/or renal disease (defined in Appendix B and

CONFIDENTIAL

## Appendix C).

- 16) Subjects must not have a laboratory abnormality that in the opinion of the Investigator is likely to introduce additional risk to the subject or might interfere with data interpretation. The specific findings listed below are excluded at Screening (a single repeat laboratory evaluation is allowed for eligibility determination, except for HIV, HbsAg and antibodies to hepatitis C virus):
  - a. Serum alanine aminotransferase (ALT)  $\geq$ 2.0x the upper limit of normal (ULN) of the reference range.
  - b. Serum aspartate aminotransferase (AST)  $\geq$ 2.0x the ULN of the reference range.
  - c. Serum total bilirubin  $\ge 1.5x$  the ULN of the reference range, unless the elevation is consistent with Gilbert's Syndrome.
  - d. Electrocardiographic QTc interval >470 msec as corrected by the Fridericia formula, or any clinically significant electrocardiographic abnormality.
  - e. Positive test for antibodies to human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or antibodies to hepatitis C virus.
- 17) Subjects of childbearing potential must not be pregnant (positive pregnancy test at Screening), lactating, or planning to become pregnant during the study period.
- 18) Subjects must not have planned surgery or other medical procedures that in the Investigator's opinion would impact compliance with the protocol.
- 19) Subjects must not have active substance abuse (e.g., drugs of any kind, including alcohol) or any other medical, psychiatric or social condition that in the Investigator's opinion would preclude compliance with the protocol.
- 20) Subjects must not have received VT-1161 study medication in a previous study.
- 21) Subjects must not have received any IMP in a clinical trial within 5 half-lives of that IMP prior to Screening (if unknown, 60 days prior to Screening).
- 22) Subjects must not have a known history of intolerance or hypersensitivity to azole antifungal drugs (e.g., fluconazole, itraconazole, voriconazole, posaconazole, and isavuconazole), or any excipients of the capsule formulation.

## **Induction Phase Treatment:** Fluconazole 150 mg tablets or capsules

#### Dose and Mode of Administration:

Oral administration of 3 sequential doses (every 72 hours) of fluconazole 150 mg starting at Screening (Day -14).

#### Maintenance Phase Test Product: VT-1161 150 mg capsules

#### Dose and Mode of Administration:

Oral administration of VT-1161 within 30 minutes after ingestion of the subject's main meal of the day (as determined by the subject and kept consistent throughout the duration of the study). Approximately 240 mL (approx. 8oz) of water is to be consumed with each dose of IMP.

Starting at Baseline (Day 1), loading doses of 150 mg (1 capsule) once daily for 7 days, followed by doses of 150 mg (1 capsule) once weekly for 11 weeks.

Duration of Administration: 12 weeks

#### Maintenance Phase Reference Product: Matching Placebo capsules

#### Dose and Mode of Administration:

Oral administration of placebo within 30 minutes after ingestion of the subject's main meal of the day (as determined by the subject and kept consistent throughout the duration of the study). Approximately 240 mL (approx. 8oz) of water is to be consumed with each dose of IMP.

Starting at Baseline (Day 1), loading doses of placebo once daily for 7 days, followed by doses of placebo (1 capsule) once weekly for 11 weeks.

Duration of Administration: 12 weeks

#### **Study Populations:**

Intent-to-Treat (ITT) Population: All randomized subjects.

Safety Population: All randomized subjects who received at least 1 dose of IMP.

<u>Per Protocol Population (PP):</u> All randomized subjects who had the following:

- Had no deviations to inclusion/exclusion criteria that could impact treatment outcome.
- Were compliant with the assigned study treatment, defined as  $\ge 80\%$  compliance during the daily dosing phase and  $\ge 50\%$  compliance during the weekly dosing phase.
- Had the Week 48 visit completed within the acceptable time window ( $\pm 14$  days).
- Had no major protocol violations that would impact treatment outcome.

Modified ITT: All randomized subjects who had the following:

- Positive KOH or Gram stain at Screening.
- Positive culture at Screening.
- Negative culture at Baseline.

#### **Criteria for Evaluation:**

#### Efficacy:

Clinical and mycological assessments will be conducted as outlined in Table 1. Schedule of Assessments and Procedures.

All efficacy analyses will be performed on the ITT, PP, and mITT Populations.

The primary efficacy outcome measure is the proportion of subjects with one or more culture-verified acute VVC episodes during the Maintenance Phase (post-randomization through Week 48) in the ITT population. An acute VVC episode during the Maintenance Phase (considered a recurrent episode) is defined as a positive culture for *Candida* species and a clinical signs and symptoms score of  $\geq 3$ .

The key secondary efficacy outcome measures include the following:

- a. Time to first recurrence of a culture-verified acute VVC episode with signs and symptoms score ≥3 during the Maintenance Phase.
- b. The proportion of subjects with at least one positive culture for Candida during the Maintenance Phase.

CONFIDENTIAL

Protocol Synopsis
Protocol VMT-VT-1161-CL-012

- c. The proportion of subjects with at least one culture-verified acute VVC episode with signs and symptoms of ≥3 post randomization through Week 24.
- d. Change from Screening through Week 48 in the SF-36 mental component score (MCS).
- e. Change from Screening through Week 48 in the SF-36 patient reported outcome survey total score.

#### Safety:

All safety analyses will be performed on the Safety Population. AEs will be collected throughout the study. Physical and vaginal examination findings and vital signs will be recorded at Screening and throughout the study per Table 1. Schedule of Assessments and Procedures. ECGs and safety laboratory tests (hematology, chemistry, and urinalysis) will be obtained throughout the study. All concomitant medications taken during the period from 30 days prior to Screening through the Week 48 (EOS) visit will be recorded in the case report form (CRF). Pertinent and all major medical conditions will be recorded on the Medical History CRF.

Subject who want to discontinue from the study should be encouraged to remain in the study for all remaining visits through Week 48 for safety and efficacy assessments. All subjects who discontinue early from the study should have all EOS procedures performed on the day of discontinuation.

## **Statistical Methods and Data Analysis:**

A statistical analysis plan will be finalized before 50% of subjects are enrolled.

#### **Efficacy Analysis:**

The primary statistical objective of this study is to determine if there are differences in the proportions of subjects with one or more episodes of culture-verified acute VVC in those receiving VT-1161 compared to those receiving placebo during the Maintenance Phase.

A sample size of 68 active subjects and 34 placebo subjects provides at least 95% power to detect a treatment difference of 35% between the VT-1161 treatment group and the placebo treatment group in percentage of subjects with at least one or more culture-verified acute VVC episodes during the Maintenance Phase (post randomization through Week 48). (PASS 2008: Fisher's exact test, two-sided alpha=0.05, and assuming 50% of placebo subjects have recurrence). Based on an estimated 20 % discontinuation rate, approximately 128 total subjects (85 active, 43 placebo) will be necessary for randomization to arrive at approximately 102 evaluable subjects.

## Safety Analysis:

AEs will be coded using the Medical Dictionary for Regulatory Activities® dictionary. The number and percentage of subjects reporting treatment-emergent AEs will be tabulated by system organ class, preferred term, and greatest severity with a breakdown by treatment group. Mean changes from pretreatment in vital signs, ECG, and clinical laboratory variables will be summarized by treatment group.

#### Pharmacokinetics:

No formal statistical hypothesis testing related to pharmacokinetics will be conducted. VT-1161 concentrations will be presented by visit with descriptive statistics. The pharmacokinetic data will be

used in a cross-population pharmacokinetic analysis that will be presented in a separate report.

## Patient Reported Outcomes:

The SF-36, EQ-5D-3L or EQ-5D-Y (for ages 12 to 17), WPAI:SHP, and PHQ-9 patient reported outcome surveys will be administered at Screening, Week 24 (EOT) and Week 48 (EOS) for all regions. At Screening, subjects will also be required to answer questions regarding their RVVC history (US only).

Protocol VMT-VT-1161-CL-012

Table 1. Schedule of Assessments and Procedures

| Table 1. Seneture of Assessments | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Activities | Screening<br>Day -14<br>(±2 days) | Baseline<br>(Day 1) | Day 14<br>(±2 days) | Week 6<br>(±7 day s) | Week 12<br>(±14 days)<br>EOT | Week 18<br>(±14 days) | Week 24 (± 14 days) | Week 30 (± 14 days) | Week 36<br>(± 14 days) | Week 42<br>(± 14 days) | Week 48<br>(± 14 days)<br>EOS | Unscheduled<br>Visit |
| Sign Informed Consent or Assent Form | X | *** | | | | | | | | | | |
| Inclusion/Exclusion Criteria | X | X | | | | | | | | | | |
| Medical/Surgical History | X | | | | | | | | , | | | |
| Prior/Concomitant Medications/Treatments <sup>a</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| Collect and Record AEs | | X | X | X | X | X | X | X | X | X | X | X |
| Patient Reported Outcome Surveysb | X | | | | 3 | | X | | | | X | X |
| RVVC History Questionnaire (US Only) | X | | | | | | | | | | () | |
| Body Height and Weight | X | | | | Xc | | Xc | | | | Xc | |
| Vital Signs <sup>d</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| Physical and Vaginal Examination | X | Xe | Xe | $\mathbf{X}^{e}$ | Xe | Xe | Xe | Xe | Xe | Xe | Xe | Xe |
| Clinical Signs and Symptoms of Vulvovaginitis | X | X | X | X | X | X | X | X | X | X | X | X |
| Local KOH Wet Mount or Gram Stain | X | | | | | | | | | | | X |
| Central Vaginal Fungal Culture | X | X | X | X | X | X | X | X | X | X | X | X |
| ECG | X | X | X | | X | | X | | | 2 2<br>3 3 | X | |
| PK Samples <sup>f</sup> | | X | X | * | X | | X | | X | | X | X |
| Clinical Laboratory Samples <sup>g</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| Urinalysis | X | X | X | | X | | X | | X | | X | |
| Hematology (CBC with differential) | X | X | X | | X | | X | | X | | X | |
| HIV Ab, HbsAg, anti-HCV | X | | | | | | | | | | | |
| Central Serum Pregnancy Testh (WOCBP) | X | X | | 2 | X | | X | | | | X | |
| Local Urine Pregnancy Testh (WOCBP) | X | X | X | X | X | X | X | X | X | X | X | X |
| Administer Fluconazole | X | | | | | | | | | | | |
| Randomization | | X | | | | | | | | | | |
| Administer and/or Review IMPi | | X | X | X | X | | | | | | | |

Abbreviations noted above – AEs: adverse events; CBC, complete blood count; ECG: electrocardiogram; EOS: End of Study; EOT: End of Treatment; HbsAg: Hepatitis B surface antigen; HCV: Hepatitis C virus; HIV: human immunodeficiency virus; IMP, investigational medicinal product; KOH: potassium hydroxide prep; PK: pharmacokinetic; WOCBP: women of childbearing potential.

Protocol VMT-VT-1161-CL-012

- a. All medication taken 30 days prior to Screening and all non-pharmacologic treatments received 72 hours prior to Screening will be recorded through the EOS visit.
- b. SF-36, EQ-5D-3L or EQ-5D-Y (for ages 12 to 17), WPAI:SHP, and PHQ-9 patient reported outcome surveys.
- c. Weight only.
- d. Vital signs include sitting heart rate, blood pressure, temperature, and respiratory rate.
- e. Limited physical examination, i.e. vaginal speculum examination plus a symptom directed physical examination.
- f. The initial PK sample must be drawn prior to the first dose of study drug (placebo/VT-1161).
- g. Serum chemistry (creatinine, BUN, AST, ALT, alkaline phosphatase, total bilirubin, conjugated bilirubin, albumin, total protein, total carbon dioxide, glucose, sodium, potassium, chloride, calcium, and phosphorus, creatine phosphokinase [CK], cholesterol, and triglycerides). Testing for HbA1c is performed for all subjects at Screening. Cultures to test for *Chlamydia trachomatis* and *Neisseria gonorrhoeae* will be taken at Screening and sent to the central lab. Testing for bacterial vaginosis will be done locally at Screening. An OSOM® Rapid test or similar test will be performed for *Trichomonas vaginalis* locally at Screening.
- h. For WOCBP, a local lab urine pregnancy test will be obtained at every study visit. A central lab serum pregnancy test will also be performed at Screening, Baseline, and Weeks 12, 24, and 48.
- i. IMP is to be administered within 30 minutes after the subject's main meal of the day (as determined by the subject) at approximately the same time of the day consistently throughout the study. Approximately 240 mL (approx. 8 oz.) of water is to be consumed with each dose of IMP. Remind subject to bring IMP to each visit to ensure compliance.
- j. All procedures listed are to be completed only for unscheduled visits where a recurrent VVC episode is suspected. If the unscheduled visit is for repeat procedures (i.e., ECG, safety labs, etc.), only those specific procedures need to be performed, along with collection of any changes in medical treatments or medications and collection of any AEs.

# TABLE OF CONTENTS

| PROTO | OCOL SIGNATURE PAGE | 2 |
|--------|------------------------------------------------------------|----|
| PROTO | OCOL SYNOPSIS | 5 |
| TABLE | OF CONTENTS | 17 |
| LIST O | F TABLES | 21 |
| LIST O | F APPENDICES | 22 |
| LIST O | F ABBREVIATIONS AND DEFINITION OF TERMS | 22 |
| 1 | INTRODUCTION | 25 |
| 1.1 | Background Information | 25 |
| 1.1.1 | Vulvovaginal Candidiasis | 26 |
| 1.2 | VT-1161 | 28 |
| 1.2.1 | Non-Clinical Pharmacology | 29 |
| 1.2.2 | Clinical Studies | 32 |
| 1.3 | Study Rationale | 41 |
| 1.3.1 | Rationale for Induction Phase Treatment | 41 |
| 1.3.2 | Dosing Regimen for VT-1161 and Matching Placebo | 42 |
| 1.4 | Potential Risks and Benefits of Participating in the Study | 42 |
| 2 | OBJECTIVES | 43 |
| 3 | STUDY ENDPOINTS | 44 |
| 4 | STUDY DESIGN | 45 |
| 4.1 | Overall Study Design | 45 |
| 4.2 | Treatment Arms and Duration of Study | 46 |
| 4.3 | Number of Subjects | 46 |
| 4.4 | Design Justification | 46 |
| 4.4.1 | Justification for Inclusion of Adolescents in the Study | 48 |
| 5 | SELECTION OF STUDY POPULATION | 50 |
| 5.1 | Inclusion Criteria | 50 |
| 5.2 | Exclusion Criteria | 52 |
| 6 | INVESTIGATIONAL MEDICINAL PRODUCT | 55 |
| 6.1 | Fluconazole | 55 |

| 6.2 | Description of Investigational Medicinal Product | 55 |
|---|---|---|
| 6.2.1 | VT-1161 | 55 |
| 6.2.2 | Placebo | 55 |
| 6.3 | Investigational Medicinal Product Labeling and Packaging | 55 |
| 6.4 | Investigational Medicinal Product Storage Conditions | 55 |
| 6.5 | Receipt of Supplies/Handling/Storage | 56 |
| 6.6 | Investigational Medicinal Product Accountability | 56 |
| 6.7 | Investigational Medicinal Product Return | 56 |
| 7 | TREATMENT OF SUBJECTS | 57 |
| 7.1 | Investigational Medicinal Product Administration and Dosing Schedule | 57 |
| 7.1.1 | Induction Phase (Screening to Day 1 Pre-Randomization) | 57 |
| 7.1.2 | Maintenance Phase (Day 1 Post Randomization to Week 12) | 57 |
| 7.2 | Method of Assigning Subjects to Treatment Groups | 58 |
| 7.3 | Dose Interruptions and Modifications | 58 |
| 7.4 | Prohibited and Permitted Medications/Non-Medications | 58 |
| 7.4.1 | Prohibited Medications/Non-Medications | 59 |
| 7.4.2 | Permitted Medications/Non-Medications | 59 |
| 7.5 | Treatment Compliance | 59 |
| 7.6 | Replacement of Study Subjects | 60 |
| 7.7 | Randomization and Blinding | 60 |
| 7.8 | Conditions for Breaking the Blind | 60 |
| 7.9 | Treatment After the End of the Study | 61 |
| 8 | STUDY PROCEDURES | 62 |
| 8.1 | Assessments and Procedures | 62 |
| 8.1.1 | Screening Assessments and Procedures (Day -14 ±2 Days) | 65 |
| 8.1.2 | Baseline (Day 1) Assessments and Procedures (Day -14 ±2 Days) | 67 |
| 8.1.3 | Day 14 (±2 Days) Assessments and Procedures | 68 |
| 8.1.4 | Week 6 (±7 Days) Assessments and Procedures | 69 |
| 8.1.5 | Week 12 (±14 Days) Assessments and Procedures | 69 |
| 8.1.6 | Week 18 (±14 Days) Assessments and Procedures | 71 |
| 8.1.7 | Week 24 (±14 Days) Assessments and Procedures | 71 |

| 8.1.8 | Week 30 (±14 Days) Assessments and Procedures | 72 |
|--------|----------------------------------------------------------------|----|
| 8.1.9 | Week 36 (±14 Days) Assessments and Procedures | 73 |
| 8.1.10 | Week 42 (±14 Days) Assessments and Procedures | 74 |
| 8.1.11 | Week 48 (±14 Days) Assessments and Procedures (End of Study) | 75 |
| 8.1.12 | Unscheduled Visit Assessment and Procedures | 76 |
| 8.2 | Exercise | 77 |
| 9 | SAFETY ASSESSMENTS | 78 |
| 9.1 | Safety Tests and Assessments | 78 |
| 9.1.1 | Height and Weight | 78 |
| 9.1.2 | Vital Signs | 78 |
| 9.1.3 | Physical Examination | 78 |
| 9.1.4 | Electrocardiograms | 78 |
| 9.1.5 | Laboratory Determinations | 79 |
| 9.1.6 | KOH Wet Mount Tests or Gram Stains and Fungal Cultures | 80 |
| 9.1.7 | Vulvovaginitis Clinical Assessment | 81 |
| 9.2 | Adverse Event Reporting | 81 |
| 9.2.1 | Definition of Adverse Events | 81 |
| 9.2.2 | Definition of a Serious Adverse Event | 82 |
| 9.2.3 | Recording of Adverse Events | 84 |
| 9.2.4 | Severity of Adverse Events | 84 |
| 9.2.5 | Causality Assessment | 85 |
| 9.2.6 | Action Taken Following Adverse Events | 87 |
| 9.2.7 | Outcome of Adverse Events | 87 |
| 9.2.8 | Other Reportable Events | 88 |
| 10 | PHARMACOKINETIC ASSESSMENTS | 89 |
| 10.1 | Sample Collection and Handling | 89 |
| 10.2 | Analytical Procedures | 89 |
| 10.3 | Pharmacokinetic Parameters | 89 |
| 11 | STUDY TERMINATION AND SUBJECT DISCONTINUATION | 90 |
| 11.1 | Screening/Baseline Failures | 90 |
| 11.2 | Subject Withdrawal or Premature Discontinuation from the Study | 90 |

| 11.3 | Subject and Study Completion | 91 |
|---|---|---|
| 11.4 | Premature Study Termination | 92 |
| 12 | STATISTICAL ANALYSIS | 93 |
| 12.1 | Determination of Sample Size | 93 |
| 12.2 | Analysis Populations | 94 |
| 12.3 | Demographic and Baseline Characteristic Analyses | 95 |
| 12.4 | Efficacy Analyses | 95 |
| 12.5 | Safety Analyses | 96 |
| 12.6 | Pharmacokinetic Analyses | 98 |
| 12.7 | Patient Reported Outcome | 98 |
| 13 | CLINICAL STUDY ADMINISTRATION/STUDY GOVERNANCE CONSIDERATIONS | 99 |
| 13.1 | Ethical Conduct of Study | 99 |
| 13.2 | Informed Consent and Assent | 99 |
| 13.3 | Quality Control (Study Monitoring) | 99 |
| 13.4 | Quality Assurance | 100 |
| 13.5 | Compliance with Standards of Medical Research/ Deviations | 100 |
| 13.6 | Data Management | 101 |
| 13.7 | Study and Site Closure | 102 |
| 13.8 | Records Retention | 102 |
| 13.9 | Disclosure of Data | 103 |
| 13.10 | Financial Disclosure | 103 |
| 13.11 | Publication Policy | 104 |
| 13.12 | Confidentiality | 104 |
| 13.12.1 | Data | 104 |
| 13.12.2 | Subject Anonymity | 104 |
| 14 | REFERENCES | 105 |

# LIST OF TABLES

| Table 1. | Schedule of Assessments and Procedures | 15 |
|----------|-------------------------------------------------------|----|
| Table 2. | Oral Agents Commonly Used to Treat VVC | 28 |
| Table 3. | VT-1161 Antifungal MIC <sub>50</sub> or Range (μg/mL) | 30 |

# **LIST OF APPENDICES**

Appendix A. Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Table (Draft November 2007)

- Appendix B. Grading of Renal Impairment
- Appendix C. Child-Pugh Classification of Hepatic Impairment
- Appendix D. SF-36<sup>TM</sup> Quality of Life Questionnaire
- Appendix E. EQ-5D-3L Health Status Questionnaire
- Appendix F. EQ-5D-Y Health Status Questionnaire
- Appendix G. Work Productivity and Activity Impairment: Specific Health Problems

Questionnaire

- Appendix H. Patient Health Questionnaire 9
- Appendix I. RVVC History Questionnaire (Version 01)
- Appendix J. Extension Study – U.S. Only
- Appendix K. Protocol Amendment Summary of Changes

# LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

AbbreviationDefinition or TermAEadverse event

ALT alanine aminotransferase
AST aspartate aminotransferase

AUC area under the curve CK creatine phosphokinase

C<sub>max</sub> maximum plasma concentration

CRF case report form

CYP51 lanosterol demethylase DDI drug-drug interaction

DMID Division of Microbiology and Infectious Diseases

ECG electrocardiogram

eCRF electronic case report form
EDC electronic data capture

EOS end of study

FDA Food and Drug Administration

GCP good clinical practice

HbsAg hepatitis B surface antigen

HIV human immunodeficiency virus

IC<sub>50</sub> half maximal inhibitory concentration ICH International Conference on Harmonization

IEC Independent Ethics Committee
IMP investigational medicinal product

IRB institutional review board

ITT intent-to-treat

IWRS interactive web response system

KOH potassium hydroxide

MedDRA Medical Dictionary for Regulatory Activities

MCS Mental Component Score

MIC<sub>50</sub> minimum inhibitory concentration NOAEL no-observed-adverse-effect-level

OM onychomycosis
Pap Papanicolaou
PK pharmacokinetic

PKE pharmacokinetic evaluation

PP per protocol

QTc Fridericia correction

RVVC recurrent vulvovaginal candidiasis

Protocol VMT-VT-1161-CL-012 Ver. 6 U.S. Only, 01 October 2019

Abbreviation **Definition or Term** serious adverse event SAE SAP statistical analysis plan

TEAE treatment-emergent adverse event

 $T_{\text{max}}$ time to reach maximum plasma concentration

TOC test of cure

ULN upper limit of normal VVC vulvovaginal candidiasis

women of childbearing potential WOCBP

Work Productivity and Activity Impairment: Specific Health Problems WPAI:SHP

## 1 INTRODUCTION

Lanosterol demethylase (CYP51), an enzyme essential for fungal growth, catalyzes an early step in the biosynthetic pathway of ergosterol, a sterol required for fungal cell membrane formation and integrity (Yoshida, 1988). Inhibition of CYP51 results in the accumulation of 14-methylated sterols, some of which are toxic to the fungus. CYP51 is the molecular target of the class of drugs referred to as 'azole antifungals'. All currently approved azole drugs contain either an imidazole or triazole ring system that binds tightly to the catalytic heme-iron of fungal CYP51 as well as to the heme-iron of many off-target mammalian cytochrome P450 enzymes. This inherent lack of selectivity is responsible for many of the side effects associated with the azole antifungals. For example, the potent inhibition of one or more human cytochrome P450 metabolizing enzymes found in the liver (e.g. CYP3A4, CYP2C9, CYP2C19) or in the adrenal and sex organs (e.g. CYP19, CYP17, CYP21), is the basis for azole drug-drug interactions (Bates and Yu, 2003) and reproductive warnings (Zarn et al., 2003), respectively. Additional azole class toxicities that are less well understood but may be related to off-target protein interactions include hepatic toxicities, skin photosensitivity, and vision impairment. In the acute care setting, these doselimiting side effects prevent attainment of plasma drug levels that might reduce the longstanding 40% mortality rate attributed to invasive fungal infections. The safety profile of the class similarly limits its use for chronic treatment of non-life-threatening fungal infections, such as onychomycosis (OM) and recurrent vulvovaginal candidiasis (VVC). A safer antifungal drug would also improve treatment options for infections seen in otherwise healthy individuals, such as OM and recurrent VVC, which require protracted treatment in a patient population where significant side-effect risks are unacceptable.

## 1.1 Background Information

Mucosal candidiasis, also known as thrush, describes a group of yeast-like fungal infections that involve the mucous membranes including the mouth, urinary tract and genitals, notably the vagina and surrounding skin in women. Infection is typically caused by *Candida albicans*, however more rare and difficult-to-treat Candida strains such as *C. glabrata* are becoming more prevalent. Mucosal candidiasis occurs more frequently in immunocompromised patients, but may also arise in immunocompetent individuals.

## 1.1.1 Vulvovaginal Candidiasis

# 1.1.1.1 Epidemiology

Symptoms of vulvovaginitis (inflammation of the vagina and vulva) are common and are among of the most frequent reasons for women's visits to physicians. Vulvovaginitis is associated with considerable morbidity including genital discomfort, decrease in sexual pleasure, loss of productivity, and psychological distress (Eschenbach, 2004). There are several etiologies for vulvovaginitis; candidiasis being the second most common after bacterial vaginitis. Vulvovaginal candidiasis is a common disorder, with nearly 75% of all adult women having had at least one "yeast infection" in their lifetime. Approximately half of these women experience a recurrence, with 5 to 8% developing recurrent VVC, defined as 3 or more episodes in one year (Sobel, 2016). Estrogen increases the glycogen concentration of the vaginal lining; glycogen is a substrate on which *C. albicans* thrives. As estrogen levels are significantly lower in both pre-menarcheal and post-menopausal females, the incidence of VVC is lower in these populations. Vulvovaginal candidiasis is most common in women aged 25 to 34 years (Foxman et al., 2013).

## 1.1.1.2 Pathophysiology

Vulvovaginal candidiasis occurs when there is an overgrowth of the normal yeast in the vagina. Most cases (85% - 95%) are caused by *C. albicans*, followed by *C. glabrata*, and infrequently by *C. parapsilosis*, *C. tropicalis*, and *C. krusei*. Vulvovaginitis caused by non-albicans Candida species, in particular *C. glabrata*, is clinically indistinguishable from *C. albicans* VVC but is more resistant to current treatments.

Candida organisms gain access to the lumen and secretions of the vagina primarily from the adjacent perianal region. Normal anti-candida defense mechanisms allow for long-term persistence of Candida as commensal organisms in the vagina without signs or symptoms of vaginitis. Factors predisposing to VVC versus asymptomatic colonization include those attributed to the health (immunosuppression, use of antibacterial agents, pregnancy, uncontrolled diabetes mellitus) and behavior (frequent intercourse, orogenital sexual activity, use of oral contraceptives or estrogen-based hormonal replacement therapy) of the host. Other dermatologic conditions such as psoriasis, lichen planus, and lichen sclerosus also predispose women to VVC (Goncalves et al., 2016).

#### 1.1.1.3 Presentation and Diagnosis

The clinical array of signs and symptoms of VVC include genital pruritus associated with edema, an erythematous rash and excoriation of the vulva and surrounding skin, a burning sensation in the vagina and vulva, and a vaginal discharge. These symptoms may persist for days to weeks, and

may also recur with each menstrual cycle. Women with VVC typically most commonly present with acute pruritus and a vaginal discharge, though neither is specific for candidiasis. The discharge may range from being watery to quite thick and "cottage-cheese-like". Common symptoms include vaginal soreness, irritation, vulvar burning, dyspareunia, and external dysuria. Physical examination typically reveals erythema and edema of the vulva with fissures and a pustulopapular rash, vaginal erythema, and a normal cervix. Symptoms often worsen the week prior to menses.

The diagnosis of VVC requires more than a history and physical examination as symptoms and signs, in particular pruritus, are often non-specific. Diagnosis is made by microscopic examination of a 10% potassium hydroxide (KOH) wet mount showing the presence of yeast cells and mycelia and the absence of both clue cells (pathognomonic of bacterial infection) and trichomonads. The vaginal pH is normal, approximately 4.0. A vaginal culture should also be performed, particularly for women with negative microscopy, as up to 50% of patients with culture-positive VVC will have no findings on microscopy (Sobel, 2007); additionally, a culture will precisely identify the organism. Papanicolaou (Pap) smears are also not reliable, typically positive in only a quarter of patients with VVC.

As up to 15% of asymptomatic women are colonized with Candida species and are thus culture positive, the final diagnosis of VVC requires a comprehensive assessment of clinical findings, microscopic examination, and vaginal culture.

## 1.1.1.4 Treatment and Outcome

In general, women who are asymptomatic carriers of Candida do not require treatment. Acute VVC in symptomatic women requires individualized treatment, the selected agent and duration of therapy being based on whether the VVC is categorized as either:

- Uncomplicated, defined as having all of the following characteristics: (mild or moderate in symptom severity, sporadic in frequency, *C. albicans* as the infecting organism, in non-pregnant women with normal immune function), or
- Complicated, defined as having any one or more of the following characteristics: severe in symptom severity, recurrent, a non-*C. albicans* organism as the infecting agent, abnormal immune function, or pregnant (Eschenbach, 2004).

Women with uncomplicated VVC can be treated with single-dose or short-course treatments, while those with complicated VVC require longer-term therapy, at least 5 to 7 days and possibly

maintenance therapy up to 6 months (Sobel et al., 2004). Pregnant women, who are at higher risk of developing VVC, can only be treated with topical agents because of the potential teratogenic effects of azoles when administered systemically. Topical agents are limited by local side effects, especially burning, and are messy to apply; therefore, most patients prefer the oral regimens. However, the systemically administered azoles listed in Table 2 are characterized by systemic toxicities and drug-drug-interactions (DDIs) and have poor activity against *C. glabrata* and fluconazole resistant C. *albicans*.

Table 2. Oral Agents Commonly Used to Treat VVC

| Agent | Formulation | Dose and Schedule |
|--------------------------|--------------------|--------------------|
| Fluconazole (Diflucan®) | 150 mg tablet (Rx) | Single dose |
| Ketoconazole (Nizoral®) | 200 mg tablet (Rx) | 2 tablets q.d. x5d |
| Itraconazole (Sporanox®) | 100 mg tablet (Rx) | 2 tablets q.d. x3d |

Abbreviations: mg = milligrams; d = day; q.d. = once daily; Rx = prescription.

## 1.1.1.5 Recurrent, Resistant and Non-Albicans VVC

Up to 20% of women will develop recurrent, resistant, or complicated VVC. In a study that compared a 6-month maintenance weekly fluconazole regimen to placebo in patients with recurrent VVC, the time to recurrence increased from 4.0 to 10.2 months, and the cure rate at 12 months doubled versus placebo from 22% to 43% (Sobel et al., 2004). However, fewer than half of patients remained disease-free after discontinuation of fluconazole which highlights the unmet medical need for these patients.

The prevalence of infection with non-albicans species, in particular *C. glabrata*, is increasing, especially in patients who are immunosuppressed and/or are diabetics; *C. glabrata* is poorly sensitive to current azole antifungal agents.

#### 1.2 VT-1161

VT-1161 is a novel oral antifungal agent with a lower affinity for heme-iron and a greater affinity for the fungal lanosterol 14  $\alpha$ -demethylase (CYP51) than the currently available azole drugs. As a result, VT-1161 more potently inhibits fungal CYP51 than current azoles and less potently inhibits host cytochrome P450 enzymes, resulting in greater cytochrome selectivity. These properties should translate to greater efficacy with an improved safety and tolerability profile.

VT-1161 is being developed for the treatment of patients with mucosal or superficial fungal infections. It is formulated with standard excipients known to be chemically stable when combined with VT-1161 into capsules for the investigational drug product.

A detailed description of the non-clinical binding and inhibition, metabolism, microbiology, toxicology, safety pharmacology, Phase 1 clinical studies in which 72 subjects were exposed to VT-1161 and Phase 2a proof-of-concept studies, in which 78 subjects were exposed to VT 1161 can be found in the VT-1161 Investigational Brochure. In the Phase 2b studies, 378 subjects were exposed to VT-1161. These studies are summarized below. The following sections provide data from non-clinical, Phase 1 and Phase 2 clinical trials supporting the use of VT-1161 for patients with recurrent vulvovaginal candidiasis (RVVC).

## 1.2.1 Non-Clinical Pharmacology

#### 1.2.1.1 Binding and Inhibition

*In vitro* pharmacology studies demonstrated that VT-1161 is a potent inhibitor of fungal CYP51 and binds more than 2200-fold more tightly to fungal CYP51 than to human CYP51. VT-1161 is also highly selective for fungal CYP51 versus key human cytochrome P450 enzymes, non-cytochrome metalloenzymes, and a broad panel of receptors, ion channels, and transporters.

#### 1.2.1.2 Metabolism

VT-1161 was not significantly metabolized when incubated with mouse, rat, dog or human hepatocytes. Only 1 possible metabolite consistent with hydroxylation and glucuronidation of VT-1161 was detected in dog hepatocytes. No additional metabolites were detected in any of the 4 species.

## 1.2.1.3 Microbiology

VT-1161 was tested against a broad range of Candida clinical isolates and showed potent activity (Table 3). It was also active against dermatophytes, including *Trichophyton rubrum*, *T. mentagrophytes*, and *T. tonsurans*.

T. tonsurans (N=5)

 $\leq 0.03 - 0.06$ 

Table 3. VT-1161 Antifungal MIC<sub>50</sub> or Range (μg/mL) Fungus (# of clinical isolates) VT-1161 Comparator C. albicans (N=10)  $\leq 0.03$ 

 $\leq 0.125$ C. glabrata (N=10) 0.25 Fluconazole C. parapsilosis (N=10) ≤0.03 0.125 0.125-0.25 C. guilliermondii (N=3) 2-8 T. mentagrophytes (N=12)0.25 0.06  $\leq 0.03$ *T. rubrum (N=41)* Itraconazole 0.03

0.06 - 0.5Abbreviations: C. = Candida; T. = Trichophyton; MIC<sub>50</sub> = minimum inhibitory concentration for 50% of isolates; μg = microgram; mL = milliliter; N = number (of clinical isolates).

In the Phase 2b RVVC study (VMT-VT-1161-CL-006), 413 clinical isolates were collected from subjects at screening visits until the end of the study. The minimum inhibitory concentration (MIC) ranges for VT-1161 and fluconazole for the isolates collected were;  $<0.0005 ->0.5 \mu g/ml$ and <0.06-32 µg/ml, respectively. The MIC<sub>50</sub> values for VT-1161 and fluconazole were 0.004 µg/ml and 0.125 µg/ml, respectively, and the MIC<sub>90</sub> values for VT-1161 and fluconazole were 0.06 μg/ml and 4 μg/ml, respectively. These data further demonstrated that VT-1161 has potent in vitro activity against the Candida strains obtained from clinical strains. For all tested isolates, the VT-1161 demonstrated MIC<sub>50</sub> and MIC<sub>90</sub> that were 5 dilutions lower than those demonstrated by fluconazole.

## 1.2.1.4 Activity in Animal Models of VVC

VT-1161 was evaluated as an oral treatment of vaginal candidiasis (C. albicans) in a murine model (Garvey et al., 2012). Three days after infection, VT-1161 was dosed orally once daily at 4, 10, or 25 mg/kg daily for 4 days. Fungal burden measured in vaginal lavage fluid was highly significantly suppressed (p <0.0002) compared to vehicle-treated controls at all doses and when measured 1 or 4 days after treatment ended. Plasma and vaginal tissue levels of the lowest dose of VT-1161 indicated that levels as low as 1 µg/mL resulted in this high degree of efficacy.

#### 1.2.1.5 Pharmacokinetics

VT-1161 formulated as a suspension in carboxymethylcellulose was well absorbed and exhibited approximately dose linear pharmacokinetics (PK) and a long plasma half-life in both rats and dogs. There was no evidence of an effect of gender on the PK of VT-1161 in either rats or dogs. VT-1161 accumulated during repeat-dosing in rats and dogs as expected based on the long half-life. VT-1161 was widely distributed into tissues and was mostly excreted in bile and feces in the rat. In vitro plasma protein binding of VT-1161 is high with approximately 99.5% binding to rat, dog and human plasma and slightly lower binding in mice (97.6%). The absolute oral

bioavailability of the capsule formulation used in Phase 1 studies administered to dogs was approximately 40% in the fasted state and approximately 100% when administered in the fed state.

## 1.2.1.6 General Toxicology

Oral VT-1161 was evaluated in general Good Laboratory Practice toxicity studies of up to 6 months and 9 months in duration in rats and dogs, respectively. Rats were more sensitive to the toxicological effects of oral administration of VT-1161 than dogs. The no observable adverse effect level (NOAEL) for the 6-month rat toxicity study was determined to be 0.5 mg/kg/day, based on an increase in incidence and severity of chronic progressive nephropathy, a rat-specific finding. The NOAEL for liver findings was 1.5 mg/kg, based on adverse findings at the high dose of 5 mg/kg/day including a minimal increase in serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) and an increase in frequency of minimal focal necrosis and single cell necrosis. Findings of liver hypertrophy, sub-capsular necrosis and multinucleated hepatocytes were considered rat-specific and associated with metabolic adaptation. Focal necrosis may be an exaggerated response to hepatocellular hypertrophy which is known to cause sub-capsular and single cell necrosis. The findings were reversible and similar to the findings observed in a prior 28-day study in the rat, providing support that the increased treatment duration in the 6-month rat study did not result in new findings of clinical concern. At the 1.5 mg/kg dose at steady state on Day 182, maximum plasma concentration (C<sub>max</sub>) was 4,055 ng/mL and area under the curve (AUC<sub>0-24</sub>) was 81,900 ng·h/mL. The NOAEL for the 9-month dog study was determined to be the high dose of 17 mg/kg/day (Day 273 C<sub>max</sub> was 74,700 ng/mL and AUC<sub>0-24</sub> was 1,675,000 ng·h/mL), as no adverse findings were identified. The NOAEL in the previous 28-day dog study was 10 mg/kg/day, based on decreased body weight and mild effects on lymphoid organs including increased 31 icromol body macrophages in the mandibular and mesenteric lymph nodes and in the Peyer's patches at 30 mg/kg and higher. These findings were largely reversed during the recovery period.

## 1.2.1.7 Genotoxicity

VT-1161 was found to be negative for genotoxicity in the Ames bacterial reverse mutation assay, the chromosome aberration assay in human peripheral lymphocytes and the *in vivo* bone marrow micronucleus assay in rats.

## 1.2.1.8 Reproductive Toxicology

VT-1161 at doses resulting in maternal toxicity (clinical signs and decrease in body weights) did not cause alterations in uterine and ovarian parameters in embryofetal development studies in rats and rabbits. Mean fetal body weights were slightly reduced in rabbits in the high dose group as a

direct result of maternal toxicity and decreased maternal body weights. No external, visceral and skeletal malformations and variations were observed at any of the dose levels evaluated. There were no effects on male or female fertility at clinically relevant doses.

## 1.2.1.9 Safety Pharmacology

The effects of VT-1161 on the neurological and pulmonary systems were evaluated in Sprague-Dawley rats. The data demonstrated that there were no VT-1161-related effects in either the neuropharmacological or pulmonary studies in rats given an oral dose of up to 1,000 mg/kg VT-1161, the highest dose tested.

Evaluation of cardiovascular function in telemetered dogs revealed no treatment-related changes in heart rate, blood pressure, cardiac rhythm or morphology, including the QT/QTc (Fridericia correction) interval, at oral doses up to 300 mg/kg, the highest dose tested.

## 1.2.1.10 In Vitro Cytochrome P450 Interactions

VT-1161 inhibited cytochrome P450 enzymes with the following potencies: CYP1A2 (half maximal inhibitory concentration [IC<sub>50</sub>]  $\geq$ 10  $\mu$ M), CYP2B6 (IC<sub>50</sub> = 4.0  $\mu$ M), CYP2C8 (IC<sub>50</sub> = 1.4  $\mu$ M), CYP2C9 (IC<sub>50</sub>  $\geq$ 10  $\mu$ M), CYP2C19 (IC<sub>50</sub> = 9.7  $\mu$ M), CYP2D6 (IC<sub>50</sub> = 9.4  $\mu$ M), and CYP3A4 (IC<sub>50</sub> = 9.6  $\mu$ M [testosterone], IC<sub>50</sub>  $\geq$ 10  $\mu$ M [midazolam]). Based on the high plasma protein binding of VT-1161, no clinically significant drug-drug interactions are expected.

#### 1.2.1.11 Effects of VT-1161 on Cardiac Repolarization

An in vitro human ether-à-go-go related gene study was conducted to assess the potential of VT-1161 to inhibit the repolarizing current of the cardiac action potential. VT-1161 inhibited the human ether-à-go-go related gene potassium current by 94.7  $\pm$  1.3% at 6  $\mu$ M. The IC<sub>50</sub> was calculated to be 1.9 µM (Hill coefficient = 2). However, a cardiovascular safety study in dogs showed that VT-1161 was well tolerated and did not induce any deleterious cardiovascular effects or affect QT intervals at test doses of up to 300 mg/kg, the highest dose tested, with exposures reaching  $24,000 \pm 6,881$  ng/mL at 30 hours post-dose.

#### 1.2.2 Clinical Studies

## 1.2.2.1 Phase 1 Studies

VT-1161 has been evaluated in 4 Phase 1 trials, a single ascending dose trial, a multiple ascending dose trial, a DDI study with midazolam as a sensitive substrate, and an ethnic PK study comparing Japanese and Western subjects. The primary objectives of these studies were to evaluate the safety and tolerability, PK and drug interaction potential of VT-1161 in healthy adult subjects. Detailed descriptions of the trials can be found in the VT-1161 Investigational Brochure.

#### 1.2.2.1.1 Single Dose-Escalation Study (Study VMT-VT-1161-CL-001)

Study VMT-VT-1161-CL-001 was a single-center, Phase 1, double-blind, randomized, placebo-controlled, dose-escalating study in healthy adult subjects. The study was designed to evaluate the safety, tolerability, and PK of single oral doses of VT-1161. Sixty-four subjects (43 males and 21 females) between 18 and 55 years of age were enrolled in 8 dose groups. Within each dose-group, 6 subjects received VT-1161 and 2 subjects received placebo. In the first 7 cohorts, escalating single oral doses (5, 10, 20, 40, 80, 160, and 320 mg) or matching placebo were administered in the fasted state. An 8<sup>th</sup> cohort received a single 320 mg oral dose of VT-1161 or matching placebo after ingesting a high-fat breakfast. Subjects in Cohorts 1 to 6 were followed for 14 days for safety and PK assessments. Visits on Days 28 and 42 were added for Cohorts 7 and 8. Dose escalation proceeded only after safety and PK of the previous dose was determined.

There were no deaths or serious adverse events (SAEs) reported. There were no treatmentemergent adverse events (TEAEs) that led to discontinuation from the study.

Overall, mean changes from baseline in safety parameters (hematology, chemistry, urinalysis, vital signs, and electrocardiogram [ECG]s) were generally small and were considered not clinically significant. None of the treatment-emergent physical examination abnormalities were of clinical significance. The maximum tolerated dose for the study was the highest dose administered, 320 mg, administered in the fed state.

Following oral administration of VT-1161 in the fasted state, median time to reach maximum plasma concentration (T<sub>max</sub>) ranged from 4 to 10 hours. Overall, C<sub>max</sub> increased slightly less than proportional to dose. The area under the plasma concentration versus time curve from time zero to infinity (AUC<sub>inf</sub>) values generally increased with increase in dose, ranging from an average of 16,145 ng•hr/mL at 20 mg to 241,971 ng•hr/mL at 320 mg. The mean half-life ranged from 393 to 1,467 hours. Administration of 320 mg VT-1161 with a standard high-fat meal resulted in higher plasma concentrations than those observed following 320 mg in the fasted state in a separate group of subjects. Average fasting C<sub>max</sub> was 338 ng/mL and this increased to 988 ng/mL in the fed state. AUC<sub>inf</sub> also increased from 241,971 ng•hr/mL when subjects were fasted to 953,119 ng•hr/mL with a high-fat meal.

## 1.2.2.1.2 Multiple Dose-Escalation Study (Study VMT-VT-1161-CL-002)

Study VMT-VT-1161-CL-002 was a Phase 1, single-center, randomized, double blind, placebo-controlled, multiple dose-escalating study in healthy adult subjects. The study was designed to evaluate the safety, tolerability, and PK of multiple oral doses of VT-1161. In addition to plasma PK, concentrations of VT-1161 in nails and skin were assessed. A total of 32 subjects participated in the study and received VT-1161 at 40, 80, 160 or 320 mg or placebo once daily for 7 days after ingestion of a high-fat meal. In each cohort of 8 subjects, 6 subjects received VT-1161, and 2 subjects received placebo. Subjects were followed for safety and PK assessments for 42 days after the last dose of study drug.

There were no deaths or SAEs reported. Most TEAEs were mild in intensity and no severe TEAEs were reported.

Mean changes from baseline in safety parameters (hematology, chemistry, coagulation, urinalysis, vital signs, and ECGs) were generally small and not considered clinically significant. There was no evidence of any clinically significant effect of VT-1161 on physical examinations in any dose group at any time point. The maximum tolerated dose for the study was the highest dose administered, 320 mg, administered once daily for 7 days in the fed state.

Following oral administration of VT-1161 in the fed state, median  $T_{max}$  values ranged from 4 to 6 hours after dosing. The increase in mean  $C_{max}$  was nearly proportional to dose over the 40 to 320 mg dose range. The concentrations were 3 to 4-fold higher on Day 7 than they were on Day 1, indicating accumulation during the 7-day dosing interval, with a mean  $C_{max}$  of 3,300 ng/mL on Day 7 at 320 mg. The area under the plasma concentration versus time curve over the dosing interval (AUC $\tau$ ) values on Day 7 also increased nearly proportionally to dose over the 40 to 320 mg dose range. The mean half-life ranged from 1,905 to 3,046 hours.

## 1.2.2.1.3 Drug-Drug Interaction Study (Study VMT-VT-1161-CL-007)

Study VMT-VT-1161-CL-007 was a Phase 1, single-center, open-label study in healthy adult subjects to evaluate the effect of single and multiple oral doses of VT-1161 when co-administered with single oral doses of midazolam (DDI cohort) and to evaluate the PK of a single oral dose of an alternate strength of VT-1161 alone (pharmacokinetic evaluation [PKE] cohort). All dosing was conducted 30 minutes after the start of a high-fat, high-calorie meal. A total of 36 subjects were enrolled in the study.

In the DDI cohort, 28 subjects were enrolled in a fixed-sequence design to receive a 2-mg oral dose of midazolam on Day 1, followed by 14 daily 600 mg oral doses of VT-1161 (4 x 150 mg
tablets) on Day 3 through Day 16 with single 2 mg oral doses of midazolam on Day 3 and Day 16. Subjects were followed for safety, tolerability and PK assessments through Day 17, 1 day after the last dose of study drug. Twenty-four subjects in the DDI cohort completed the study and 4 subjects withdrew from the study prior to completion; 2 subjects voluntarily withdrew consent and 2 subjects withdrew due to an AE (discussed in more detail below).

There were no deaths reported in the study. One SAE (acute psychosis) was reported in a subject in the DDI cohort on Day 11 of the study, leading to discontinuation. The Investigator determined the subject likely had a pre-existing psychiatric condition based on patient report and assessed causality as unlikely-related to VT-1161. One additional subject in the DDI cohort withdrew from the study due to an AE of abnormal ECG on Day 3 of the study. The AE occurred prior to the first dose of VT-1161; the Investigator assessed causality as unrelated to study drug. Otherwise, mean changes from baseline in safety parameters (hematology, chemistry, coagulation, urinalysis, vital signs, and ECGs) in both the DDI and PKE cohorts were generally small and not considered clinically significant and there was no evidence of any clinically significant effect of VT-1161 on physical examinations in either cohort.

In the DDI cohort, midazolam mean plasma C<sub>max</sub> increased 30% and AUC<sub>inf</sub> decreased 15% on Day 3 (after the first dose of VT-1161) relative to Day 1 (midazolam alone). Midazolam mean plasma C<sub>max</sub> decreased 3% and AUC<sub>inf</sub> decreased 37% on Day 16 (after 14 daily doses of VT-1161) relative to Day 1 (midazolam alone).

In the PKE cohort, 8 subjects were enrolled to receive a single 600 mg oral dose of VT-1161 (2 x 300 mg tablets) on Day 1. Subjects in the PKE cohort were followed for safety, tolerability and PK assessments through Day 2, 1 day after the dose of study drug. All 8 subjects in the PKE cohort completed the study. VT-1161 mean plasma C<sub>max</sub> and AUC<sub>0-24</sub> values after a single oral administration of 600 mg VT-1161 (2 x 300 mg) on Day 1 were 1,946 ng/mL and 28,070 ng•hr/mL, respectively. These values are similar to VT-1161 mean plasma C<sub>max</sub> and AUC<sub>0-24</sub> values after a single oral administration of 600 mg VT-1161 (4 x 150 mg) in the DDI cohort (1,994 ng/mL and 25,330 ng•hr/mL, respectively), indicating the comparative bioavailability of the 2 strengths of tablets is similar.

### 1.2.2.1.4 Japanese Bridging Study (Study VMT-VT-1161-CL-008)

Study VMT-VT-1161-CL-008 was a single-center, open-label study in healthy adult Japanese and Western subjects. The objective of this ethno-bridging study was to evaluate the safety, tolerability, and PK of VT-1161 in these 2 ethnic populations after subjects received 14 once daily

oral doses of VT-1161 administered in the fed state. There was a total of 51 subjects enrolled. In the 300-mg dosage-group, there were 13 Japanese and 14 Western subjects. In the 600 mg dosage group, there were 12 Japanese and 12 Western subjects. The mean age of subjects was 36.5 years, ranging from 19 to 55 years across treatment groups. The subjects were evenly divided by sex across all groups and the race of the Western subjects was evenly divided by white and black.

The study drug was overall well tolerated by both Western and Japanese subjects. There were no significant differences between the 2 populations in any of the safety assessments. A slight increase in AEs was seen in the 600 mg dosage group as compared with the 300 mg dosage group, but no SAEs were observed. Only 1 subject was withdrawn from the study for an AE of rash (subject request), which was categorized as an unlikely-related TEAE. There was 1 pregnancy in a subject who was non-compliant with contraception requirements, which was electively terminated by the subject.

Of the 51 subjects enrolled in the study, 11 Japanese subjects from both dose groups and 12 Western subjects from both dose groups were included in the full PK analysis population. Trough concentrations on Days 1 through 14 rose each day; thus, steady-state conditions had not been met by Day 14. Larger differences between the 2 ethnic groups were seen in C<sub>max</sub> and AUC<sub>0-72</sub> following the 300 mg dose compared with the 600 mg dose. At the 300 mg dose, C<sub>max</sub> and AUC<sub>0-72</sub> were approximately 40% higher in Japanese subjects compared with Western subjects. At the 600-mg dose, C<sub>max</sub> and AUC<sub>0-72</sub> were approximately 10% higher in Japanese subjects compared with Western subjects. However, median T<sub>max</sub> was similar across doses at 4 hours for Japanese subjects at both the 300 mg and 600 mg dosages and 6 hours for Western subjects at both the 300 mg and 600 mg dosages. The terminal elimination phase was very flat and half-life exceeded 1800 hours. Total clearance following the 300-mg dose was 1.642 L/hr for the Japanese subjects compared with 2.332 L/hr for the Western subjects. Following the 600 mg dose, clearance was similar for the Japanese and Western subjects (2.000 and 2.086 L/hr, respectively).

### 1.2.2.2 Phase 2 Studies

### 1.2.2.2.1 Dose Ranging Study in Tinea Pedis (Study VMT-VT-1161-CL-003)

VMT-VT-1161-CL-003 was a Phase 2a, randomized, double-blind, dose-ranging study to evaluate the efficacy and safety of VT-1161 over-encapsulated tablets compared to placebo in the treatment of subjects with moderate to severe interdigital tinea pedis. A total of 50 subjects participated in the study across 4 dose groups: 1) VT-1161 200 mg once daily for 4 days, followed by 50 mg once daily for 10 days (low dose); 2) VT-1161 600 mg once daily for 4 days, followed by 150 mg once

daily for 10 days (mid-dose); 3) 600 mg twice daily for 4 days, followed by 300 mg once daily for 10 days (high dose; or 4) placebo matching the VT-1161 treatment regimen. VT-1161 plasma concentrations increased with dose and were as high as 6,230 ng/mL on Day 14 in the 600 mg twice daily/300 mg once daily dose group. Subjects were enrolled into the high-dose cohort following an interim analysis that included safety data generated through the test of cure (TOC) visit (Day 42) of the 2 lower dose groups.

VT-1161 was safe and well tolerated at all dose levels through 6 months of follow up. No SAEs were reported. Most AEs reported were mild to moderate in severity and considered unrelated to study drug. A single VT-1161 treatment related AE was reported (rash) that was considered by the Investigator to be "possibly related." The subject discontinued treatment after the first dose, and the rash completely resolved by the following day. There were no clinically significant treatment-emergent changes in vital signs, physical findings, ECGs, or laboratory parameters. One subject experienced a significant elevation of creatine kinase (CK) along with a slight increase in ALT and AST that was associated with a rigorous exercise program. These changes were considered unrelated to treatment and all enzyme levels returned to normal at a subsequent follow-up visit.

At the Day 42 TOC visit, 42%, 42%, 50% and 0% of subjects receiving low dose, mid-dose or high dose VT-1161 or placebo were determined to have achieved effective therapeutic cure (defined as having a total severity score of  $\leq$ 2 with no individual severity score of  $\geq$ 1, and also, having negative mycology [culture and KOH]) in the intent-to-treat (ITT) population.

# 1.2.2.2.2 Dose Ranging Study in Acute Vulvovaginal Candidiasis (Study VMT-VT-1161-CL-004)

VMT-VT-1161-CL-004 was a randomized Phase 2a, double-blind, dose ranging study to evaluate the efficacy and safety of VT-1161 over-encapsulated tablets compared to fluconazole in the treatment of 55 subjects with moderate to severe acute VVC. A total of 55 subjects with moderate-to-severe acute VVC (severity score ≥6 and a positive fungal KOH test) participated in the study across 4 dose groups: 1) VT 1161 300 mg once daily for 3 days, 2) 600 mg once daily for 3 days, 3) 600 mg twice daily for 3 days, or 4) a single dose of fluconazole 150 mg followed by matching placebo. Subjects were enrolled into the high-dose cohort following an interim analysis that included safety data generated through the TOC visit (Day 28) of the 2 lower dose groups. An additional interim analysis was conducted when the high-dose subjects had completed their TOC visit.

VT-1161 was determined to be safe and well tolerated at all dose levels through Day 28. No SAEs were reported and no subjects discontinued because of an AE. Most AEs reported were considered unrelated to study drug and were mild in severity. There were few treatment-related TEAEs of clinical concern. Most TEAEs were reported in the low- and mid-dose cohorts and only 1 TEAE (insomnia) was noted in the high-dose cohort. One subject developed urticaria that was considered possibly related to study drug and which resolved with prednisone. There were no clinically significant treatment-emergent changes in vital signs, physical findings, ECGs or laboratory parameters.

The efficacy of VT-1161 in the treatment of moderate-to-severe acute VVC was evaluated at the TOC visit in the ITT population (defined as all randomized subjects receiving at least 1 dose of study drug) and the per protocol (PP) population (defined as subjects that were compliant with all key aspects of the protocol). Subjects in the ITT population were randomized into the VT-1161 300 mg once daily for 3 days (n = 14), VT-1161 600 mg once daily for 3 days (n = 12), VT-1161 600 mg twice daily for 3 days (n = 14) or fluconazole (n = 15). Effective clinical cure rate (defined as having a total severity score of 0 or 1 and a negative culture) were 29%, 83%, 86% and 73%, respectively. Subjects in the PP population achieved effective therapeutic cure at a rate of approximately 87%, 86%, 86% and 75%, respectively, in the low-dose, mid-dose, or high-dose VT-1161 or fluconazole groups at the Day 28 TOC visit.

# 1.2.2.2.3 Phase 2b Study in Subjects with Distal and Lateral Subungual Onychomycosis of the Toenail (VMT-VT-1161-CL-005)

In this Phase 2b study, the safety, tolerability, PK and efficacy of VT-1161 in subjects with distal and lateral subungual onychomycosis of the toenail were evaluated. A total of 259 subjects participated in the study in 5 treatment groups and were administered either:

- Low dose 12-week: Loading doses of 300 mg once daily for 2 weeks, then 300 mg once weekly for 10 weeks, followed by placebo for 12 weeks.
- Low dose 24-week: Loading doses of 300 mg once daily for 2 weeks, then 300 mg once weekly for 22 weeks.
- High dose 12-week: Loading doses of 600 mg once daily for 2 weeks, then 600 mg once weekly for 10 weeks, followed by placebo for 12 weeks.
- High dose 24-week: Loading doses of 600 mg once daily for 2 weeks, then 600 mg once weekly for 22 weeks.

## · Matching placebo

Subjects in all cohorts were followed for 60 weeks. Consenting subjects were enrolled into an extension study to assess the long-term safety and PK of VT-1161 through Week 96.

The incidence of adverse events (AEs) was balanced across the VT-1161 treatment arms and placebo. A total of 148 subjects (57%) had at least 1 TEAE, and the frequency was within the range of 49% to 67% for all treatment groups. The majority of TEAEs were considered by the Investigator to be mild or moderate and unrelated to study drug. Most TEAEs were transient and occurred during the first 12 weeks of treatment for all treatment groups, including placebo. Nineteen subjects reported related TEAEs through Week 60. Sixteen subjects were on VT-1161 and three subjects were on placebo. The only related TEAE reported by more than 2 subjects was nausea. Eleven subjects reported a total of 16 SAEs, which were considered unrelated to study drug.

The incidence of study drug related TEAEs was within the range of 6% to 11% for all treatment groups, with the highest frequency in the 600 mg 24-week group. The most common (≥2 total subjects) TEAEs that were considered related to VT-1161 were nausea, dysgeusia, dizziness, constipation, and decreased appetite. The most common TEAE that was considered related to placebo was dizziness.

The incidence of TEAEs leading to study drug discontinuation was low, in the range of 0% to 6% for all treatment groups.

There were no clinically-relevant findings noted by the Investigators with vital signs, physical exam findings or ECGs.

There was no obvious clinically-relevant effect of VT-1161 on chemistry, hematology or urinalysis parameters.

Overall, VT-1161 was safe and well-tolerated at all doses and treatment durations including the highest dose and longest duration evaluated of 600 mg 24-week treatment group. The TEAEs were typical of the subject population being studied and were generally balanced across the VT-1161 treatment and placebo group.

The primary efficacy endpoint was complete cure at Week 48. The proportion of subjects in the ITT population with complete cure at Week 48 ranged from 32% to 42% in the VT-1161 treatment groups, with the lowest rate in the 300 mg 12—week treatment group and the highest rate in the

600 mg 12—week treatment group. No subjects receiving placebo experienced complete cure at Week 48. The proportion of ITT subjects with complete cure was statistically significantly higher for all VT-1161 treatment groups compared with placebo at Week 48 (p<0.001).

Overall, the efficacy at Week 48 was clearly demonstrated in all the VT-1161 treatment groups, with little to no improvement seen in the placebo group.

### 1.2.2.2.4 Phase 2b Study in Subjects with Recurrent Vulvovaginal Candidiasis

In this Phase 2b study, the safety, tolerability, PK and efficacy of VT-1161 in subjects with recurrent vulvovaginal candidiasis was evaluated. A total of 215 subjects participated in the study, were randomized to 5 treatment groups and were administered either:

- Low dose 12-week: Loading doses of 150 mg once daily for 7 days, then 150 mg once weekly for 11 weeks, followed by placebo for 12 weeks.
- Low dose 24-week: Loading doses of 150 mg once daily for 7 days, then 150 mg once weekly for 23 weeks.
- High dose 12-week: Loading doses of 300 mg once daily for 7 days, then 300 mg once weekly for 11 weeks, followed by placebo for 12 weeks.
- High dose 24-week: Loading doses of 300 mg once daily for 7 days, then 300 mg once weekly for 23 weeks.
- Matching placebo

In general, the incidence of AEs was balanced across the VT-1161 treatment arms and placebo. Two subjects discontinued VT-1161 because of a TEAE. Of these two, only one TEAE was considered related to VT-1161 by the study investigator. Most TEAEs were considered unrelated to study drug and were mild or moderate in severity. Six SAEs were reported through Week 48 of the study, none of which were considered related to study drug by the investigator. Interestingly, a higher incidence of bacterial vaginosis and urinary tract infections was reported in the placebo arm.

There were no clinically-relevant findings noted by the investigators regarding vital signs, physical exam findings or ECGs. There was no obvious clinically-relevant effect of VT-1161 on chemistry, hematology or urinallysis parameters.

The primary efficacy outcome measure was the proportion of subjects with one or more culture-verified acute VVC episodes during the Maintenance Phase through Week 48 of the study in the ITT population. Culture-verified acute VVC was defined as a positive fungal culture for Candida species associated with a clinical signs and symptoms score of  $\geq 3$ . The proportion of subjects with one or more culture-verified acute VVC episode through Week 48 was lower in VT-1161 dosing regimens: 4.8% in 150 mg 12 weeks, 7.0% in 150 mg 24 weeks, 0.0% in 300 mg 12 weeks, and 4.9% in 300 mg 24 weeks, treatment groups compared with 52.2% in the placebo group. The difference was statistically significant in the VT-1161 dosing regimens compared with placebo (p<0.0001).

In conclusion, VT-1161 was determined to be efficacious, safe and well tolerated at all dose levels through the final visit at Week 48 of the study.

### 1.3 Study Rationale

RVVC can be treated with topical and/or oral agents and patients may receive maintenance treatment for up to 6 months or longer once the acute infection has resolved. For most patients, available agents do not provide the desired delay to recurrence of an acute VVC episode, underlining the need for more effective treatments for RVVC. Fluconazole has been used to treat acute VVC episodes in patients with recurrent disease. However, fluconazole has relatively lesser activity against some non-albicans species that are more common in patients with complicated VVC.

While oral antifungal agents offer better efficacy, they suffer from safety issues associated with their narrow therapeutic windows and off target toxicity. Several properties of VT-1161 suggest that it has the potential to be a best-in-class oral agent for the treatment of RVVC, including its ability to effectively inhibit growth of causative fungal pathogens at achievable plasma levels. The in vitro potency against Candida species is greater than fluconazole. Also, because it is much more selective for fungal CYP51 and CYP metabolizing enzymes than currently used oral agents, the probability of both hepatotoxicity and DDIs should be significantly reduced. Its PK profile and extended half-life should also limit recurrence of VVC. A weekly dosing regimen after the loading dose may improve patient compliance.

### 1.3.1 Rationale for Induction Phase Treatment

Fluconazole is an approved treatment for acute VVC and is used off-label to treat patients with recurrent disease. The proposed dose regimen of 3 doses of fluconazole taken 72 hours apart corresponds to a regimen that is often used as the standard of care and has been regularly employed

during the induction phase of similar clinical studies designed to study RVVC. Treatment of the acute infection with fluconazole in the Induction Phase allows for a more controlled assessment of recurrence in the VT-1161 treatment group versus placebo.

### 1.3.2 Dosing Regimen for VT-1161 and Matching Placebo

Following cure of the acute infection by 3 doses of fluconazole every 72 hours, subjects will be randomly assigned to receive one of the following treatment groups:

- VT-1161: Loading dose of 150 mg once daily for 7 days, then 150 mg once weekly for 11 weeks.
- Placebo: Matching VT-1161 capsules.

The rationale for dose selection is provided in Section 4.4, Design Justification.

### 1.4 Potential Risks and Benefits of Participating in the Study

The Phase 1, Phase 2a, and Phase 2b studies with VT-1161 incorporated monitoring for AEs often reported with other azole antifungal drugs. No clinically significant study drug related AEs were observed in clinical studies with VT-1161, suggesting that it may be better tolerated than commonly used azole agents.

# **2 OBJECTIVES**

# Primary:

• To evaluate the efficacy of oral VT-1161 in the treatment of RVVC through Week 48.

# Secondary:

- To evaluate the safety and tolerability of oral VT-1161 in the treatment of RVVC through Week 48.
- To evaluate the impact of oral VT-1161 treatment on patient reported outcomes through Week 48.

### 3 STUDY ENDPOINTS

The primary efficacy outcome measure is the proportion of subjects with one or more culture-verified acute VVC episodes during the Maintenance Phase in the ITT population. The Maintenance Phase is defined as post randomization through Week 48 of the study. An acute VVC episode during the Maintenance Phase (considered a recurrent episode) is defined as a positive culture for Candida species and a clinical signs and symptoms score of  $\geq 3$ .

### Secondary:

- Time to first recurrence of a culture-verified acute VVC episode with signs and symptoms score ≥3 during the Maintenance Phase.
- The proportion of subjects with at least one positive culture for Candida during the Maintenance Phase.
- The proportion of subjects with at least one culture-verified acute VVC episode with signs and symptoms ≥3 post randomization through Week 24.
- Change from Screening through Week 48 in the SF-36 mental component score (MCS).
- Change from Screening through Week 48 in the SF-36 patient reported outcome survey total score.

Product: VT-1161 IND 111675 Ver. 6 U.S. Only, 01 October 2019

### **STUDY DESIGN**

### **Overall Study Design**

This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled, parallel-group study. The study is designed to evaluate the efficacy and safety of oral VT-1161 capsules in the treatment of subjects with RVVC. The impact of oral VT-1161 treatment on the quality of life will also be evaluated using data collected from patient reported outcome assessments.

Subjects must have a history of RVVC, defined as at least 3 episodes of acute VVC in the past 12 months, as described below:

- Subjects must have an acute VVC episode at the time of Screening, with a documented positive KOH or Gram stain performed at the investigative site
- Subjects must also have had 2 or more additional episodes of acute VVC in the past 12 months, with at least 1 of the episodes documented by a positive confirmatory laboratory test (i.e., culture, PCR, Affirm test, KOH test, Gram stain, a documented Pap test, or other approved diagnostic test)

The study consists of two Phases: 1) an open-label Induction Phase for the treatment of the acute VVC infection with 3 sequential 150 mg oral doses (every 72 hours) of fluconazole, and 2) a Maintenance Phase in which subjects will be randomly assigned to receive VT-1161 or placebo for 7 daily doses followed by 11 weekly doses and then enter a 36-week follow-up period.

Once subjects have provided informed consent or assent (for those ages 12 to 17), the investigational site will evaluate all subjects by completing a review of pertinent medical history, obtaining vital signs, weight and height, ECG and laboratory tests, reviewing clinical signs and symptoms of vulvovaginitis, performing a complete physical examination including speculum examination of the vagina, performing a KOH wet mount test or Gram stain from a vaginal smear to confirm the presence of yeast, and collecting vaginal swabs to establish a baseline culture for identification of fungal species. Patient reported outcome surveys (SF-36, EQ-5D-3L or EQ-5D-Y [for ages 12 to 17], WPAI:SHP, PHQ-9) for all regions and questions regarding their RVVC history (US only) will also be administered. Eligible subjects will have a composite vulvovaginal signs and symptom score of  $\geq 3$  as outlined in Section 9.1.7, a positive local KOH or Gram stain that confirmed the presence of yeast, and must meet other initial entry criteria.

Once eligibility is confirmed, subjects will enter the Induction Phase. During the Induction Phase, the presenting acute VVC infection will be treated with 3 sequential 150 mg oral doses (every 72 hours) of fluconazole. Subjects will return approximately 14 days after the first dose of fluconazole for evaluation and, if the acute VVC infection has resolved (defined by a signs and symptoms score of <3), they will be randomized in a 2:1 ratio to receive either VT-1161 or a matching placebo regimen. Day 1 (Baseline) is defined as the first day of investigational medicinal product (IMP) administration and subsequent study days are defined by the number of consecutive days thereafter. If the acute VVC has not resolved (defined by a signs and symptoms score of  $\ge 3$ ), the subject will be considered a screen failure and encouraged to see their physician for further evaluation and follow-up care.

### 4.2 Treatment Arms and Duration of Study

Subjects will be randomized in a 2:1 ratio to receive VT-1161 or placebo.

The duration of individual subject participation will be approximately 50 weeks: including the 2-week Induction Phase with fluconazole administration, followed by 12 weeks for IMP administration, and 36 weeks of follow-up. Assessments and procedures will be performed as outlined in Table 1. Schedule of Assessments and Procedures. Subjects who return to the clinic for a recurrent VVC episode should be evaluated as per the unscheduled visit noted in the Schedule of Assessment and Procedures.

The planned study duration is 26 months from Screening of the first subject until the last follow-up of the last subject.

### 4.3 Number of Subjects

Approximately 600 screened and 300 randomized subjects are planned for this study. Assuming a 20% discontinuation rate for the remainder of the study, approximately 240 subjects are expected to complete the study.

Subjects will be enrolled at 60 to 80 sites in North America and Europe.

### 4.4 Design Justification

The VT-1161 dose and duration selection in the planned Phase 3 studies is based primarily on the results of VMT-VT-1161-CL-006; "A Phase 2, Randomized, Double Blind, Placebo-Controlled, Dose Ranging Study to Evaluate the Efficacy and Safety of VT-1161 Oral Tablets in the Treatment of Patients with Recurrent Vulvovaginal Candidiasis." The study was designed to be consistent with the principles put forth in the ICH E4 Guideline, "Dose-Response Information to Support Drug Registration."

Given VT-1161's large therapeutic window and favorable safety profile as demonstrated in the single- and multiple-ascending dose Phase 1 studies as well as Phase 2a studies, the Phase 2b RVVC study was designed to demonstrate prolonged remission following short courses of VT-1161 dosing.

The proportion of subjects in the ITT population with one or more culture verified acute VVC episodes through Week 48 was lower in the VT 1161 dose groups; 4.8% in the 150 mg/12-week, 7.1% in the 150 mg/24-week, 0.0% in the 300 mg/12-week, and 4.9% in the 300 mg/24-week treatment groups, compared to 52.2% in the placebo group. This difference was statistically significant in all VT-1161 groups compared to placebo (p<0.0001). However, the study was not designed to demonstrate a statistical difference between the VT-1161 dosing regimens.

In the PP population, the proportion of subjects with one or more culture-verified acute VVC episodes through Week 48 in VT-1161 dose groups were 3.3% in the 150 mg/12-week, 10.7% in the 150 mg/24-week, 0.0% in the 300 mg/12-week, and 0.0% in the 300 mg/24-week treatment groups, compared to 65.6% in the placebo group, indicating a numerically higher rate of recurrence in the lower VT-1161 dose groups. A similar trend was observed in subjects with one or more positive cultures through Week 48; 13.3% in the 150 mg/12-week; 25.0% in the 150 mg/24-week; 16.1% in the 300 mg/12-week; and 3.2% in the 300 mg/24-week treatment groups, compared to 84% in the placebo group. The mean plasma concentrations for the VT-1161 150 mg/12-week treatment group was 1.3  $\mu$ g/mL at the start of weekly dosing (Day 7), 2.6  $\mu$ g/mL at the end of the dosing phase (Week 12), and was followed by a slow decay to reach 0.75  $\mu$ g/mL at Week 48. Based on the PP analysis, it appears that the 150 mg/12-week treatment group is at or near a minimally effective dose and duration of therapy.

In the Kaplan-Meier analysis (ITT population), most recurrent episodes occurred in the early phase of the study. In total, 7 subjects across all the VT-1161 dose groups exhibited a culture-verified recurrence while on study with 5 of 7 subjects having a recurrence in the first 5 weeks of the study. Notably, 3 of these 5 subjects (all in the 150 mg group) experienced a recurrence by Day 7. Taken together, the data suggest that these subjects in the VT-1161 low dose (150 mg) treatment groups may have not attained effective therapeutic drug levels early enough to prevent the early recurrences. Therefore, a lower than 150 mg VT-1161 starting dose cannot be justified given the potential that more patients would experience recurrence, especially for less susceptible non-albicans strains.

The dose selection for the Phase 3 study is further supported by the safety and tolerability profile of VT-1161. The frequency of AEs across all VT-1161 treatment groups in the Phase 2b study

Protocol VMT-VT-1161-CL-012

was similar to the placebo group. There were also no meaningful differences observed between placebo and the VT-1161 treatment groups in other safety parameters including chemistry, hematology and ECG analyses. To that end, from a safety perspective any of the dosing groups tested in the Phase 2b study could be potentially selected for the Phase 3 studies. This is important since, in addition to exhibiting excellent safety and tolerability, all VT-1161 treatment groups also achieved clinical outcomes that were far superior to fluconazole historic data where approximately 60% of RVVC patients experienced one or more acute culture-verified VVC recurrences within 6 months after the cessation of weekly prophylactic/maintenance therapy. (Sobel et al. 2004).

The proposed dosing regimen for the Phase 3 studies, incorporates a 7-day 150 mg loading dose phase to minimize early breakthroughs, followed by a 150 mg once weekly maintenance dose phase for 11 weeks. Based on the PK results from the Phase 2b study, the proposed dosing regimen of 150 mg daily for 7 days followed by a 150 mg once weekly maintenance dose is expected to provide a mean plasma concentration of approximately 2.5  $\mu$ g/mL at the end of the dosing period (Week 12).

### 4.4.1 Justification for Inclusion of Adolescents in the Study

Vulvovaginal candidiasis, and especially RVVC, is rare in pre-menarcheal girls (typically pre-adolescents less than 12 years of age) and epidemiological data is generally lacking for this population.

Adolescent females (ages 12 to 17 years, inclusive) represent a menarcheal population that is newly influenced by reproductive hormones. The changes in reproductive hormones in adolescents cause vast changes in tissues and may increase the susceptibility to VVC. In this population, cases of VVC and RVVC exist but are substantially less common than in adult females. While 75% of healthy women will likely experience one episode of VVC in their lifetime, and potentially 9% will be characterized as having recurrent disease, the prevalence of symptomatic acute VVC in adolescents is less than 2% of the population and there is no published data that addresses the incidence of RVVC in this patient population (Fidel, 2002; Blostein, 2017; Barousse, 2004). Presenting symptoms of VVC in menarcheal adolescents are similar to those in the adult population, and treatment typically consists of topical antifungal preparations while oral antifungal agents are prescribed only in severe or complicated cases (Joishy, 2005). The dose and administration of the agents used in adolescents are the same as those used in adult females with VVC and RVVC.

The United States FDA Draft Guidance *Vulvovaginal Candidiasis: Developing Drugs for Treatment* states that while uncomplicated VVC is unlikely to occur in healthy pre-menarcheal girls, post-menarcheal adolescent girls with VVC should be included in Phase 3 trials. Accordingly, the present study will follow guidance received by the United States FDA reviewers and will allow enrollment of subjects 12 to 17 years of age (inclusive) to collect as much information as possible on the treatment of the adolescent population with RVVC.

In Hungary, Romania, Ukraine, and Czech Republic, only subjects 18 years of age or older will be enrolled in the study.

#### 5 SELECTION OF STUDY POPULATION

The following criteria for enrollment must be followed explicitly. A subject will not be enrolled unless the following inclusion/exclusion criteria are met. The Investigator or other study site personnel must record in the source documents (e.g., the site's chart) and case report form (CRF) that the informed consent document (or assent for those 12-17) was signed and dated prior to any study procedures. The presence of inclusion criteria and absence of exclusion criteria will be verified by the Investigator in the subject's clinic chart.

### 5.1 Inclusion Criteria

- 1. Subjects must be generally healthy, post-menarchal, non-pregnant females 12 years of age and older as of Screening. In Hungary, Romania, Ukraine, and Czech Republic only, subjects must be generally healthy, post-menarchal, non-pregnant females 18 years of age and older as of Screening.
- 2. Subjects must have a history of recurrent VVC as defined by three (3) or more patient reported and/or laboratory confirmed episodes of acute VVC in the past 12 months including the episode confirmed at Screening, with at least one episode (not including the current episode) documented by a positive culture, PCR, Affirm test, KOH test, Gram stain, or a documented Pap test in the prior 12 months revealing filamentous hyphae/pseudohyphae and/or budding yeast cells, or other approved diagnostic tests.
- 3. Subjects must have an acute VVC infection at Screening, defined as:
  - a. a total signs and symptoms score of  $\geq 3$  and
  - b. a positive KOH wet mount preparation or Gram stain from a vaginal smear revealing filamentous hyphae/pseudohyphae and/or budding yeast cells.
- 4. Subjects must have a composite vulvovaginal signs and symptoms score of <3 at the Baseline (Day 1) Visit.
- 5. Subjects must have a documented Pap test at Screening or within the timeline per current standard of care guidelines for the appropriate age requirement. Results must be either "negative for intraepithelial lesion or malignancy" or "ASCUS-atypical squamous cells of undetermined significance" (not applicable to subjects with a history of total hysterectomy).
- 6. Subjects must be suitable candidates for oral therapy and be able to swallow capsules intact.
- 7. Subjects must be willing and able to provide written informed consent or assent (for those ages 12 to 17) and authorization for use of protected health information.

- 8. Subjects must be willing and able to comply with protocol requirements, instructions, and protocol-stated restrictions and be likely to complete the study as planned.
- 9. Subjects of non-childbearing potential must meet the requirements defined below:
  - a. Pre-menopausal with documentation of surgical sterilization (i.e., hysterectomy, bilateral tubal ligation, bilateral oophorectomy, or bilateral salpingectomy) at least 3 months prior to Screening.
  - b. Post-menopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments at Screening.
- 10. Subjects of childbearing potential (includes ages 12 to 17) must use 1 of the following methods of contraception during the study through Week 48:

**OPTION 1** – Highly effective methods that can be used alone:

- i. Copper intrauterine device
- ii. Levonorgestrel-releasing intrauterine system
- iii. Progestin implant
- iv. Monogamous with a vasectomized male partner
- v. Abstinence<sup>a</sup>

**OPTION 2** – Acceptable first and second barrier methods to be used in combination:

FIRST (Hormonal Contraception)<sup>b</sup>

- 1. Estrogen & progestin oral contraceptives, transdermal patch or vaginal ring.
- 2. Progestin only oral contraceptives or injection

SECOND (Barrier Method)

- 1. Diaphragm (with spermicide)
- 2. Cervical cap (with spermicide)
- 3. Male condom (with or without spermicide)

In addition to OPTIONS 1 and 2, subjects of childbearing potential (includes ages 12-17) may also use 1 of the following methods of contraception after completing the Induction Phase on Study Day 1 through Week 48:

**OPTION 3 (Day 1 – Week 48)**<sup>c</sup> – Acceptable first and second barrier methods to be used in combination:

FIRST (Barrier Method)

1. Diaphragm (with spermicide)

# 2. Cervical cap (with spermicide)

### SECOND (Barrier Method)

1. Male condom (with or without spermicide)

- <sup>a</sup> Sexual abstinence is defined as refraining from heterosexual intercourse during the entire study period and where this is the usual life style of the subject. Periodic abstinence (calendar, symptothermal, postovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not considered to be acceptable methods of contraception.
- <sup>b</sup> Subjects who started taking a hormonal contraceptive less than 3 months prior to the first dose of fluconazole must agree to use a double-barrier method (i.e. diaphragm plus spermicide or condom) through 3 months after starting the hormonal contraceptive.
- <sup>c</sup> Because of the teratogenic risk associated with repeat dosing of fluconazole, OPTION 3 contraceptive methods cannot be used during Screening and the Induction Phase of the study [from Screening (Day 1) until Day 14 of the study].

### 5.2 Exclusion Criteria

- 1. Subjects must not have the presence of concomitant vulvovaginitis caused by other pathogens (e.g., bacterial vaginosis, *Trichomonas vaginalis*, *Chlamydia trachomatis*, or *Neisseria gonorrhoeae*) at Screening visit and at the Day 1 visit if an infection is suspected.
- 2. Subjects must not have an active HPV infection as evidenced by visible condylomas on vulvovaginal examination at Screening and Day 1 visits.
- 3. Subjects must not have the presence or a history of another vaginal or vulvar condition(s) that in the Investigator's opinion would confound the interpretation of clinical response.
- 4. Subjects must not have a history of cervical cancer.
- 5. Subjects must not use any systemic (e.g., oral or injectable) corticosteroid therapy during the study or within 30 days prior to Screening, nor use of topical vulvar or vaginal steroids during the study or within 7 days prior to Screening. However, use of topical (no vulvar or vaginal steroids), inhaled, ophthalmic, collunarium/nasal, intraarticular and intralesional steroids is permitted.
- 6. Subjects must not use any systemic (e.g., oral or injectable) or topical (applied to the vulva or vaginal area) antifungal, antibacterial, or antitrichomonal drugs or vaginal douches during the study (unless prescribed by the Investigator) or within 7 days prior to Screening.

- 7. Subjects must not be using drugs with a narrow therapeutic index that are metabolized by CYP3A4 and sensitive to induction of CYP3A4 during the study (carbamazepine, cyclosporine, fentanyl, quinidine, sirolimus and tacrolimus).
- 8. Subjects must not use any vaginal estrogen replacement therapy, ospemifene, Vitamin E gel capsules (vaginally) or lubricants within 7 days prior to Screening.
- 9. Subjects must not have a condition that would require treatment during the study with concomitant topical (applied to vulva and vagina) or systemic antimicrobial therapy for any reason.
- 10. Subjects must not have received an immunosuppressive medication (e.g. cyclosporine, tacrolimus, methotrexate, 6 mercaptopurine, mycophenolate, etc.), or radiation therapy within 3 months prior to Screening or have a medical condition where it would be likely that the subject may need to use these therapies during the study.
- 11. Subjects must not have evidence of any clinically significant major organ disease or current clinically significant infection or any other conditions (with the exception of acute VVC) that may affect the clinical assessment of RVVC per Investigator judgment.
- 12. Subjects must not have any comorbid condition that in the opinion of the Investigator would preclude the safe participation of the subject in the study or would prevent the subject from meeting the study requirements.
- 13. Subjects must not have any condition that in the opinion of the Investigator could impact drug absorption (e.g. gastrectomy, Roux-en-Y gastric bypass surgery, gastric bands or staples, etc.), distribution, or elimination.
- 14. Subjects must not have poorly controlled diabetes mellitus (HbA1c  $\geq$ 8.5% at Screening).
- 15. Subjects must not have moderate or severe hepatic and/or renal disease (defined in Appendix B and Appendix C).
- 16. Subjects must not have a laboratory abnormality that in the opinion of the Investigator is likely to introduce additional risk to the subject or might interfere with data interpretation. The specific findings listed below are excluded at Screening (a single repeat laboratory evaluation is allowed for eligibility determination, except for HIV, HbsAg and antibodies to hepatitis C virus):

- a. Serum ALT  $\geq$ 2.0x the upper limit of normal (ULN) of the reference range.
- b. Serum AST  $\geq 2.0x$  the ULN of the reference range.
- c. Serum total bilirubin  $\ge 1.5x$  the ULN of the reference range, unless the elevation is consistent with Gilbert's Syndrome.
- d. Electrocardiographic QTc interval >470 msec as corrected by the Fridericia formula, or any clinically significant electrocardiographic abnormality.
- e. Positive test for antibodies to human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or antibodies to hepatitis C virus.
- 17. Subjects of childbearing potential must not be pregnant (positive pregnancy test at Screening), lactating, or planning to become pregnant during the study period.
- 18. Subjects must not have planned surgery or other medical procedures that in the Investigator's opinion would impact compliance with the protocol.
- 19. Subjects must not have active substance abuse (e.g., drugs of any kind, including alcohol) or any other medical, psychiatric or social condition that in the Investigator's opinion would preclude compliance with the protocol.
- 20. Subjects must not have received VT-1161 study medication in a previous study.
- 21. Subjects must not have received any IMP in a clinical trial within 5 half-lives of that IMP prior to Screening (if unknown, 60 days prior to Screening).
- 22. Subjects must not have a known history of intolerance or hypersensitivity to azole antifungal drugs (e.g., fluconazole, itraconazole, voriconazole, posaconazole, and isavuconazole), or any excipients of the capsule formulation.

### 6 INVESTIGATIONAL MEDICINAL PRODUCT

All protocol-specific criteria for administration of study treatments must be met and documented prior to IMP administration. Study treatments will be administered only to eligible subjects under the supervision of the Investigator.

### 6.1 Fluconazole

Fluconazole tablets or capsules containing 150 mg of active pharmaceutical ingredient for the Induction Phase of the study will be provided by Mycovia Pharmaceuticals (or its designee) or by the Investigator for use in the Induction Phase and for treatment of acute VVC episodes during the Maintenance Phase (as described in Section 7.4.2).

### 6.2 Description of Investigational Medicinal Product

### 6.2.1 VT-1161

Active IMP will be supplied by Mycovia Pharmaceuticals (or its designee) as capsules containing 150 mg of VT-1161.

### 6.2.2 Placebo

Placebo will be supplied by Mycovia Pharmaceuticals (or its designee) as capsules matching the appearance of VT-1161 capsules.

# 6.3 Investigational Medicinal Product Labeling and Packaging

Mycovia Pharmaceuticals (or its designee) will package the VT-1161 and placebo capsules. IMP will be supplied according to applicable regulatory requirements. Information pertaining to labeling and a description of the specific packaging and storage conditions will be supplied to the Investigator or designee.

VT-1161 and placebo will be provided in bottles for daily dosing on Days 1-7 and weekly dosing through Week 12 of the study.

# 6.4 Investigational Medicinal Product Storage Conditions

IMP will be stored in a secure location at a controlled room temperature of 15°C to 25°C (59°F to 77°F) and protected from light and moisture. The storage of IMP will be locked with limited access, available to appropriate study personnel only.

# 6.5 Receipt of Supplies/Handling/Storage

Only subjects enrolled in the study may receive study treatment, and only authorized site staff may supply or administer study treatment. All study treatments must be stored in a secure environmentally controlled and monitored area in accordance with the labelled storage conditions with access limited to the Investigator and authorized staff.

Further guidance and information for final disposition of unused study treatments are provided in the Study Procedures Manual.

# 6.6 Investigational Medicinal Product Accountability

Mycovia Pharmaceuticals will provide the Investigator with sufficient amounts of IMP. It is the responsibility of the Investigator to ensure that a current record of inventory/IMP accountability is maintained.

### 6.7 Investigational Medicinal Product Return

Upon the completion or termination of the study, and with supporting documentation from Mycovia Pharmaceuticals (or designee), all unused and/or partially used IMP should be returned to Sponsor or its designee or destroyed at the investigational site per the site's standard operating procedure (SOP) for IMP destruction. Prior to destruction of any used or unused IMP at a site, Mycovia Pharmaceuticals (or designee) must review and provide written documentation that:

- 1. The site SOP for IMP destruction is acceptable.
- 2. The clinical site monitor has conducted and documented full accountability of the IMP.

### 7 TREATMENT OF SUBJECTS

### 7.1 Investigational Medicinal Product Administration and Dosing Schedule

### 7.1.1 Induction Phase (Screening to Day 1 Pre-Randomization)

All subjects will receive 3 sequential 150 mg doses of fluconazole that are administered 72 hours apart.

Regarding the dosing of fluconazole in adolescent subjects (12 to 17 years of age, inclusive), fluconazole exposure at the planned dose is anticipated to be similar to that in adults and proportional to weight. AEs associated with fluconazole would also be expected to be similar in adolescents as in adults. There are currently no United States FDA- or European-approved doses or regimens of fluconazole for treatment of VVC or RVVC in adolescents. While the United States FDA-approved labeling for fluconazole (Diflucan, Pfizer 2017) is silent on treatment of adolescents with VVC, the European prescribing information for fluconazole (Diflucan® Summary of Product Characteristics [2017]) provides the following guidance; "If treatment is imperative in adolescents (from 12 to 17 years old), the posology should be the same as in the adult population." Therefore, adolescent subjects (ages 12 to 17 years) enrolled in the study will receive the same 150 mg doses of fluconazole as adult subjects.

In Hungary, Romania, Ukraine, and Czech Republic, only subjects 18 years of age or older will be enrolled in the study.

### 7.1.2 Maintenance Phase (Day 1 Post Randomization to Week 12)

Subjects will receive either:

- 150 mg once daily dose of VT-1161 for 7 days followed by a 150-mg once weekly dose of VT-1161 for 11 weeks, or
- a matching placebo regimen for 12 weeks.

All subjects will take 1 capsule once daily on Days 1 to 7 and 1 capsule once weekly starting at Week 2 (7 days after the completion of daily dosing) through Week 12 of the study.

Subjects will be instructed to take the doses of VT-1161 within 30 minutes after ingestion of the subject's main meal (as determined by the subject), at approximately the same time of the day consistently throughout the study. Subjects should consume approximately 240 mL (approximately 8 oz.) of water with each dose of IMP.

IND 111675 Ver. 6 U.S. Only, 01 October 2019

Using similar rationale as above for fluconazole, the exposure after dosing of VT-1161 at 150 mg doses is anticipated to be similar in adolescents as in adults and proportional to weight. Therefore, adolescents (ages 12 to 17 years) enrolled into the study will receive the same dosing regimen as adult subjects. It should also be noted that the United States FDA has reviewed this protocol and accepted the planned dosing regimen for fluconazole and VT-1161 in adolescent subjects.

# 7.2 Method of Assigning Subjects to Treatment Groups

Each subject who completes the study Screening assessments, meets all eligibility criteria, and is accepted for the study will be assigned a unique sequential identification number and will receive the corresponding treatment according to the randomization scheme described in the Statistical Analysis Plan (SAP). For more information on subject randomization, see Section 7.7.

# 7.3 Dose Interruptions and Modifications

If any subject experiences a Grade 3 AE that is considered possibly related, or related to IMP, dosing will be discontinued in that subject and the AE will be followed until resolution (refer to Section 9.2 for AE reporting). Dosing of IMP will not be re-initiated in any subject who experiences a possibly related or related Grade 3 AE. Although these subjects should stop the study drug, they are encouraged to return for their remaining study visits. Elevation in laboratory values that do not require medical or surgical treatment or discontinuation from the study will not be considered AEs (Section 9.2.1).

If any subject experiences a Grade 4 AE that is considered possibly related or related to IMP, the subject may be unblinded at the discretion of the Investigator and dosing of IMP will be discontinued and the AE will be followed until resolution. Dosing of IMP will not be re-initiated in any subject who experiences a possibly related or related Grade 4 AE.

### 7.4 Prohibited and Permitted Medications/Non-Medications

All medications taken 30 days prior to the Screening visit including all prescription and non-prescription medications (e.g., herbal and/or vitamin supplements), through the End of Study (EOS) visit will be recorded for each subject.

All concomitant therapies and procedures (including any surgical and diagnostic procedures) that were performed 72 hours prior to Screening through the EOS visit will be recorded for each subject.

#### 7.4.1 Prohibited Medications/Non-Medications

The following prescription and over-the-counter drug products are prohibited during the study and will be considered a protocol deviation:

- 1. Topical or oral antifungal drugs (with the exception of fluconazole when prescribed by the Investigator to treat a subject with a recurrent VVC episode; refer to Section 8.1.12 on treatment options if fluconazole is ineffective).
- 2. Topical products applied to the vulva or vagina (e.g. antibiotic, antitrichomonal, corticosteroids, or anti-inflammatory agents).
- 3. Oral antibacterial or antitrichomonal agents for the treatment of bacterial vaginosis, trichomonas, or other concomitant (urogenital) infection unless prescribed by the Investigator.
- 4. Oral or injectable corticosteroid or immunosuppressive drugs for the duration of the study. Use of topical (no vulvar or vaginal steroids), inhaled, ophthalmic, collunarium/nasal, or intraarticular and intralesional steroids is permitted.
- 5. Drugs with a narrow therapeutic index that are metabolized by CYP3A4 and sensitive to the induction of CYP3A4 (carbamazepine, cyclosporine, fentanyl, quinidine, sirolimus and tacrolimus).
- 6. Vaginal douches or benzalkonium chloride disinfectant during the study.

### 7.4.2 Permitted Medications/Non-Medications

The Investigator may prescribe a single dose of fluconazole to treat an acute VVC recurrence during the Maintenance Phase, when confirmed by a positive local KOH or Gram stain showing presence of yeast and clinical signs and symptoms score of  $\geq 3$ .

Medications to treat any AEs the subject experiences during the study are permitted. If a subject is unable to comply with the excluded medications criteria (Section 7.4.1), the subject's continued participation in the study will be re-evaluated by the Investigator, in consultation with Mycovia Pharmaceuticals' Medical Monitor.

# 7.5 Treatment Compliance

IMP will be administered or dispensed only to eligible subjects under the supervision of the Investigator.

# 7.6 Replacement of Study Subjects

Any subject who receives  $\geq 1$  dose of study drug will be considered evaluable and will not be replaced.

# 7.7 Randomization and Blinding

A randomized design through an interactive web response system (IWRS) will be used to assign subjects in a 2:1 ratio to the dose regimen of VT-1161 or placebo. Day 1 (Baseline) is defined as the first day of VT-1161/Placebo administration and subsequent study days are defined by the number of consecutive days thereafter.

The subjects, study Investigators and their staff, all clinical staff members within Mycovia Pharmaceuticals, the clinical study monitor, the study project team, and the study Medical Monitor(s) will remain blinded to individual treatment assignments until the completion of the study. The Unblinded Statistician responsible for creating the final randomization list and the IWRS personnel responsible for loading the final randomization list into the IWRS will be unblinded to the treatments. The bioanalytical personnel responsible for assay of VT-1161 in plasma samples will also be unblinded to subject treatments.

# 7.8 Conditions for Breaking the Blind

In the event the breaking of the blind is required, the following will apply:

- The Investigator may unblind a subject's treatment assignment only in the case of an emergency (i.e., a Grade 4 AE) OR in the event of a serious medical condition when knowledge of the study treatment is essential for the appropriate clinical management or welfare of the subject as judged by the Investigator (ICH GCP 4.3.1). If the SAE requires that an expedited regulatory report be sent to 1 or more regulatory agencies, a copy of the report, identifying the subject's treatment assignment, may be sent to Investigators in accordance with local regulations.
- The Investigator must contact the Medical Monitor or appropriate Mycovia Pharmaceuticals study personnel to communicate the reasons for unblinding the subject's treatment assignment immediately after the unblinding occurred (ICH GCP 4.7).
- If unblinding is required, the Mycovia Pharmaceuticals' Medical Monitor and Investigator will be provided with the treatment assigned to the subject. The Investigator must NOT disclose the treatment assignment to the subject and/or other study personnel including other site

personnel, monitors, or the Sponsor's project team; nor should there be any written or verbal disclosure of the code in any of the corresponding subject documents. The treatment assignment of the subject is to be revealed only if that information is important to the safety of subjects currently in the study.

• The date and reason for unblinding must be fully documented in the eCRF.

# 7.9 Treatment After the End of the Study

After the completion of the study, Mycovia Pharmaceuticals will follow local regulatory/International Conference on Harmonisation (ICH) guidelines for any follow-up treatment provided to subjects. The Investigator is responsible for ensuring that consideration has been given to the post-study care of a subject's medical condition.

# 8 STUDY PROCEDURES

# 8.1 Assessments and Procedures

The study subjects should be seen within the timeframes noted in the Table 1. Schedule of Assessments and Procedures. All study visits should be scheduled within the visit windows and projected from the Baseline (Day 1) visit.

Table 1. Schedule of Assessments and Procedures

| Activities | Screening<br>Day -14<br>(±2 days) | Baseline<br>(Day 1) | Day 14<br>(±2 days) | <b>Week 6</b> (±7 days) | Week 12<br>(±14 days)<br>EOT | Week 18<br>(±14 days) | Week 24<br>(± 14 days) | Week 30<br>(± 14 days) | Week 36<br>(± 14 days) | Week 42<br>(± 14 days) | Week 48<br>(± 14 days)<br>EOS | Unscheduled<br>Visit <sup>j</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Sign Informed Consent or Assent Form | X | 7. | | | | | | | | | | 1 |
| Inclusion/ Exclusion Criteria | X | X | | | - | | | | - | | | |
| Medical/Surgical History | X | Λ | | | | | | | | | | |
| Prior/Concomitant Medications/ Treatments <sup>a</sup> | X | X | v | v | X | v | X | v | v | v | X | X |
| Collect and record AEs | Λ | X | X | X | X | X | X | X | X | X | X | X |
| 1 - 5 - C | X | Λ | Λ | Λ | Λ | A | X | Λ | Λ | Λ | X | X |
| Patient Reported Outcome Surveys <sup>b</sup> | X | | | | | | Λ | | | | Λ | Λ |
| RVVC History Questionnaire (US Only) | X | | s. | | 370 | | 3/C | 8 | | 7 | 370 | |
| Body height and weight Vital signs <sup>d</sup> | X | 37 | v | v | X <sup>c</sup> | V | X <sup>c</sup> | v | v | v | X <sup>c</sup> | 37 |
| | | X | X | X | | X | | X | X | X | | X |
| Physical and Vaginal Examination | X | Xe | Xe | Xe | Xe | Xe | Xe | Xe | Xe | Xe | Xe | Xe |
| Clinical Signs & Symptoms of Vulvovaginitis | X | X | X | X | X | X | X | X | X | X | X | X |
| Local KOH Wet Mount or Gram stain | X | | | | | | | | | | | X |
| Central Vaginal Fungal Culture | X | X | X | X | X | X | X | X | X | X | X | X |
| ECG | X | X | X | | X | | X | 3<br>8 | | | X | |
| PK Samples <sup>f</sup> | | X | X | | X | | X | | X | | X | X |
| Clinical Laboratory Samples | X | X | X | X | X | X | X | X | X | X | X | X |
| Urinalysis | X | X | X | | X | | X | | X | | X | |
| Hematology (CBC with differential) | X | X | X | | X | | X | | X | | X | |
| HIV Ab, HbsAg, anti-HCV | X | | | | | | | | | | | |
| Central Serum Pregnancy Testh (WOCBP) | X | X | | | X | | X | | | | X | |
| Local Urine Pregnancy Testh (WOCBP) | X | X | X | X | X | X | X | X | X | X | X | X |
| Administer Fluconazole | X | | | | | | | | | | | |
| Randomization | | X | | | | | | | | | | |
| Administer and/or Review IMPi | | X | X | X | X | | | | | | | |

#### Protocol VMT-VT-1161-CL-012

Abbreviations noted above – AEs: adverse events; CBC, complete blood count; ECG: electrocardiogram; EOS: End of Study; HbsAg: Hepatitis B surface antigen; HCV: Hepatitis C virus; HIV: human immunodeficiency virus; IMP, investigational medicinal product; KOH: potassium hydroxide prep; PK: pharmacokinetic; WOCBP: women of childbearing potential.

- a. All medication taken 30 days prior to Screening and all non-pharmacologic treatments received 72 hours prior to Screening will be recorded through the EOS visit.
- b. SF-36, EQ-5D-3L or EQ-5D-Y (for ages 12 to 17), WPAI:SHP, and PHQ-9 patient reported outcome surveys.
- c. Weight only
- d. Vital signs include sitting heart rate, blood pressure, temperature, and respiratory rate.
- e. Limited Physical Examination, i.e. vaginal speculum examination plus a symptom directed physical examination
- f. The initial PK sample must be drawn prior to the first dose of study drug (placebo/VT-1161).
- g. Serum chemistry (creatinine, BUN, AST, ALT, alkaline phosphatase, total bilirubin, conjugated bilirubin, albumin, total protein, total carbon dioxide, glucose, sodium, potassium, chloride, calcium, and phosphorus, creatine phosphokinase [CK], cholesterol, and triglycerides). Testing for HbA1c is performed for all subjects only at Screening. Cultures to test for *Chlamydia trachomatis* and *Neisseria gonorrhoeae* will be taken at Screening and sent to the central lab. Testing for *Bacterial vaginosis* will be done locally at Screening. An OSOM® Rapid test or similar test will be performed for *Trichomonas vaginalis* locally at Screening.
- h. For WOCBP, a local lab urine pregnancy test will be obtained at every study visit. A central lab serum pregnancy test will be performed at Screening, Baseline, and Weeks 12, 24, and 48.
- i. IMP is to be administered within 30 minutes after the subject's main meal of the day (as determined by the subject) at approximately the same time of the day consistently throughout the study. Approximately 240 mL (64icromo. 8 oz.) of water is to be consumed with each dose of IMP. Remind subject to bring IMP to each visit to ensure compliance.
- j. All procedures listed are to be completed only for unscheduled visits where a recurrent VVC episode is suspected. If the unscheduled visit is for repeat procedures (i.e., ECG, safety labs, etc.), only those specific procedures need to be performed, along with collection of any changes in medical treatments or medications and collection of any AEs.

### 8.1.1 Screening Assessments and Procedures (Day -14 ±2 Days)

Subjects will be screened 14 days prior to randomization. The subject will start open-label fluconazole treatment at Screening if the subject has met all preliminary enrollment criteria, (central lab results are not required to initiate fluconazole treatment). Proper written informed consent (or assent for those ages 12 to 17) must be obtained from all subjects prior to any study procedures, see Section 13.2 for more information. Once the subject has signed the Institutional Review Board (IRB) / Independent Ethic Committee (IEC) approved informed consent document or assent the following evaluations will be performed to assess subject eligibility:

- 1. Review Inclusion and Exclusion criteria.
- 2. Document subject demographics, including date of birth, race, and ethnic origin.
- 3. Document and review medical/medication and surgical history, including all current, pertinent and major past illnesses and surgical procedures. All concomitant therapies or procedures (including any surgical or diagnostic procedures) that were performed 72 hours prior to the Screening will be recorded.
- 4. Review alcohol and tobacco history (previous 12 months).
- 5. Record all medications, including prescription and non-prescription medications, herbal products, and vitamin/mineral supplements taken within 30 days prior to Screening.
- 6. Administer the SF-36, EQ-5D-3L or EQ-5D-Y (for ages 12 to 17), WPAI:SHP, and PHQ-9 Patient Reported Outcomes Surveys for all regions and RVVC History Questionnaire (US only).
- 7. Assess height and weight to determine the body mass index.
- 8. Obtain vital signs in the sitting position (blood pressure, heart rate, respiratory rate, and temperature).
- 9. Conduct a comprehensive physical examination, including vaginal exam, as described in Section 9.1.3. For proper assessment, it is best the subject is not menstruating at time of the visit.

- 10. Recording of clinical signs and symptoms of vulvovaginitis, as outlined in Section 9.1.7. Subjects must be cautioned to not use any treatment (topical or systemic) for their infection during the Screening period.
- 11. KOH wet mount test or Gram stain, performed locally (Section 9.1.6).
- 12. Vaginal swab for culture will be obtained and sent to the central mycology laboratory (Section 9.1.6).
- 13. Standard 12-lead ECG will be obtained in the supine position (Section 9.1.4).
- 14. Clinical chemistries, hematology, and urinalysis for study eligibility as outlined in Section 9 and the Schedule of Assessments and Procedures. Cultures for testing of *Chlamydia trachomatis* and *Neisseria gonorrhoeae* will also be taken. Vaginal pH will be determined. Local testing will be done for *Bacterial vaginosis* and an OSOM® Rapid test or similar test will be performed locally for *Trichomonas vaginalis*.
- 15. Testing for HbsAg, HCV, and HIV as outlined in Section 9.1.5.2 and the Schedule of Assessments and Procedures. (Results for these tests are not required for the start of Induction Phase- treatment with fluconazole).
- 16. A urine pregnancy test will be performed locally and a serum pregnancy test will be obtained and sent to the central laboratory for all women of childbearing potential (WOCBP).
- 17. Provide subject with 3 doses of fluconazole. The subject should be advised to take one fluconazole tablet or capsule on the day of the visit (day 1) and on days 4 and 7 at home, at approximately the same time of the day.
- 18. Remind subject to return for Day 1 visit.

Central laboratory results are not required prior to start of treatment with fluconazole.

Subjects may be eligible for re-screening, one time. The investigative site is to refer to the Study Procedures Manual and contact the study clinical monitor for guidance.

### 8.1.2 Baseline (Day 1) Assessments and Procedures (Day -14 ±2 Days)

The subjects will return to the investigative site for the following evaluations:

- 1. Confirm all Inclusion and Exclusion criteria have been met
- 2. Record all medications taken since the previous visit, including all prescription and non-prescription medications, herbal products, and vitamin/mineral supplements. All concomitant therapies or procedures (including any surgical or diagnostic procedures) that were performed since the last visit will be recorded.
- 3. Review and record any AEs.
- 4. Obtain vital signs in the sitting position, (blood pressure, heart rate, respiratory rate, and temperature).
- 5. Limited physical examination, includes vaginal exam (as described in Section 9.1.3). For proper assessment, it is best the subject is not menstruating at time of the visit.
- 6. Recording of clinical signs and symptoms of vulvovaginitis, as outlined in Section 9.1.7. Subjects must be cautioned to not use any treatment (topical or systemic) for vulvovaginitis except study drug.
- 7. Vaginal swab for culture will be obtained and sent to the central mycology laboratory (Section 9.1.6).
- 8. Standard 12-lead ECG will be obtained in the supine position (Section 9.1.4).
  - 9. Obtain PK plasma specimen. The initial PK sample must be drawn prior to the first dose of study drug (placebo/VT-1161).

10.

- 11. Obtain clinical chemistries, hematology, and urinalysis as outlined in Section 9 and the Schedule of Assessments and Procedures.
- 12. A urine pregnancy test will be performed locally and a serum pregnancy test will be obtained and sent to the central laboratory for all WOCBP.
- 13. IWRS randomization of the subject to a treatment arm.
- 14. Provide bottle for IMP daily dosing to subject along with instructions.

15. Remind subject to return for Day 14 ( $\pm 2$  days) visit.

### 8.1.3 Day 14 (±2 Days) Assessments and Procedures

Subjects will return to the investigative site for follow-up evaluation as follows:

- 1. Record all medications taken since the previous visit, including all prescription and non-prescription medications, herbal products, and vitamin/mineral supplements. All concomitant therapies or procedures (including any surgical or diagnostic procedures) that were performed since the previous visit.
- 2. Review and record any AEs.
- 3. Obtain vital signs in the sitting position, (blood pressure, heart rate, respiratory rate, and temperature).
- 4. Limited physical examination, includes vaginal exam (as described in Section 9.1.3). For proper assessment, it is best the subject is not menstruating at time of the visit.
- 5. Recording of clinical signs and symptoms of vulvovaginitis, as outlined in Section 9.1.7. Subjects must be cautioned to not use any treatment (topical or systemic) for vulvovaginitis except study drug.
- 6. Vaginal swab for culture will be obtained and sent to the central mycology laboratory (Section 9.1.6).
- 7. Standard 12-lead ECG will be obtained in the supine position (Section 9.1.4).
- 8. Obtain PK plasma specimen.
- 9. Obtain clinical chemistries, hematology, and urinalysis as outlined in Section 9 and the Schedule of Assessments and Procedures.
- 10. A urine pregnancy test will be performed locally for all WOCBP.
- 11. Collect and review accountability of IMP daily dose bottle with the subject for compliance.
- 12. Dispense bottle for IMP weekly dosing to the subject along with instructions
- 13. Remind subject to return for Week 6 ( $\pm$ 7 days) visit.

Ver. 6 U.S. Only, 01 October 2019

### 8.1.4 Week 6 (±7 Days) Assessments and Procedures

Subjects will return to the investigative site for follow-up evaluation as follows:

- 1. Record all medications taken since the previous visit, including all prescription and nonprescription medications, herbal products, and vitamin/mineral supplements. All concomitant therapies or procedures (including any surgical or diagnostic procedures) that were performed since the previous visit.
- 2. Review and record any AEs.
- 3. Obtain vital signs in the sitting position, (blood pressure, heart rate, respiratory rate, and temperature).
- 4. Limited physical examination, includes vaginal exam (as described in Section 9.1.3). For proper assessment, it is best the subject is not menstruating at time of the visit.
- 5. Recording of clinical signs and symptoms of vulvovaginitis, as outlined in Section 9.1.7. Subjects must be cautioned to not use any treatment (topical or systemic) for vulvovaginitis except study drug.
- 6. Vaginal swab for culture will be obtained and sent to the central mycology laboratory (Section 9.1.6).
- 7. Obtain clinical chemistries, as outlined in Section 9.1.5.3.
- 8. A urine pregnancy test will be performed locally for all WOCBP.
- 9. Review accountability of IMP weekly dose bottle with the subject for compliance.
- 10. Remind subject to return for Week 12 ( $\pm$ 14 days) visit.

### 8.1.5 Week 12 (±14 Days) Assessments and Procedures

The subjects will return to the investigative site for the following evaluations:

- 1. Record all medications taken since the previous visit, including all prescription and nonprescription medications, herbal products, and vitamin/mineral supplements. All concomitant therapies or procedures (including any surgical or diagnostic procedures) that were performed since the previous visit.
- 2. Review and record any AEs.

- 3. Obtain body weight.
- 4. Obtain vital signs in the sitting position, (blood pressure, heart rate, respiratory rate, and temperature).
- 5. Limited physical examination, includes vaginal exam (as described in Section 9.1.3). For proper assessment, it is best the subject is not menstruating at time of the visit.
- 6. Recording of clinical signs and symptoms of vulvovaginitis, as outlined in Section 9.1.7. Subjects must be cautioned to not use any treatment (topical or systemic) for vulvovaginitis except study drug.
- 7. Vaginal swab for culture will be obtained and sent to the central mycology laboratory (Section 9.1.6).
- 8. Standard 12-lead ECG will be obtained in the supine position (Section 9.1.4).
- 9. Obtain PK plasma specimen.
- 10. Obtain clinical chemistries, hematology, and urinalysis as outlined in Section 9 and the Schedule of Assessments and Procedures.
- 11. A urine pregnancy test will be performed locally and a serum pregnancy test will be obtained and sent to the central laboratory for all WOCBP.
- 12. Collect and conduct final review accountability of IMP **weekly dose** bottle with the subject for compliance.
- 13. Remind subject to return for Week 18 ( $\pm$ 14 days) visit.
# 8.1.6 Week 18 (±14 Days) Assessments and Procedures

The subjects will return to the investigative site for the following evaluations:

- 1. Record all medications taken since the previous visit, including all prescription and non-prescription medications, herbal products, and vitamin/mineral supplements. All concomitant therapies or procedures (including any surgical or diagnostic procedures) that were performed since the previous visit.
- 2. Review and record any AEs.
- 3. Obtain vital signs in the sitting position, (blood pressure, heart rate, respiratory rate, and temperature).
- 4. Limited physical examination, includes vaginal exam (as described in Section 9.1.3). For proper assessment, it is best the subject is not menstruating at time of the visit.
- 5. Recording of clinical signs and symptoms of vulvovaginitis, as outlined in Section 9.1.7. Subjects must be cautioned to not use any treatment (topical or systemic) for vulvovaginitis except study drug.
- 6. Vaginal swab for culture will be obtained and sent to the central mycology laboratory (Section 9.1.6).
- 7. Obtain clinical chemistries, as outlined in Section 9.1.5.3.
- 8. A urine pregnancy test will be performed locally for all WOCBP.
- 9. Remind subject to return for Week 24 (±14 days) visit.

#### 8.1.7 Week 24 (±14 Days) Assessments and Procedures

- 1. Record all medications taken since the previous visit, including all prescription and non-prescription medications, herbal products, and vitamin/mineral supplements. All concomitant therapies or procedures (including any surgical or diagnostic procedures) that were performed since the previous visit.
- 2. Review and record any AEs.

- 3. Administer the SF-36, EQ-5D-3L or EQ-5D-Y (for ages 12 to 17), WPAI:SHP, and PHQ-9 Patient Reported Outcomes Surveys.
- 4. Obtain body weight.
- 5. Obtain vital signs in the sitting position, (blood pressure, heart rate, respiratory rate, and temperature).
- 6. Limited physical examination, includes vaginal exam (as described in Section 9.1.3). For proper assessment, it is best the subject is not menstruating at time of the visit.
- 7. Recording of clinical signs and symptoms of vulvovaginitis, as outlined in Section 9.1.7. Subjects must be cautioned to not use any treatment (topical or systemic) for vulvovaginitis except study drug.
- 8. Vaginal swab for culture will be obtained and sent to the central mycology laboratory (Section 9.1.6).
- 9. Standard 12-lead ECG will be obtained in the supine position (Section 9.1.4).
- 10. Obtain PK plasma specimen.
- 11. Obtain clinical chemistries, hematology, and urinalysis as outlined in Section 9 and the Schedule of Assessments and Procedures.
- 12. A urine pregnancy test will be performed locally and a serum pregnancy test will be obtained and sent to the central laboratory for all WOCBP.
- 13. Remind subject to return for Week 30 ( $\pm$ 14 days) visit.

# 8.1.8 Week 30 (±14 Days) Assessments and Procedures

- 1. Record all medications taken since the previous visit, including all prescription and non-prescription medications, herbal products, and vitamin/mineral supplements. All concomitant therapies or procedures (including any surgical or diagnostic procedures) that were performed since the previous visit.
- 2. Review and record any AEs.

- 3. Obtain vital signs in the sitting position, (blood pressure, heart rate, respiratory rate, and temperature).
- 4. Limited physical examination, includes vaginal exam (as described in Section 9.1.3). For proper assessment, it is best the subject is not menstruating at time of the visit.
- 5. Recording of clinical signs and symptoms of vulvovaginitis, as outlined in Section 9.1.7. Subjects must be cautioned to not use any treatment (topical or systemic) for vulvovaginitis except study drug.
- 6. Vaginal swab for culture will be obtained and sent to the central mycology laboratory (Section 9.1.6).
- 7. Obtain clinical chemistries, as outlined in Section 9.1.5.3.
- 8. A urine pregnancy test will be performed locally for all WOCBP.
- 9. Remind subject to return for Week 36 ( $\pm 14$  days) visit.

# 8.1.9 Week 36 (±14 Days) Assessments and Procedures

- 1. Record all medications taken since the previous visit, including all prescription and non-prescription medications, herbal products, and vitamin/mineral supplements. All concomitant therapies or procedures (including any surgical or diagnostic procedures) that were performed since the previous visit.
- 2. Review and record any AEs.
- 3. Obtain vital signs in the sitting position, (blood pressure, heart rate, respiratory rate, and temperature).
- 4. Limited physical examination, includes vaginal exam (as described in Section 9.1.3). For proper assessment, it is best the subject is not menstruating at time of the visit.
- 5. Recording of clinical signs and symptoms of vulvovaginitis, as outlined in Section 9.1.7. Subjects must be cautioned to not use any treatment (topical or systemic) for vulvovaginitis except study drug.

- 6. Vaginal swab for culture will be obtained and sent to the central mycology laboratory (Section 9.1.6).
- 7. Obtain PK plasma specimen.
- 8. Obtain clinical chemistries, hematology, and urinalysis as outlined in Section 9 and the Schedule of Assessments and Procedures.
- 9. A urine pregnancy test will be performed locally for all WOCBP.
- 10. Remind subject to return for Week 42 ( $\pm 14$  days) visit.

#### 8.1.10 Week 42 (±14 Days) Assessments and Procedures

- 1. Record all medications taken since the previous visit, including all prescription and non-prescription medications, herbal products, and vitamin/mineral supplements. All concomitant therapies or procedures (including any surgical or diagnostic procedures) that were performed since the previous visit.
- 2. Review and record any AEs.
- 3. Obtain vital signs in the sitting position, (blood pressure, heart rate, respiratory rate, and temperature).
- 4. Limited physical examination, includes vaginal exam (as described in Section 9.1.3). For proper assessment, it is best the subject is not menstruating at time of the visit.
- 5. Recording of clinical signs and symptoms of vulvovaginitis, as outlined in Section 9.1.7. Subjects must be cautioned to not use any treatment (topical or systemic) for vulvovaginitis except study drug.
- 6. Vaginal swab for culture will be obtained and sent to the central mycology laboratory (Section 9.1.6).
- 7. Obtain clinical chemistries, as outlined in Section 9.1.5.3.
- 8. A urine pregnancy test will be performed locally for all WOCBP.
- 9. Remind subject to return for Week 48 ( $\pm 14$  days) visit.

# 8.1.11 Week 48 (±14 Days) Assessments and Procedures (End of Study)

- 1. Record all medications taken since the previous visit, including all prescription and non-prescription medications, herbal products, and vitamin/mineral supplements. All concomitant therapies or procedures (including any surgical or diagnostic procedures) that were performed since the previous visit.
- 2. Review and record any AEs.
- 3. Administer the SF-36, EQ-5D-3L or EQ-5D-Y (for ages 12 to 17), WPAI:SHP, and PHQ-9 Patient Reported Outcomes Surveys.
- 4. Obtain body weight.
- 5. Obtain vital signs in the sitting position, (blood pressure, heart rate, respiratory rate, and temperature).
- 6. Limited physical examination, includes vaginal exam (as described in Section 9.1.3). For proper assessment, it is best the subject is not menstruating at time of the visit.
- 7. Recording of clinical signs and symptoms of vulvovaginitis, as outlined in Section 9.1.7. Subjects must be cautioned to not use any treatment (topical or systemic) for vulvovaginitis except study drug.
- 8. Vaginal swab for culture will be obtained and sent to the central mycology laboratory (Section 9.1.6).
- 9. Standard 12-lead ECG will be obtained in the supine position (Section 9.1.4).
- 10. Obtain PK plasma specimen.
- 11. Obtain clinical chemistries, hematology, and urinalysis as outlined in Section 9 and the Schedule of Assessments and Procedures.
- 12. A urine pregnancy test will be performed locally and a serum pregnancy test will be obtained and sent to the central laboratory for all WOCBP.

If the Investigator suspects the subject is experiencing a recurrent episode at a regular study visit, a local KOH wet mount test or Gram stain is to be performed to confirm whether filamentous hyphae/pseudohyphae and/or budding yeast cells are present.

#### **8.1.12** Unscheduled Visit Assessment and Procedures

Subjects should be encouraged to return for an unscheduled visit if they experience a recurrence of VVC anytime during the study. The following evaluations are to be performed:

- 1. Record all medications taken since the previous visit, including all prescription and non-prescription medications, herbal products, and vitamin/mineral supplements. All concomitant therapies or procedures (including any surgical or diagnostic procedures) that were performed since the previous visit.
- 2. Review and record any AEs.
- 3. Administer the SF-36, EQ-5D-3L or EQ-5D-Y (for ages 12 to 17), WPAI:SHP, and PHQ-9 Patient Reported Outcomes Surveys.
- 4. Obtain vital signs in the sitting position, (blood pressure, heart rate, respiratory rate, and temperature).
- 5. Limited physical examination, includes vaginal exam (as described in Section 9.1.3). For proper assessment, it is best the subject is not menstruating at time of the visit.
- 6. Recording of clinical signs and symptoms of vulvovaginitis, as outlined in Section 9.1.7. Subjects must be cautioned to not use any treatment (topical or systemic) for vulvovaginitis except study drug.
- 7. KOH wet mount test or Gram stain, performed locally (Section 9.1.6).
- 8. Vaginal swab for culture will be obtained and sent to the central mycology laboratory (Section 9.1.6).
- 9. Obtain PK plasma specimen.
- 10. A urine pregnancy test will be performed locally for all WOCBP.
- 11. Obtain clinical chemistries, as outlined in Section 9.1.5.3.

If a subject has a recurrent acute VVC episode prior to the end of treatment at Week 12, the subject will continue her assigned treatment through Week 12 and will receive one dose of fluconazole to treat her acute VVC infection. Throughout the Maintenance Phase, the Investigator is to prescribe one dose of fluconazole to treat the acute VVC episode, once confirmed by a positive KOH or Gram stain to show presence of yeast and if the clinical signs and symptoms score is  $\geq 3$ . If the subject fails to respond to fluconazole treatment, the Investigator may employ treatment options corresponding to the site's standard of care treatment for treating the infection upon consultation with the Medical Monitor.

If a subject comes in for an unscheduled visit to repeat a procedure (i.e., ECG, safety labs, etc.), only those specific procedures need to be performed, along with collection of any changes in medical treatments, medications and collection of any AEs.

If subjects experience any AEs other than a potential recurrent VVC episode they may be evaluated at the site at the Investigators discretion.

# 8.2 Exercise

Subjects will be encouraged, if possible, to avoid engaging in strenuous activity within 48 hours prior to study visits. Walking at a normal pace during these periods is acceptable.

# 9 SAFETY ASSESSMENTS

# 9.1 Safety Tests and Assessments

Safety assessments will include attention to relevant changes in the following parameters, which are identified as occurring after the start of IMP, regardless of whether the change is in an examination finding, test result, or symptom(s) reported by a subject, and regardless of presumed relationship to IMP (VT-1161 or placebo). The Investigator will follow all clinically significant abnormal findings after IMP treatment until resolution, return to baseline, or permanent documented change in medical history.

# 9.1.1 Height and Weight

Height and body weight will be collected at times specified in the Table 1. Schedule of Assessments and Procedures.

#### 9.1.2 Vital Signs

Vital signs to include body temperature, heart rate (pulse), breathing rate, and blood pressure will be obtained in a sitting position at times specified in the Table 1. Schedule of Assessments and Procedures.

#### 9.1.3 Physical Examination

Comprehensive Physical Examination: general appearance; head, eyes, ears, nose, and throat; thyroid/neck (endocrine); chest and lungs; cardiovascular system, abdomen, pelvic exam, musculoskeletal system, lymph nodes, extremities/skin, and neurological system will be performed at Screening. Special attention should be given during the vulvovaginal examination to erythema, edema, and excoriation. For proper assessment, it is best the subject is not menstruating at time of the study visits.

Symptom Directed Physical Examination: A symptom directed physical exam consists of a very brief history of present illness. Investigators should use the symptom directed exam for all study visits after the Screening visit. If the subject has no present illness this should be documented by the Investigator or qualified designee.

#### 9.1.4 Electrocardiograms

Standard 12-lead ECGs to assess heart rate, rhythm, and interval information such as PR, QRS, QT, and QTc will be obtained in the supine position at times specified in the Table 1. Schedule of Assessments and Procedures.

# **9.1.5 Laboratory Determinations**

After the Baseline (Day 1) visit, laboratory test values that fall outside the reference range on the laboratory reports and are deemed clinically significant by the Investigator may be repeated at the discretion of the Investigator. Those values deemed clinically significant should be followed until resolution or permanent documented change in medical history.

The following laboratory samples will be obtained at times specified in the Schedule of Assessments and Procedures and analyzed by the central laboratory:

# 9.1.5.1 Pregnancy Testing

All WOCBP must undergo urine and serum pregnancy testing at Screening and Baseline to assess protocol eligibility. Urine pregnancy testing will be performed at every study visit. Serum pregnancy tests will be performed periodically throughout the study as specified in the Schedule of Assessments and Procedures.

# **9.1.5.2 Immunology**

HIV antibody, HbsAg, anti-HCV at Screening. Laboratory results are not required prior to start of treatment with fluconazole. Investigators are to follow local and/or state laws in regards to parental disclosure of any positive pregnancy tests or reportable and treatable serologies or STDs in adolescents.

# 9.1.5.3 Clinical Chemistry Panel

Creatinine, blood urea nitrogen, AST, ALT, alkaline phosphatase, total bilirubin, conjugated bilirubin, albumin, total protein, total carbon dioxide, glucose, sodium, potassium, chloride, calcium, phosphorus, CK, cholesterol, and triglycerides. Testing for HbA1c should be performed for all subjects at Screening. Central laboratory results are not required prior to start of treatment with fluconazole.

After the Baseline (Day 1) visit, subjects may be re-tested for ALT, AST and total bilirubin to confirm any abnormal values and to determine if they are increasing or decreasing. The Investigator will also assess the subject for any associated emergent symptoms.

# 9.1.5.4 Hematology

A complete blood count with differential to include red blood cell count, total and differential white blood cell counts, hemoglobin, hematocrit, RBC, MCV, MCH, MCHC, RDW and platelet count will be performed at times specified in the Table 1. Schedule of Assessments

and Procedures. Central laboratory results are not required prior to start of treatment with fluconazole.

#### **9.1.5.5** Urinalysis

Testing for glucose, ketones, leukocyte esterase, nitrite, blood, pH, protein, and specific gravity will be performed at times specified in the Schedule of Assessments and Procedures. Central laboratory results are not required prior to start of treatment with fluconazole.

# 9.1.5.6 Chlamydia Trachomatis and Neisseria Gonorrhoeae

Cultures to test for *Chlamydia trachomatis* and *Neisseria gonorrhoeae* will be taken at Screening and sent to the central laboratory.

# 9.1.5.7 Trichomonas Vaginalis

An OSOM® Rapid test or similar test will be performed for *Trichomonas vaginalis* locally at Screening. Instructions for collecting, processing, storing, and shipping samples to the central laboratory are outlined in the laboratory manual.

# 9.1.5.8 Bacterial Vaginosis

Testing for *Bacterial vaginosis* will be done locally.

# 9.1.6 KOH Wet Mount Tests or Gram Stains and Fungal Cultures

A local KOH wet mount test or Gram stain will be performed locally at the Screening visit and at unscheduled visits where a recurrent VVC episode is suspected. The investigative site is to use the same local mycology test (KOH wet mount or Gram stain) consistently for all subjects throughout the study.

A vaginal fungal culture will be obtained at Screening and all subsequent visits and sent to the central mycology laboratory for fungal identification and susceptibility testing according to approved Clinical Laboratory Standards Institute methods. Subjects should not be menstruating at time of the study visits to ensure proper sample collection of the vaginal fluid. Details as to the collection of samples, shipping, testing methods and analysis will be delineated in a laboratory manual. Mycology samples may be retained for future analysis for a period of up to 15 years, after which time the samples will be destroyed.

# 9.1.7 Vulvovaginitis Clinical Assessment

Vulvovaginal signs and symptoms will be evaluated at the Screening and each subsequent study visit. Each of the following vulvovaginal signs and symptoms will be scored and the individual scores combined for a maximum score of 18, using the following scale:

- a. Signs: erythema, edema, and excoriation
- b. Symptoms: itching, burning, and irritation

Scoring Scale: Each score should be objectively defined on a scale of 0 to 3 as follows:

- 0 = none (complete absence of any signs or symptoms)
- 1 = mild (slight)
- 2 = moderate (definitely present)
- 3 = severe (marked, intense)

# 9.2 Adverse Event Reporting

#### 9.2.1 Definition of Adverse Events

Monitoring of all AEs will be conducted throughout the study as specified in the Schedule of Assessments and Procedures.

An AE is any untoward, undesired, unplanned clinical event in the form of signs, symptoms, disease, or laboratory or physiological observations occurring in a human participating in a clinical study with a Mycovia Pharmaceuticals product, regardless of causal relationship. A "pre-existing" condition is one that is present prior to the start of IMP administration and is reported as part of the subject's medical history. Pre-existing conditions should be reported as AEs only if the frequency, intensity, or character of the pre-existing condition worsens during the study.

Any abnormal safety assessments, such as ECGs, radiological scans, vital sign measurements, that are judged by the Investigator to be clinically significant should be recorded as an AE or SAE provided it meets one of those definitions. Laboratory abnormalities generally are not considered AEs unless they are associated with clinical signs or symptoms, or require medical intervention. A laboratory abnormality (e.g., a clinically significant change detected on clinical chemistry, hematology) that is independent from a known underlying medical condition and that requires medical or surgical intervention, or leads to IMP interruption or discontinuation, should be considered an AE.

Clinically significant abnormal laboratory findings or other abnormal assessments that are associated with the disease being studied are not considered AEs unless their severity is greater than expected in the judgement of the Investigator.

In addition, the following apply:

 All AEs, including clinically significant laboratory abnormalities, will be documented as an AE and followed until resolution.

All AEs and SAEs will be collected from the start of taking the first dose of fluconazole
until the last follow-up visit of the study, at the time points specified in the Schedule of
Assessments and Procedures.

• Medical occurrences that begin prior to the start of fluconazole but after obtaining informed consent should be recorded in the medical history section of the eCRF.

• Investigators are not obligated to actively seek AEs or SAEs in former study subjects. However, if the Investigator learns of an SAE, including a death, at any time after a subject has been discharged from the study, and he/she considers the event reasonably related to the study treatment or study participation, the Investigator must promptly notify Mycovia Pharmaceuticals.

#### 9.2.2 Definition of a Serious Adverse Event

An SAE is any AE occurring after the first administration of fluconazole that results in any of the following outcomes:

- Death<sup>a</sup>
- Is a life-threatening experience<sup>b</sup>
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in a persistent or significant disability/incapacity<sup>c</sup>
- Results in a congenital anomaly/birth defect
- Additionally, important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, may jeopardize the subject and may require medical or surgical intervention to

prevent 1 of the outcomes listed above. Example: allergic bronchospasm requiring intensive treatment in an emergency room or at home.

#### NOTES:

a. "Death" is an outcome and is NOT the AE. In the event of death, the cause of death should be recorded as the SAE. The only exception is "sudden death" when the cause is unknown.

b. Life-threatening SAEs include any adverse drug experience, which, in the view of the Investigator, places the subject at immediate risk of death from the reaction as it occurs. It does not include a reaction that, had it occurred in a more serious form, might have caused death.

c. Disability is defined as a substantial disruption in a person's ability to conduct normal life functions.

All SAEs, regardless of causal relationship, must be reported to Mycovia Pharmaceuticals (or designee) within 24 hours of the site's knowledge of the event. The initial report must be captured in the electronic SAE CRFs within 1 business day.

The SAE report should provide as much of the required information as is available at the time. The following minimum information is required for reporting an SAE: subject identification number, reporting source, and an event outcome. Supplemental information may be entered into the electronic SAE CRFs and should not delay the initial report. Mycovia Pharmaceuticals (or designee) may contact the investigational site to solicit additional information or to follow-up on the event.

If there is any doubt whether the information constitutes an SAE, the information will be treated as an SAE for the purposes of this protocol.

All SAEs will be followed until resolution, return to baseline (when worsening of a pre-existing condition is reported), or permanent documented change in medical history.

All relevant documentation pertaining to the SAE (additional laboratory tests, consultation reports, discharge summaries, post-mortem reports, etc.) will be provided by the Investigator to Mycovia Pharmaceuticals (or designee) in a timely manner.

# 9.2.3 Recording of Adverse Events

Subjects should be instructed to report all AEs to the Investigator. In addition, the Investigator should seek to elicit any clinical or objective reactions by open-ended questioning ("How have you been feeling?") and, as appropriate, by examination. All AE information obtained during the subject questioning should be documented in the subjects' clinical records and entered into the CRF. All clearly related signs, symptoms, and results of diagnostic procedures performed because of an AE should be grouped together and recorded as a single diagnosis. The component parts of the diagnosis may be listed for verification. If the AE is a laboratory abnormality that is part of a clinical condition or syndrome, it should be recorded as the syndrome or diagnosis rather than the individual laboratory abnormality. It should also be documented, verbatim, directly on the laboratory report.

To avoid vague, ambiguous, or colloquial expressions, all AEs should be recorded in standard medical terminology on the CRF and on the medical record rather than in the subject's own words. Each AE will also be described in terms of duration (start and stop date), severity, association with the IMP, action(s) taken, and outcome.

# 9.2.4 Severity of Adverse Events

All AEs and SAEs will be assessed by the Investigator or MD designee for severity, according to the Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Table, (Draft, November 2007) Appendix A. For AEs involving a body system or laboratory value which is not addressed in the DMID Adult Toxicity Table, the most recent version of the Common Terminology Criteria for Adverse Events, version 4.0 published by the National Cancer Institute will be used.

Where discrepancies in the ULN and lower limit of normal (LLN) laboratory ranges occur between those included in the DMID and those of the central laboratory that performs the assays, the values provided by the central laboratory will be used for assignment of severity grade.

For AEs involving a body system or laboratory value not addressed in the DMID Adult Toxicity Table, the following general scale may be used with Investigator discretion to assign severity:

• **GRADE 1 Mild**: An event easily tolerated by the subject; transient or mild discomfort (usually < 48 hours); no medical intervention/therapy required.

- **GRADE 2 Moderate**: An event that may interfere with normal, everyday activities; some assistance may be needed; no or minimal medical intervention/therapy required.
- GRADE 3 Severe: An event that prevented the subject from performing their normal, everyday activities; some assistance usually required; medical intervention/therapy required; hospitalizations possible.
- GRADE 4 Life-threatening: At the time of the event the subject was at risk of death or the event resulted in a persistent or significant disability or incapacity.
- **GRADE 5 Death**: An event that resulted in death.

When changes in the severity of an AE occur more frequently than once a day, the maximum severity for the experience that day should be noted. If the severity category changes over several days, then those changes should be recorded separately (with distinct onset dates).

NOTE: An AE that is assessed as severe should not be confused with an SAE. Severity is a category utilized for rating the intensity of an event (such as mild, moderate, or severe myocardial infarction). However, the event itself may be of relatively minor medical significance, (such as a severe headache), and both AE(s) and SAE(s) can be assessed as severe. An event is defined as 'serious' when it meets one of the pre-defined outcomes as described in Section 9.2.2.

Where discrepancies in the ULN and lower limit of normal of laboratory ranges occur between those included in the DMID tables and those of the central laboratory that performs the assays, the values provided by the central laboratory will be used for assignment of severity grade.

# 9.2.5 Causality Assessment

The Investigator is obligated to assess the relationship between the IMP and the occurrence of each AE or SAE by using his or her best clinical judgment. It should be clearly documented in the medical notes that he/she has reviewed the AE/SAE and that they are the ones providing the assessment of causality. Other elements to be considered, such as the history of the underlying disease, concomitant therapy, other risk factors, and the temporal relationship of the event to the IMP will be considered and investigated. The Investigator will also consult the VT-1161 Investigational Brochure and the study Medical Monitor in estimating the relationship.

An SAE may be recorded when the Investigator has minimal information to include in the initial report. However, the Investigator must always make an assessment of causality for every event prior to reporting the SAE report. The Investigator may change his or her opinion of the causality upon evaluation of follow-up information or discussions with the study Medical Monitor with subsequent amendment of the SAE report. *Causality assessment is one of the criteria used to determine regulatory reporting requirements and should not be left blank.* 

For each reported adverse reaction, the Investigator must assess the relationship of the event to the IMP using the following scale:

# **Unrelated:**

- Does not follow a known response pattern to the suspect IMP (if response pattern is previously known).
- Can clearly be explained by the known characteristics of the subject's clinical state or other modes of therapy administered to the subject.

# **Unlikely Related:**

- The temporal sequence from administration of the IMP suggests that a relationship is unlikely.
- Follows a response pattern that is unlike that of the suspect IMP (if response pattern is previously known).
- Could be reasonably explained by the subject's clinical state or other modes of therapy administered to the subject.

# **Possibly Related:**

- Follows a reasonable temporal sequence from administration of the IMP.
- May follow a known response pattern to the suspect IMP (if response pattern is previously known).
- Could also be reasonably explained by the subject's clinical state or other modes of therapy administered to the subject.

# Related:

- Follows a reasonable temporal sequence from administration of the IMP.
- Could not be reasonably explained by the known characteristics of the subject's clinical state or any other modes of therapy administered to the subject.
- Is confirmed by improvement on stopping or slowing administration of the IMP, if applicable.

If an assessment is not provided, the event will be treated as Possibly Related for purposes of regulatory reporting.

# 9.2.6 Action Taken Following Adverse Events

For each reported AE and SAE, the Investigator must document the action taken according to the following criteria:

- No action taken
- Non-pharmacologic treatment added
- New drug therapy added
- IMP interrupted
- Discontinued from study
- New or prolonged hospitalization

#### 9.2.7 Outcome of Adverse Events

For each reported AE and SAE, the Investigator must document the outcome according to the following criteria:

- Resolved
- Ongoing
- Unknown
- Death

The appropriate AE or SAE report page will be updated once the outcome is determined. The Investigator will also ensure that additional follow-up information includes any supplemental data that may explain causality of the event(s).

For SAEs, new or updated information will be recorded on the originally completed SAE report, with all changes signed and dated by the Investigator or designee. The updated SAE report will then be signed by the Investigator and resubmitted to Mycovia Pharmaceuticals (or designee).

# 9.2.8 Other Reportable Events

Reports of overdose (with or without an AE), abuse, dependency, inadvertent or accidental exposure, pregnancy and unexpected therapeutic benefit should be forwarded to Mycovia Pharmaceuticals (or designee) in the same time frame as an SAE.

Overdose occurs when a subject is administered or has taken a dose substantially greater than the intended or scheduled dose specified by the protocol.

All pregnancies occurring from the time the subject takes their first dose of IMP through the last study visit (Week 48) must be followed for information regarding the course of pregnancy, delivery, and condition of the newborn. Follow-up should be provided by the Investigator to Mycovia Pharmaceuticals in a timely manner.

Ver. 6 U.S. Only, 01 October 2019

# 10 PHARMACOKINETIC ASSESSMENTS

# 10.1 Sample Collection and Handling

Blood samples for determination of VT-1161 plasma concentrations will be collected at visits specified in Schedule of Assessments and Procedures. Timing of samples will be with respect to the day and time study drug is administered. The initial PK sample must be drawn prior to the first dose of study drug (placebo/VT-1161). The date and time of each PK sample will be recorded in the CRF. PK samples should be stored frozen at -20°C or colder. Detailed shipping instructions will be provided in the lab manual.

# **10.2 Analytical Procedures**

Plasma samples will be analyzed to determine concentrations of VT-1161 using a validated, specific and sensitive liquid chromatography/tandem mass spectrometry method at a bioanalytical laboratory designated by Mycovia Pharmaceuticals. Pharmacokinetic samples may be retained for future analysis of the metabolite profile for a period of up to 15 years, after which time the samples will be destroyed.

# 10.3 Pharmacokinetic Parameters

For subjects in the VT-1161 treatment arm, VT-1161 concentrations will be presented by visit with descriptive statistics. The PK data may be used in a cross-population PK analysis that may be presented in a separate report.

# 11 STUDY TERMINATION AND SUBJECT DISCONTINUATION

# 11.1 Screening/Baseline Failures

Subjects who sign and date the informed consent form or assent (for those ages 12 to 17) but fail to be randomized are defined as screen failures. Site personnel should maintain documentation for all subjects who sign an informed consent or assent.

# 11.2 Subject Withdrawal or Premature Discontinuation from the Study

The following actions must be taken in relation to a subject who fails to attend the clinic for a required study visit:

- The site must attempt to contact the subject and reschedule the missed visit as soon as possible.
- The site must counsel the subject on the importance of maintaining the assigned visit schedule and ascertain whether or not the subject wishes to and/or should continue in the study.
- In cases where the subject is deemed 'lost to follow-up', the Investigator or designee must
  make every effort to regain contact with the subject (e.g., multiple telephone calls on
  various dates/time, a certified letter to the subject's last known mailing address, or
  equivalent methods). These contact attempts should be documented in the subject's source
  documents.
- Should the subject continue to be unreachable, only then will they be considered to have withdrawn from the study with a primary reason of "Lost to Follow-up".

A subject may withdraw from the study at any time at his/her own request, or may be withdrawn at any time at the discretion of the Investigator for safety, behavioral, or administrative reasons. If a subject withdraws from the study, he/she may request destruction of any laboratory samples taken, and the Investigator must document this in the site study records and communicate this request to Mycovia Pharmaceuticals.

A subject may be withdrawn due to lack of tolerability or safety concerns, including study drug-related AEs or development of clinically-significant study drug-related laboratory abnormalities. If a subject is withdrawn from treatment, the subject must be followed clinically until the event is resolved or deemed stable. A subject must be discontinued from the study

drug if ALT or/and AST is  $> 5 \times$  the upper limit of normal (ULN) or ALT or/and AST is  $> 3 \times$  ULN and serum total bilirubin is > 2.0 ULN. (Refer to 7.3).

Subject who want to discontinue from the study should be encouraged to remain in the study for all remaining visits through Week 48 for safety and efficacy assessments. All subjects who do discontinue early from the study should have all EOS procedures performed on the day of discontinuation.

If a subject is prematurely discontinued from study treatment for any reason other than withdrawal of consent, the Investigator (or designee) should request that the subject continues to participate in the study, attending all remaining visits in accordance with the Schedule of Assessments and Procedures. Subjects who prematurely discontinue study medication, but remain in the study, may be treated according to the standard local practice. If the subject does not agree to remain in the study, the Investigator (or designee) must make every effort to perform the early withdrawal visit/EOS visit procedures.

# 11.3 Subject and Study Completion

A completed subject is one who has completed all visits, Screening through Week 48 (EOS), as defined in the Schedule of Assessments and Procedures. Study completion is defined as when the last subject has completed their last study visit.

Ver. 6 U.S. Only, 01 October 2019

# 11.4 Premature Study Termination

Reasons for discontinuation of the study at the investigative site may include, but are not limited to, the following:

- The incidence or severity of AEs in the study indicates a potential health hazard to subjects.
- Subject wishes to withdraw consent for reasons other than an AE.
- Subject non-compliance or unwillingness to comply with the procedures required by the protocol.
- Investigator request to withdraw from participation.
- Sponsor decision.
- Serious and/or persistent non-compliance by the Investigator with the protocol, the clinical research agreement, the Form Food and Drug Administration 1572, or applicable regulatory guidelines in conducting the study.
- Decision by the IRB/IEC to terminate or suspend approval for the investigation or the Investigator.
- Investigator fraud (altered data, omitted data, or manufactured data).

# 12 STATISTICAL ANALYSIS

The SAP will provide a detailed description of the proposed data analysis methods and procedures. The SAP was drafted and submitted to regulatory bodies prior to the start of the study and will be finalized before 50% of subjects are enrolled. The SAP contains all the details for the analysis of the primary and secondary endpoints as well as the sensitivity analyses planned for all endpoints. The additions to the SAP since that initial submission include additional sensitivity analyses,

The handling of missing data is explained in detail in the SAP including the descriptions of the sensitivity analyses that will be performed for each endpoint in order to assess the impact of the handling of the missing data on the results. Any deviation from the analyses outlined in the protocol will be described in the SAP. The primary statistical objective of this study is to determine if there are differences in the proportions of subjects with one or more culture-verified acute VVC episodes with signs and symptoms of  $\geq 3$  during the Maintenance (post randomization through Week 48) in those receiving VT-1161 compared to those receiving placebo during the Maintenance Phase.

# 12.1 Determination of Sample Size

For the primary efficacy endpoint determination, a sample size of 68 active subjects and 34 placebo subjects provides at least 95% power to detect a treatment difference of 35% between the VT-1161 treatment group and the placebo treatment group in percentage of subjects with one or more culture-verified acute VVC episodes during the Maintenance Phase (post randomization through Week 48). (PASS 2008: Fisher's exact test, two-sided alpha = 0.05, and assuming 50% of placebo subjects have recurrence). Based on an estimated 20% discontinuation rate, approximately 128 total subjects (85 active, 43 placebo) will be necessary for randomization to arrive at approximately 102 evaluable subjects.

The placebo rate was based on data generated in the Phase 2b RVVC study; the primary efficacy outcome measure in this study was the proportion of subjects with one or more culture-verified acute VVC episodes during the Maintenance Phase through Week 48 of the study in the ITT population (all randomized subjects). Culture-verified acute VVC was defined as a positive fungal culture for Candida species associated with a total signs and symptoms score of  $\geq 3$ . The proportion of subjects with one or more culture-verified acute VVC episodes through Week 48 was lower in the VT-1161 dosing regimens (0-7%) compared with the placebo group (52.2%). This difference was statistically significant in all VT-1161 treatment groups compared with placebo (p<0.0001). When powering the VMT-VT-1161-CL-012 study, it was determined that a separation of at least 35% between the treatment groups would be a

clinically meaningful separation. Thus, the sample size was powered to pick up at least a 35% separation between the treatment groups.

While 102 total subjects will provide more than 90% power to detect reasonable differences between treatment groups in most of the pre-specified key secondary endpoints a sample size of 160 active subjects and 80 placebo subjects is needed to provide 80% power to detect a treatment difference of 3.9 between the VT-1161 treatment group and the placebo group in the change from screening through Week 48 in the SF-36 MCS with a standard deviation of 10 points. (PASS 2008: two-sample t-test, alpha = 0.05). Therefore, with the expected discontinuation rate, approximately 300 subjects will be necessary for randomization to arrive at approximately 240 evaluable subjects. Approximately 600 subjects will be screened to randomize approximately 300 subjects that would meet the inclusion/ exclusion criteria.

# 12.2 Analysis Populations

ITT Population: All randomized subjects.

Safety Population: All randomized subjects who received at least 1 dose of IMP.

PP Population: All randomized subjects who had the following:

- Had no deviations to inclusion/exclusion criteria that could impact treatment outcome.
- Were compliant with the assigned study treatment, defined as  $\ge 80\%$  compliance during the daily dosing phase and  $\ge 50\%$  compliance during the weekly dosing phase.
- Had the Week 48 visit completed within the acceptable time window ( $\pm 14$  days).
- Had no major protocol violations that would impact treatment outcome.

Modified ITT: All randomized subjects who had the following:

- Positive KOH or Gram stain at Screening.
- Positive culture at Screening.
- Negative culture at Baseline.

All statistical populations will be defined in the SAP.

# 12.3 Demographic and Baseline Characteristic Analyses

Subject disposition, demographics, baseline characteristics and study drug exposure will be summarized by treatment group.

# 12.4 Efficacy Analyses

Clinical and mycological assessments will be conducted as outlined in the Schedule of Assessments and Procedures.

The primary efficacy outcome measure is the proportion of subjects with one or more culture-verified acute VVC episodes during the Maintenance Phase (post randomization through Week 48 of the study) in the ITT population. An acute VVC episode in the Maintenance Phase (considered a recurrent episode) is defined as a positive culture for Candida species and a clinical signs and symptoms score of  $\geq 3$ .

The primary method of analysis is a Chi-square test for active treatment versus placebo based on the ITT population.

The number and percentage of subjects with one or more culture-verified acute VVC episodes with signs and symptoms of  $\geq 3$  post randomization through Week 48 will be summarized across treatment groups including a 95% exact confidence interval and odds ratio. The percentages will also be plotted by treatment group.

The key secondary efficacy outcome measures include the following:

- Time to first recurrence of a culture-verified acute VVC episode with signs and symptoms score ≥3 during the Maintenance Phase.
- The proportion of subjects with at least one positive culture for Candida species during the Maintenance Phase.
- The proportion of subjects with at least one culture-verified acute VVC episode with signs and symptoms ≥3 post randomization through Week 24.
- Change from Screening through Week 48 in the SF-36 patient mental component score (MCS).

• Change from Screening through Week 48 in the SF-36 patient reported outcome survey total score.

Subjects who want to discontinue from the study should be encouraged to remain in the study for all remaining visits through Week 48 for safety and efficacy assessments. Subjects who do discontinue early from the study should have all Week 48/EOS assessments performed on the day of discontinuation.

Every effort will be made to obtain required data at each scheduled evaluation from all subjects who have been randomized, including those who discontinue the study prior to the EOS Week 48 visit.

For scheduled visits where the investigator's assessment of clinical signs and symptoms or the culture result is missing, missing values will be imputed using the method of multiple imputation. For subjects who discontinue the study early and have missing assessments for all visits after discontinuation, the missing values for the expected scheduled visits will be imputed using the method of multiple imputation. The missing values will be imputed using the following auxiliary information: region, treatment, baseline BMI, baseline age, ethnicity, and visit. The procedure PROC MI in SAS will be used to generate 10 possible imputed datasets. Using these multiple imputation datasets, determination of meeting the primary endpoint of a culture-verified acute VVC episode during the Maintenance Phase will be Subjects with a culture-verified acute VVC episode at any point from post randomization through Week 48 (including unscheduled visits) will be counted as having an episode when calculating the primary endpoint. The multiple datasets containing the primary endpoint will be analyzed using a Chi-square test and the results will be combined using PROC MIANALYZE to obtain an inferential result. Sensitivity analyses will be performed for the primary endpoint to assess the impact of missing/censored data on the results using different time to event and censoring calculations. Further details on the steps of these analyses are presented in the VMT-VT-1161-CL-012 SAP.

# 12.5 Safety Analyses

To meet the safety dataset requirement, approximately 600 subjects will be screened to randomize approximately 300 subjects that would meet the inclusion/ exclusion criteria. Assuming a 20% discontinuation rate, it is expected that approximately 240 subjects will complete the study.

All subjects who receive at least one dose of IMP will be included in the safety analyses. Subjects will be analyzed as per the treatment they receive. The number and percentage of subjects having TEAEs will be tabulated by system organ class and preferred term with a breakdown by treatment group. Mean changes from pre-treatment in vital signs, ECGs, and clinical laboratory variables will be summarized by treatment group.

AEs will be collected from the date of the first dose of fluconazole through Week 48 (EOS). Physical examination findings, vital signs, ECGs and safety laboratory tests (hematology and chemistry) will be obtained throughout the study as outlined in the Schedule of Assessments and Procedures. All concomitant medications taken during the period from 30 days prior to Screening through the Week 48 (EOS) visit will be recorded in the CRF. Pertinent and all major medical conditions will be recorded on the Medical History CRF.

For subjects discontinuing early from the study, every effort will be made for all EOS procedures to be performed as outlined in the Schedule of Assessments and Procedures. AEs will be coded with the Medical Dictionary for Regulatory Activities (MedDRA®) version 21 dictionary, or higher. The number and percentage of subjects having treatment-emergent AEs will be tabulated by system organ class and MedDRA® preferred term with a breakdown by treatment group. Mean changes from pre-treatment in vital signs, ECG, and clinical laboratory variables will be summarized by treatment group. The AE profile will be characterized with severity and relationship to IMP. SAEs and AEs resulting in discontinuation of IMP will be identified.

Treatment-emergent abnormal laboratory test results will be identified. Treatment-emergent abnormal laboratory tests results are those in which the baseline value is within normal laboratory limits and at least 1 post-baseline value is outside normal laboratory limits. Baseline will be defined as the last clinical laboratory result obtained before the first dose of IMP. Per protocol, the baseline for laboratory values should be obtained at the Day 1 (Baseline) visit.

Change from baseline to the minimum, maximum, and final vital sign value after first dosing will be summarized descriptively.

ECG measurements will include heart rate, QT interval, QTc interval, PR interval, and QRS interval. Baseline for ECG measurements is defined per protocol as the value pre-dosing at the Day 1 (Baseline) visit. Change from baseline will be summarized descriptively at each scheduled evaluation. Subjects with clinically significant changes in ECG rhythm or waveform will be identified. Subjects who meet each of the following criteria from ICH Guideline E14 "Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic

Potential for Non-Antiarrhythmic Drugs" (October 2005) for QT and corrected QT intervals will be identified.

- QT or Fridericia-corrected QT >450 msec
- QT or Fridericia-corrected QT >480 msec
- QT or Fridericia-corrected QT >500 msec
- QT or Fridericia-corrected QT increases from baseline by at least 30 msec
- QT or Fridericia-corrected QT increases from baseline by at least 60 msec

# 12.6 Pharmacokinetic Analyses

For subjects in the VT-1161 treatment arms, VT-1161 concentrations will be presented by visit with descriptive statistics. The PK data may be used in a cross-population PK analysis that may be presented in a separate report.

# 12.7 Patient Reported Outcome

Validated Patient Reported Outcomes, SF-36<sup>TM</sup>, EQ-5D-3L or EQ-5D-Y (for ages 12 to 17), WPAI:SHP, and PHQ-9 Health Surveys, will be administered for all regions participating in this study (see Appendices D, E, F, G, and H, respectively). Data will be reviewed for overall quality of life changes from the Screening visit to the Week 48 visit. For US only, questions regarding RVVC history will be administered at Screening using the RVVC History Questionnaire (see Appendix I) to collect information on the disease, diagnosis, and treatment profile for the subjects enrolled in the study.

Ver. 6 U.S. Only, 01 October 2019

# 13 CLINICAL STUDY ADMINISTRATION/STUDY GOVERNANCE CONSIDERATIONS

# 13.1 Ethical Conduct of Study

The study will be conducted in accordance with ICH Good Clinical Practice (GCP), all applicable subject privacy requirements, the guiding principles of the current version of the Declaration of Helsinki, and applicable country-specific regulatory requirements. This includes, but is not limited to, the following:

- IRB/IEC review and favorable opinion/approval of the study protocol and amendments, as applicable, informed consent and assent (for those ages 12 to 17) documents, and investigational brochure.
- Signed informed consent form or assent (for those ages 12 to 17) to be obtained for each subject before participation in the study (and for amendments as applicable).
- Investigator reporting requirements (e.g., continuing reviews, reporting of AEs/SAEs/protocol deviations to the IRB/IEC).
- If any documents are translated, an official certificate of translation must be maintained.

# 13.2 Informed Consent and Assent

Written informed consent or assent (for ages 12 to 17) must be obtained from all subjects. The informed consent or assent document must be signed and dated prior to the initiation of study-related tests and prior to administration of fluconazole. The original signed informed consent or assent for each participating subject shall be filed with records kept by the Investigator(s). A copy of the informed consent or assent document must be provided to the subject. If applicable, it will be provided in a certified translation of the local language.

# 13.3 Quality Control (Study Monitoring)

In accordance with applicable regulations, including GCP, the representative(s) or the designated clinical study monitor of Mycovia Pharmaceuticals will contact the site staff prior to the start of the study to review the protocol, study requirements, and their responsibilities to satisfy regulatory, ethical, and Mycovia Pharmaceuticals' requirements. When reviewing the data collection procedures, the discussion will also include identification, agreement, and documentation of data items that will serve as the source document.

Mycovia Pharmaceuticals representative(s) or the designated clinical study monitor will monitor the study and site activity at regular intervals throughout the study to verify the following:

- Data are authentic, accurate, and complete.
- Safety and rights of subjects are being protected.
- Study is conducted in accordance with the currently approved protocol and any other study agreements, GCP, and all applicable regulatory requirements.

The Investigator and the head of the medical institution (where applicable) agrees to allow the clinical study monitor direct access to all relevant documents.

Relevant documents or source documents are defined as the results of original observations and activities of a clinical investigation. Source documents may include, but are not limited to, study progress notes, e-mail correspondences, computer printouts, laboratory data, and drug accountability records.

# 13.4 Quality Assurance

To ensure compliance with GCP and all applicable regulatory requirements, Mycovia Pharmaceuticals may conduct a quality assurance assessment and/or audit of the site records, and the regulatory agencies may conduct a regulatory inspection at any time during or after the completion of the study. In the event of an assessment, audit or inspection, the Investigator (and institution) must agree to grant the advisor(s), auditor(s), and inspector(s) direct access to all relevant documents and to allocate their time and the time of their staff to discuss the conduct of the study, any findings/relevant issues, and to implement any corrective and/or preventative actions to address any findings/issues identified.

# 13.5 Compliance with Standards of Medical Research/ Deviations

This protocol will be conducted in accordance with the applicable ICH guidelines and GCP. Any instance of non-compliance with the protocol will result in a documented deviation. If a change is deemed necessary to protect the safety, rights or welfare of a subject, Mycovia Pharmaceuticals and IRB/IEC should be notified as soon as possible and preferably prior to introducing the deviation. Major deviations are defined as, but not limited to, the following:

• Subjects who did not meet entry criteria.

- Subjects who developed withdrawal criteria during the study but were not withdrawn.
- Subjects who received the wrong treatment or incorrect dose.
- Subjects who were <80% IMP compliant in the Induction Phase or <50% IMP compliant in the Maintenance Phase.
- Subjects who received an excluded concomitant medication or treatment.

# 13.6 Data Management

Electronic case report forms (eCRFs) will be used to capture study results and data. The study coordinator or other authorized site study personnel will transcribe data from source documents into the eCRFs. All eCRFs will be reviewed and source verified by the clinical study monitor during periodic site visits, and the clinical study monitor will ensure that all data in the eCRF are correct and complete. Prior to or between visits, the Medical Monitor or clinical study monitor may request copies of the eCRFs for preliminary medical review. Once the eCRFs are complete and source verified, the Investigator must sign and date all required pages, verifying the accuracy of all data contained within the eCRF.

Training will be provided for the Electronic Data Capture (EDC) system. All personnel using the EDC system must have the appropriate education, training, and experience, or any combination thereof. The Investigator will be provided with SOPs (contained in the Study Procedures Manual or a vendor-specific SOP) on the use of the EDC system. Documentation for employee education, training, and previous experience that pertains to the EDC system must be present in the Investigator files.

If electronic data systems other than those provided and maintained by Mycovia Pharmaceuticals are used for documentation and data capture, the Investigator must ensure that the systems are validated and ensure regular data back-up.

The eCRF will be signed by the Principal Investigator listed on the Food and Drug Administration (FDA) 1572 form. It is the responsibility of the Principal Investigator to ensure the eCRFs are completed and submitted to Mycovia Pharmaceuticals (or designee) in an accurate and timely manner. The processing of eCRFs will include an audit trail (to include changes made, reason for change, date of change, and person making change). At the completion of the study, the Investigator will be provided with a final copy of the eCRFs for their subjects. Mycovia Pharmaceuticals will be provided with a final copy of all subject eCRF data for the study.

Management of clinical data will be performed in accordance with applicable Mycovia Pharmaceuticals standards and data cleaning procedures to ensure the integrity of the data (e.g., removing errors and inconsistencies in the data). AEs and concomitant medications will be coded using MedDRA®. Electronic CRFs (including queries and audit trails) will be retained by the Mycovia Pharmaceuticals and copies will be sent to the Investigator to maintain as the Investigator copy.

# 13.7 Study and Site Closure

Upon completion or premature discontinuation of the study, the representative (or designated clinical study monitor) of Mycovia Pharmaceuticals will conduct site closure activities with the Investigator or site staff, as appropriate, in accordance with applicable regulations including GCP. Mycovia Pharmaceuticals reserves the right to temporarily suspend or prematurely discontinue this study at any time for reasons including, but not limited to, safety or ethical issues or severe non-compliance. For multicenter studies, this can occur at 1 or more or at all sites. If the Sponsor determines such action is needed, Mycovia Pharmaceuticals will discuss the reasons for taking such action with the Investigator or head of the medical institution (where applicable). When feasible, Mycovia Pharmaceuticals will provide advance notification to the Investigator or head of the medical institution (where applicable) of the impending action. If the study is suspended or prematurely discontinued for safety reasons, Mycovia Pharmaceuticals will promptly inform all Investigators, heads of medical institutions (where applicable), and/or institutions conducting the study. Mycovia Pharmaceuticals will also promptly inform the relevant regulatory authorities of the suspension or premature discontinuation of the study and the reason(s) for the action. If required by applicable regulations, the Investigator must inform the IRB/IEC promptly and provide the reason(s) for the suspension or premature discontinuation.

# 13.8 Records Retention

Following closure of the study, the Investigator must maintain all site study records (except for those required by local regulations to be maintained elsewhere), in a safe and secure location. The records must be maintained to allow easy and timely retrieval when needed (e.g., for a Mycovia Pharmaceuticals audit or regulatory inspection) and must be available for review in conjunction with the assessment of the facility, supporting systems, and relevant site staff. When permitted by local laws/regulations or institutional policy, some or all of the records can be maintained in a format other than hard copy (e.g., microfiche, scanned, electronic); however, caution needs to be exercised before such action is taken. The Investigator must ensure that all reproductions are legible and are a true and accurate copy of the original and

meet accessibility and retrieval standards, including regenerating a hard copy, if required. Furthermore, the Investigator must ensure there is an acceptable back-up of these reproductions and that an acceptable quality control process exists for making these reproductions.

Investigators are required to retain essential documents pertaining to the conduct of this study for at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product, per ICH guidelines. The minimum retention time will meet the strictest standard applicable to that site for the study, as dictated by any institutional requirements, local laws or regulations, or Mycovia Pharmaceuticals' standards/procedures. The Investigator must notify Mycovia Pharmaceuticals of any changes to the archival arrangements, including, but not limited to, archival at an off-site facility or transfer of ownership of the records in the event the Investigator is no longer associated with the site.

# 13.9 Disclosure of Data

The Investigator agrees by his/her participation that the results of this study may be used for submission to national and/or international registration and supervising authorities. If required, these authorities will be provided with the names of Investigators, their addresses, qualifications, and extent of involvement. It is understood that the Investigator is required to provide Mycovia Pharmaceuticals with all study data, complete reports, and access to all study records.

Data generated by this study must be available for inspection by the United States FDA and other regulatory authorities, by Mycovia Pharmaceuticals, and the IRB/IEC as appropriate. At a subject's request, medical information may be given to his or her personal physician or other appropriate medical personnel responsible for his or her welfare. Subject medical information obtained during this study is confidential and disclosure to third parties other than those noted above is prohibited.

# 13.10 Financial Disclosure

The United States FDA Financial Disclosure by Clinical Investigators (21 Code of Federal Regulations 54) regulations require Sponsors to obtain certain financial information from Investigators participating in covered clinical studies; each Principal Investigator and Sub-Investigator is required to provide the required financial information and to promptly update Mycovia Pharmaceuticals with any relevant changes to their financial information throughout the course of the clinical study and for up to 1 year after its completion. This rule

applies to all Investigators and Sub-Investigators participating in covered clinical studies to be submitted to the FDA in support of an application for market approval.

# **13.11 Publication Policy**

The publication policy is outlined in the Clinical Trial Agreement.

# **13.12** Confidentiality

Confidentiality is outlined in the Clinical Trial Agreement.

#### 13.12.1 Data

All information about the nature of the proposed investigation provided by Mycovia Pharmaceuticals or the designated clinical study monitor to the Investigator (with the exception of information required by law or regulations to be disclosed to the IRB/IEC, the subject, or the appropriate regulatory authority) must be kept in confidence by the Investigator.

# 13.12.2 Subject Anonymity

The anonymity of participating subjects must be maintained. Subjects will be identified by an assigned subject number on CRFs and other documents retrieved from the site or sent to the designated clinical study monitor, Sponsor, regulatory agencies, or central laboratories/reviewers. Documents that identify the subject (e.g., the signed informed consent document, subject identification record) must be maintained in strict confidence by the Investigator, except to the extent necessary to allow auditing by the appropriate regulatory authority, the clinical study monitor, or Mycovia Pharmaceuticals representatives.

# 14 REFERENCES

Barousse, M., et al. Vaginal yeast 105icromole105a105, prevalence of vaginitis, and associated local immunity in adolescents. Sexually Transmitted Infections, 2004;80(1):48-53.

Bates DW and Yu DT. Clinical impact of drug-drug interactions with systemic azole antifungals. Drugs Today 2003; 39: 801-813.

Blostein, F., et al. Recurrent vulvovaginal candidiasis. Annals of Epidemiology, 2017: In press.

Diflucan® 150 Capsules [Summary of Product Characteristics]. Pfizer Limited. Sandwich, UK. Accessed through http://www.medicines.org.uk/emc/medicine/1458/spc. Last updated 19-May-2017.

Eschenbach DA. Chronic Vulvovaginal Candidiasis. New Engl J Med 2004; 351: 851-852.

Fidel, P., Jr. and J. Sobel. Host defense against vaginal candidiasis. Candida and candidiasis, ed. R. Calderone. Washington, D.C.: ASM Press. 2002, 193-209.

Foxman B, Muraglia R, Dietz JP, et al. Prevelence of recurrent Vulvovaginal Candidiasis in 5 European countries and the United States: results from an internet panel survey. Am Soc of Colposcopy and Cervical Path 2013; 17(3): 340-345.

Garvey EP, Fidel PL, Lilly EA, et al. The clinical antifungal agent VT-1161 is orally efficacious in a murine model of C. albicans vaginitis. Presented at the 11<sup>th</sup> American Society for Microbiology Conference on Candida and Candidiasis, San Francisco, CA. Abstract #33C (2012).

Goncalves B, Ferreira C, Alves CT, et al. Vulvovaginal candidiasis: epidemiology, microbiology and risk factors. Crit Rev Microbiol 2016; 42(2): 905-927.

Joishy, M., et al., Do we need to treat vulvovaginitis in prepubertal girls? British Medical Journal, 2005;330(7484):186-188.

Pfizer, I. Diflucan®, fluconazole tablet, <a href="https://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?setid=f694c617-3383-416c-91b6-b94fda371204">https://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?setid=f694c617-3383-416c-91b6-b94fda371204</a> (2017).

Sobel JD. Recurrent vulvovaginal candidiasis. Am J Obstet Gynecol. 2016 (1):6.

Sobel JD, Wiesenfeld HC, Martens M, et al. Maintenance fluconazole therapy for recurrent Vulvovaginal Candidiasis. New Engl J Med 2004; 351:876-883.

Sobel JD. Vulvovaginal Candidosis. Lancet 2007; 369:1961-1971.

VT-1161 Investigational Brochure, v005. Durham, NC. Mycovia Pharmaceuticals Inc. (2017).

Yoshida Y. Cytochrome P450 of fungi: primary target for azole antifungal agents. Curr Top Med Mycol 1988; 2: 388-418.

Zarn JA, Bruschweiler BJ, Schlatter JR. Azole fungicides affect mammalian steroidogenesis by inhibiting sterol  $14\alpha$ -demethylase and aromatase. Env Health Pers 2003; 111: 255-261.

# **APPENDICES**
Ver. 6 U.S. Only, 01 October 2019

# Appendix A. Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Table (Draft November 2007) Modified for Use in VMT-VT-1161-CL-012 Study

### **ABBREVIATIONS:** Abbreviations utilized in the Table:

ULN = Upper Limit of Normal LLN = Lower Limit of Normal

Rx = Therapy Req = Required
Mod = Moderate IV = Intravenous
ADL = Activities of Daily Living Dec = Decreased

#### ESTIMATING SEVERITY GRADE

For abnormalities NOT found elsewhere in the Toxicity Tables use the scale below to estimate grade of severity:

**GRADE 1** Mild: Transient or mild discomfort (<48 hours); no medical intervention/therapy required

**GRADE 2 Moderate**: Mild to moderate limitation in activity – some assistance may be needed; no or minimal medical intervention/therapy required

**GRADE 3** Severe: Marked limitation in activity, some assistance usually required; medical intervention/therapy required, hospitalizations possible.

**GRADE 4 Life-threatening**: Extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or hospice care probable

### **SERIOUS OR LIFE-THREATENING AES**

ANY clinical event deemed by the clinician to be serious or life-threatening should be considered a Grade 4 event.

### **LABORATORY RANGES**

Where discrepancies in the ULN and LLN of laboratory ranges occur between those included in this document and those of the laboratory that performs the assays, the values provided by the laboratory will be used for assignment of severity grade.

<sup>\*</sup>This toxicity table is applicable for subjects ages 12-17 years of age.

| HEMATOLOGY | | | | * |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hemoglobin | 9.5 - 10.5 gm/dL | 8.0 - 9.4 gm/dL | 6.5 - 7.9 gm/dL | < 6.5 gm/dL |
| <u> </u> | 5.9 – 6.5 mmol/L | 5.0 - 5.8 mmol/L | 4.0 – 4.9 mmol/L | < 4.0 mmol/L |
| Absolute Neutrophil | $1000 - 1500 / \text{mm}^3$ | 750 – 999/mm <sup>3</sup> | $500 - 749 \text{/mm}^3$ | <500/mm <sup>3</sup> |
| Count | Colores July Colors positively date | SERVINE INCOME. | ceamores as consistent unos | |
| Platelets | 75,000 - | 50,000 - | 20,000 - | <20,000/mm <sup>3</sup> |
| | 99,999/mm <sup>3</sup> | 74,999/mm <sup>3</sup> | 49,999/mm <sup>3</sup> | |
| WBCs | 11,000 - 13,000/ | 13,000 - 15,000 | 15,000 - | >30,000 or <1,000 |
| 28 | $\mathrm{mm}^3$ | $/\mathrm{mm}^3$ | $30,000/\text{mm}^3$ | $\mathrm{mm}^3$ |
| % Polymorphonuclear | >80% | 90 – 95% | >95% | |
| Leukocytes + Band | | | | |
| Cells | | | | |
| Activated Partial | $1.01 - 1.66 \times ULN$ | $1.67 - 2.33 \times ULN$ | $2.34 - 3 \times ULN$ | $> 3 \times ULN$ |
| Thromboplastin | | | | |
| (APTT) | | | | |
| CHEMISTRIES | | | T | |
| Marine and a second and a second and a second and | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyponatremia | 130 – 135 mEq/L | 123 – 129 mEq/L | 116 – 122 mEq/L | < 116 mEq/L or |
| | or mmol/L | or mmol/L | or mmol/L | mmol/L OR |
| | | | | abnormal sodium |
| | | | | with mental status |
| · • | 116 150 5 7 | 4.54 4.55 75 75 | 1.50 1.55 E /T | changes or seizures |
| Hypernatremia | 146 – 150 mEq/L | 151 – 157 mEq/L | 158 – 165 mEq/L | > 165 mEq/L or |
| | or mmol/L | or mmol/L | or mmol/L | mmol/L OR |
| | | | | abnormal sodium with mental status |
| | | | | 727 |
| Hypokalemia | 3.0 – 3.4 mEq/L or | 2.5 – 2.9 mEq/L or | 2.0 – 2.4 mEq/L or | changes or seizures<br>< 2.0 mEq/L or |
| пуроканиа | mmol/L | mmol/L | mmol/L OR | mmol/L OR |
| | IIIIIOI/L | IIIIIOD L | intensive | abnormal |
| | | | replacement | potassium with |
| | | | therapy or | paresis, ileus or |
| | | | hospitalization | life-threatening |
| | | | required | arrhythmia |
| Hyperkalemia | 5.6 - 6.0 mEq/L or | 6.1 - 6.5 mEq/L or | 6.6 - 7.0 mEq/l or | >7.0 mEq/L or |
| | mmol/L | mmol/L | mmol/L | mmol/L OR |
| | | | | abnormal |
| | | | | potassium with life- |
| | | | | threatening |
| ** | | | | arrhythmia |
| Hypoglycemia | 55 – 64 mg/dL | 40 - 54 mg/dL | 30 – 39 mg/dL | <30 mg/dL or |
| | | | | abnormal glucose |
| | | | | with mental status |
| | | | | changes or coma |

Protocol VMT-VT-1161-CL-012

| | | Service California Marco | Inches and the second | Tr. 100 Parks |
|---|---|---|---|---|
| | 3.1 - 3.6 mmol/L | 2.2 - 3.0 mmol/L | 1.7 – 2.2 mmol/L | <1.7 mmol/L or |
| | | | | abnormal glucose |
| | | | | with mental status |
| | | | | changes or coma |
| Hyperglycemia (non- | 116 – 160 mg/dL | 161-250 mg/dL | 251 - 500 mg/dL | > 500 mg/dL or |
| fasting and no prior | 110 100 1119 022 | 101 200 mg uz | 201 DOO ING GE | abnormal glucose |
| diabetes) | | | | with ketoacidosis or |
| diabetes) | | | | seizures |
| | C 4 0 0 1/T | 0.0 10.0 1/7 | 100 000 1/7 | |
| | 6.4 - 8.9 mmol/L | 8.9 – 13.9 mmol/L | 13.9 – 27.8 mmol/L | |
| | | | | abnormal glucose |
| | | | | with ketoacidosis |
| | | | | or seizures |
| CHEMISTRIES | | | 7<br>2 | es es |
| 8 | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hypocalcemia | 8.4 - 7.8 mg/dL | 7.7 - 7.0 mg/dL | 6.9 - 6.1 mg/dL | < 6.1 mg/Dl or |
| (corrected for | | | | abnormal calcium |
| albumin) | | | | with life- |
| , | | | | threatening |
| | | | | arrhythmia or |
| | | | | tetany |
| | 2.10 1.04 | 1.02 1.75 | 1.74 1.60 mm = 1/T | |
| | 2.10 – 1.94 IIIII0I/L | 1.93 – 1.75 IIIIIOI/L | 1.74 – 1.60 mmol/L | |
| | | | | abnormal calcium |
| | | | | with life- |
| | | | | threatening |
| | | | | arrhythmia or |
| | | | | tetany |
| Hypercalcemia | 10.6 - 11.5 mg/dL | 11.6 - 12.5 mg/dL | 12.6 - 13.5 mg/dL | > 13.5 mg/dL or |
| (correct for albumin) | | | | abnormal calcium |
| | | | | with life- |
| | | | | threatening |
| | | | | arrhythmia |
| | 2.64 2.97 mm a1/I | 2.00 2.12 mm a1/T | 3.13 – 3.37 mmol/L | |
| | 2.04 - 2.8 / IIIIIOI/L | 2.88 - 5.12 HIIIIOI/L | 3.13 - 3.3 / HIIIOI/L | |
| | | | | abnormal calcium |
| | | | | with life- |
| | | | | threatening |
| st . | | | | arrhythmia |
| Hypomagnesemia | 1.4 - 1.2 mEq/L | 1.1 - 0.9 mEq/L | 0.8 - 0.6 mEq/L | < 0.6 mEq/L or |
| anticisis SSSS | | 525 | 107 | abnormal |
| | | | | magnesium with |
| | | | | life-threatening |
| | | | | arrhythmia |
| | 0.58 - 0.49 mmol/L | 0.48 - 0.37 mmol/L | 0.36 - 0.25 mmol/L | |
| | J IIIII D. D. | o.c. minor D | in the state of th | abnormal |
| | | | | magnesium with |
| | | | | life-threatening |
| 10 | | | | arrhythmia |

| | PRODUCE SINCE THE STATE OF THE | TANDON CONTROL WAS ASSESSED. | The second secon | 2 on on 12,000 on 12 |
|---|---|---|---|---|
| Hypophosphatemia | 2.0 - 2.4 mg/dL | 1.5 - 1.9 mg/dL or | 1.0 - 1.4 mg/dL | < 1.0 mg/dL or |
| 699, ATA 1091, 8 1099) | V700 | replacement Rx | intensive therapy or | abnormal |
| | | required | hospitalization | phosphate with life- |
| | | 1 | required | threatening |
| | | | required | arrhythmia |
| | 0.65 0.77 | 0.40 0.64 | 0.22 0.47 | |
| | 0.65 - 0.77 IIIIIIOI/L | 0.48 - 0.64 HIIII0I/L | 0.32 - 0.47 mmol/L | A STATE OF THE PARTY OF THE PAR |
| | | | | abnormal |
| | | | | phosphate with life- |
| | | | | threatening |
| 19 | | | | arrhythmia |
| Hyperbilirubinemia | 1.1 - < 1.25 x ULN | 1.25 - <1.5 x ULN | 1.5 – 1.75 x ULN | > 1.75 x ULN |
| (when accompanied by | | | | |
| any increase in other | | | | |
| liver function test) | | | | |
| Hyperbilirubinemia | 1.1 – <1.5 x ULN | 1.5 – <2.0 x ULN | 2.0 – 3.0 x ULN | > 3.0 x ULN |
| (when other liver | 1.1 \1.5 X OLIV | 1.5 \2.0 A OLIV | 2.0 J.0 A OLIV | J.O A OLIV |
| The second secon | | | | |
| function is in normal | | | | |
| range) | 105 05 1773 | 26 5 17737 | 5.1 10 THAT | . 10 11131 |
| BUN | 1.25 – 2.5 x ULN | 2.6 – 5 x ULN | 5.1 – 10 x ULN | > 10 x ULN |
| Hyperuricemia (uric | 7.5 - 10.0 mg/dL | 10.1 - 12.0 mg/dL | 12.1 – 15.0 mg/dL | >15.0 mg/dL |
| acid) | 446 – 594 μmol/L | 595 – 714 μmol/L | 715 – 892 μmol/L | >892 μmol/L |
| Creatinine | 1.1 – 1.5 x ULN | 1.6 - 3.0 x ULN | $3.1 - 6 \times ULN$ | > 6 x ULN or |
| | | | | dialysis required |
| ENZYMES | | | | |
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| 7 | TO A SHIP BOA DADGER OF HOLD | A COLUMN TO SECURE STATE OF THE SECURE STATE O | | Grade 4 |
| AST (SGOT) | 1.1 – <2.0 x ULN | 2.0 – <3.0 x ULN | 3.0 – 8.0 x ULN | > 8 x ULN |
| AST (SGOT)<br>ALT (SGPT) | 1.1 – <2.0 x ULN<br>1.1 – <2.0 x ULN | 2.0 – <3.0 x ULN<br>2.0 – <3.0 x ULN | 3.0 – 8.0 x ULN<br>3.0 – 8.0 x ULN | > 8 x ULN<br>> 8 x ULN |
| AST (SGOT)<br>ALT (SGPT)<br>Alkaline Phosphatase | 1.1 – <2.0 x ULN | 2.0 – <3.0 x ULN | 3.0 – 8.0 x ULN | > 8 x ULN |
| AST (SGOT)<br>ALT (SGPT) | 1.1 – <2.0 x ULN<br>1.1 – <2.0 x ULN<br>1.1 – <2.0 x ULN | 2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN | 3.0 - 8.0 x ULN<br>3.0 - 8.0 x ULN<br>3.0 - 8.0 x ULN | > 8 x ULN<br>> 8 x ULN<br>> 8 x ULN |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS | 1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>Grade 1 | 2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>Grade 2 | 3.0 - 8.0 x ULN<br>3.0 - 8.0 x ULN<br>3.0 - 8.0 x ULN<br>Grade 3 | > 8 x ULN<br>> 8 x ULN<br>> 8 x ULN<br>Grade 4 |
| AST (SGOT)<br>ALT (SGPT)<br>Alkaline Phosphatase | 1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>Grade 1<br>1+ or 200 mg - 1 | 2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>Grade 2<br>2-3+ or 1- 2 gm | 3.0 - 8.0 x ULN<br>3.0 - 8.0 x ULN<br>3.0 - 8.0 x ULN<br>Grade 3<br>4+ or 2-3.5 gm | > 8 x ULN<br>> 8 x ULN<br>> 8 x ULN<br>Grade 4<br>nephrotic syndrome |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS | 1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>Grade 1 | 2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>Grade 2 | 3.0 - 8.0 x ULN<br>3.0 - 8.0 x ULN<br>3.0 - 8.0 x ULN<br>Grade 3 | > 8 x ULN<br>> 8 x ULN<br>> 8 x ULN<br>Grade 4<br>nephrotic syndrome<br>or |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS Proteinuria | 1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>Grade 1<br>1+ or 200 mg - 1 | 2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>Grade 2<br>2-3+ or 1- 2 gm<br>loss/day | 3.0 – 8.0 x ULN<br>3.0 – 8.0 x ULN<br>3.0 – 8.0 x ULN<br>Grade 3<br>4+ or 2-3.5 gm<br>loss/day | > 8 x ULN<br>> 8 x ULN<br>> 8 x ULN<br>> 8 x ULN<br>Grade 4<br>nephrotic syndrome<br>or<br>> 3.5 gm loss/day |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS | 1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>Grade 1<br>1+ or 200 mg - 1 | 2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>Grade 2<br>2-3+ or 1- 2 gm | 3.0 - 8.0 x ULN<br>3.0 - 8.0 x ULN<br>3.0 - 8.0 x ULN<br>Grade 3<br>4+ or 2-3.5 gm | > 8 x ULN<br>> 8 x ULN<br>> 8 x ULN<br>Grade 4<br>nephrotic syndrome<br>or |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS Proteinuria | 1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>Grade 1<br>1+ or 200 mg - 1<br>gm loss/day | 2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>Grade 2<br>2-3+ or 1- 2 gm<br>loss/day<br>gross, no clots | 3.0 – 8.0 x ULN<br>3.0 – 8.0 x ULN<br>3.0 – 8.0 x ULN<br>Grade 3<br>4+ or 2-3.5 gm<br>loss/day<br>gross, with or | > 8 x ULN<br>> 8 x ULN<br>> 8 x ULN<br>> 8 x ULN<br>Grade 4<br>nephrotic syndrome<br>or<br>> 3.5 gm loss/day<br>obstructive or |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS Proteinuria | 1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>Grade 1<br>1+ or 200 mg - 1<br>gm loss/day | 2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>Grade 2<br>2-3+ or 1- 2 gm<br>loss/day | 3.0 – 8.0 x ULN<br>3.0 – 8.0 x ULN<br>3.0 – 8.0 x ULN<br>Grade 3<br>4+ or 2-3.5 gm<br>loss/day<br>gross, with or<br>without clots, OR | > 8 x ULN<br>> 8 x ULN<br>> 8 x ULN<br>> 8 x ULN<br>Grade 4<br>nephrotic syndrome<br>or<br>> 3.5 gm loss/day<br>obstructive or<br>required |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS Proteinuria Hematuria | 1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>Grade 1<br>1+ or 200 mg - 1<br>gm loss/day<br>microscopic only<br><10 rbc/hpf | 2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>Grade 2<br>2-3+ or 1- 2 gm<br>loss/day<br>gross, no clots | 3.0 – 8.0 x ULN<br>3.0 – 8.0 x ULN<br>3.0 – 8.0 x ULN<br>Grade 3<br>4+ or 2-3.5 gm<br>loss/day<br>gross, with or<br>without clots, OR | > 8 x ULN<br>> 8 x ULN<br>> 8 x ULN<br>> 8 x ULN<br>Grade 4<br>nephrotic syndrome<br>or<br>> 3.5 gm loss/day<br>obstructive or |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS Proteinuria | 1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>Grade 1<br>1+ or 200 mg - 1<br>gm loss/day<br>microscopic only<br><10 rbc/hpf | 2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>Grade 2<br>2-3+ or 1- 2 gm<br>loss/day<br>gross, no clots<br>>10 rbc/hpf | 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN Grade 3 4+ or 2-3.5 gm loss/day gross, with or without clots, OR red blood cell casts | > 8 x ULN > 8 x ULN > 8 x ULN > 8 x ULN Grade 4 nephrotic syndrome or > 3.5 gm loss/day obstructive or required transfusion |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS Proteinuria Hematuria CARDIOVASCULAR | 1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>Grade 1<br>1+ or 200 mg - 1<br>gm loss/day<br>microscopic only<br><10 rbc/hpf | 2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>Grade 2<br>2-3+ or 1- 2 gm<br>loss/day<br>gross, no clots<br>>10 rbc/hpf | 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN Grade 3 4+ or 2-3.5 gm loss/day gross, with or without clots, OR red blood cell casts Grade 3 | > 8 x ULN > 8 x ULN > 8 x ULN Say ULN Grade 4 nephrotic syndrome or > 3.5 gm loss/day obstructive or required transfusion Grade 4 |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS Proteinuria Hematuria | 1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>Grade 1<br>1+ or 200 mg - 1<br>gm loss/day<br>microscopic only<br><10 rbc/hpf | 2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>Grade 2<br>2-3+ or 1- 2 gm<br>loss/day<br>gross, no clots<br>>10 rbc/hpf | 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN Grade 3 4+ or 2-3.5 gm loss/day gross, with or without clots, OR red blood cell casts Grade 3 recurrent/persistent | > 8 x ULN > 8 x ULN > 8 x ULN Crade 4 nephrotic syndrome or > 3.5 gm loss/day obstructive or required transfusion Grade 4 unstable |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS Proteinuria Hematuria CARDIOVASCULAR | 1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>Grade 1<br>1+ or 200 mg - 1<br>gm loss/day<br>microscopic only<br><10 rbc/hpf | 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN Grade 2 2-3+ or 1- 2 gm loss/day gross, no clots >10 rbc/hpf Grade 2 asymptomatic, transient signs, no | 3.0 - 8.0 x ULN 3.0 - 8.0 x ULN 3.0 - 8.0 x ULN 3.0 - 8.0 x ULN Grade 3 4+ or 2-3.5 gm loss/day gross, with or without clots, OR red blood cell casts Grade 3 recurrent/persistent symptomatic Rx | > 8 x ULN > 8 x ULN > 8 x ULN > 8 x ULN Grade 4 nephrotic syndrome or > 3.5 gm loss/day obstructive or required transfusion Grade 4 unstable dysrythmia; |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS Proteinuria Hematuria CARDIOVASCULAR | 1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>Grade 1<br>1+ or 200 mg - 1<br>gm loss/day<br>microscopic only<br><10 rbc/hpf | 2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>2.0 - <3.0 x ULN<br>Grade 2<br>2-3+ or 1- 2 gm<br>loss/day<br>gross, no clots<br>>10 rbc/hpf | 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN Grade 3 4+ or 2-3.5 gm loss/day gross, with or without clots, OR red blood cell casts Grade 3 recurrent/persistent | > 8 x ULN > 8 x ULN > 8 x ULN > 8 x ULN Grade 4 nephrotic syndrome or > 3.5 gm loss/day obstructive or required transfusion Grade 4 unstable dysrythmia; hospitalization and |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS Proteinuria Hematuria CARDIOVASCULAR Cardiac Rhythm | 1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>1.1 - <2.0 x ULN<br>Grade 1<br>1+ or 200 mg - 1<br>gm loss/day<br>microscopic only<br><10 rbc/hpf | 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN Grade 2 2-3+ or 1- 2 gm loss/day gross, no clots >10 rbc/hpf Grade 2 asymptomatic, transient signs, no Rx required | 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN Grade 3 4+ or 2-3.5 gm loss/day gross, with or without clots, OR red blood cell casts Grade 3 recurrent/persistent symptomatic Rx required | > 8 x ULN > 8 x ULN > 8 x ULN Say ULN Grade 4 nephrotic syndrome or > 3.5 gm loss/day obstructive or required transfusion Grade 4 unstable dysrythmia; hospitalization and treatment required |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS Proteinuria Hematuria CARDIOVASCULAR | 1.1 - <2.0 x ULN 1.1 - <2.0 x ULN 1.1 - <2.0 x ULN 1.1 - <2.0 x ULN Grade 1 1+ or 200 mg - 1 gm loss/day microscopic only <10 rbc/hpf Grade 1 transient increase | 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN Grade 2 2-3+ or 1- 2 gm loss/day gross, no clots >10 rbc/hpf Grade 2 asymptomatic, transient signs, no Rx required recurrent, chronic | 3.0 - 8.0 x ULN 3.0 - 8.0 x ULN 3.0 - 8.0 x ULN 3.0 - 8.0 x ULN Grade 3 4+ or 2-3.5 gm loss/day gross, with or without clots, OR red blood cell casts Grade 3 recurrent/persistent symptomatic Rx required acute treatment | > 8 x ULN > 8 x ULN > 8 x ULN > 8 x ULN Grade 4 nephrotic syndrome or > 3.5 gm loss/day obstructive or required transfusion Grade 4 unstable dysrythmia; hospitalization and treatment required end organ damage |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS Proteinuria Hematuria CARDIOVASCULAR Cardiac Rhythm | 1.1 - <2.0 x ULN 1.1 - <2.0 x ULN 1.1 - <2.0 x ULN 1.1 - <2.0 x ULN Grade 1 1+ or 200 mg - 1 gm loss/day microscopic only <10 rbc/hpf Grade 1 transient increase > 20 mm/Hg; no | 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN Grade 2 2-3+ or 1- 2 gm loss/day gross, no clots >10 rbc/hpf Grade 2 asymptomatic, transient signs, no Rx required recurrent, chronic increase | 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN Grade 3 4+ or 2-3.5 gm loss/day gross, with or without clots, OR red blood cell casts Grade 3 recurrent/persistent symptomatic Rx required acute treatment required; outpatient | > 8 x ULN > 8 x ULN > 8 x ULN > 8 x ULN Grade 4 nephrotic syndrome or > 3.5 gm loss/day obstructive or required transfusion Grade 4 unstable dysrythmia; hospitalization and treatment required end organ damage or hospitalization |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS Proteinuria Hematuria CARDIOVASCULAR Cardiac Rhythm | 1.1 - <2.0 x ULN 1.1 - <2.0 x ULN 1.1 - <2.0 x ULN 1.1 - <2.0 x ULN Grade 1 1+ or 200 mg - 1 gm loss/day microscopic only <10 rbc/hpf Grade 1 transient increase | 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN Grade 2 2-3+ or 1- 2 gm loss/day gross, no clots >10 rbc/hpf Grade 2 asymptomatic, transient signs, no Rx required recurrent, chronic | 3.0 - 8.0 x ULN 3.0 - 8.0 x ULN 3.0 - 8.0 x ULN 3.0 - 8.0 x ULN Grade 3 4+ or 2-3.5 gm loss/day gross, with or without clots, OR red blood cell casts Grade 3 recurrent/persistent symptomatic Rx required acute treatment | > 8 x ULN > 8 x ULN > 8 x ULN > 8 x ULN Grade 4 nephrotic syndrome or > 3.5 gm loss/day obstructive or required transfusion Grade 4 unstable dysrythmia; hospitalization and treatment required end organ damage |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS Proteinuria Hematuria CARDIOVASCULAR Cardiac Rhythm | 1.1 - <2.0 x ULN 1.1 - <2.0 x ULN 1.1 - <2.0 x ULN 1.1 - <2.0 x ULN Grade 1 1+ or 200 mg - 1 gm loss/day microscopic only <10 rbc/hpf Grade 1 transient increase > 20 mm/Hg; no | 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN Grade 2 2-3+ or 1- 2 gm loss/day gross, no clots >10 rbc/hpf Grade 2 asymptomatic, transient signs, no Rx required recurrent, chronic increase | 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN Grade 3 4+ or 2-3.5 gm loss/day gross, with or without clots, OR red blood cell casts Grade 3 recurrent/persistent symptomatic Rx required acute treatment required; outpatient | > 8 x ULN > 8 x ULN > 8 x ULN > 8 x ULN Grade 4 nephrotic syndrome or > 3.5 gm loss/day obstructive or required transfusion Grade 4 unstable dysrythmia; hospitalization and treatment required end organ damage or hospitalization |
| AST (SGOT) ALT (SGPT) Alkaline Phosphatase URINALYSIS Proteinuria Hematuria CARDIOVASCULAR Cardiac Rhythm | 1.1 - <2.0 x ULN 1.1 - <2.0 x ULN 1.1 - <2.0 x ULN 1.1 - <2.0 x ULN Grade 1 1+ or 200 mg - 1 gm loss/day microscopic only <10 rbc/hpf Grade 1 transient increase > 20 mm/Hg; no | 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN 2.0 - <3.0 x ULN Grade 2 2-3+ or 1- 2 gm loss/day gross, no clots >10 rbc/hpf Grade 2 asymptomatic, transient signs, no Rx required recurrent, chronic increase > 20mm/Hg. | 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN 3.0 – 8.0 x ULN Grade 3 4+ or 2-3.5 gm loss/day gross, with or without clots, OR red blood cell casts Grade 3 recurrent/persistent symptomatic Rx required acute treatment required; outpatient treatment or | > 8 x ULN > 8 x ULN > 8 x ULN > 8 x ULN Grade 4 nephrotic syndrome or > 3.5 gm loss/day obstructive or required transfusion Grade 4 unstable dysrythmia; hospitalization and treatment required end organ damage or hospitalization |

| Hypotension Pericarditis | transient orthostatic<br>hypotension with<br>heart rate increased<br>by <20 beat/min or<br>decreased by <10<br>mm Hg systolic<br>BP, no treatment<br>required<br>minimal effusion | orthostatic hypotension or BP decreased by <20 mm Hg systolic; correctable with oral fluid treatment mild/moderate asymptomatic effusion, no | requires IV fluids;<br>no hospitalization<br>required<br>symptomatic<br>effusion; pain;<br>ECG changes | mean arterial pressure <60mm/ Hg or end organ damage or shock; requires hospitalization and vasopressor treatment tamponade; pericardiocentesis or surgery required |
|---|---|---|---|---|
| Hemorrhage, Blood | microscopic/occult | treatment<br>mild, no | gross blood loss; | massive blood loss; |
| Loss | landress opin social | transfusion | | > 3 units transfused |
| RESPIRATORY | | | | |
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Cough | transient- no<br>treatment | persistent cough;<br>treatment<br>responsive | Paroxysmal cough;<br>uncontrolled with<br>treatment | |
| Bronchospasm, Acute | transient; no<br>treatment;<br>70% – 80% FEV <sub>1</sub><br>of peak flow | requires treatment;<br>normalizes with<br>bronchodilator;<br>FEV <sub>1</sub> 50% – 70%<br>(of peak flow) | no normalization<br>with<br>bronchodilator;<br>FEV <sub>1</sub> 25% – 50%<br>of peak flow; or<br>retractions present | cyanosis: FEV <sub>1</sub> < 25% of peak flow or intubation necessary |
| Dyspnea | dyspnea on exertion | dyspnea with normal activity | Dyspnea at rest | Dyspnea requiring oxygen therapy |
| GASTROINTESTINA | | V 1490 V | · | |
| <u>s</u> | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Nausea | mild or transient;<br>maintains<br>reasonable intake | moderate<br>discomfort; intake<br>decreased<br>significantly; some<br>activity limited | no significant<br>intake; requires IV<br>fluids | hospitalization<br>required; |
| Vomiting | 1 episode in 24<br>hours | 2-5 episodes in 24 hours | >6 episodes in 24<br>hours or needing<br>IV fluids | physiologic<br>consequences<br>requiring<br>hospitalization or<br>requiring parenteral<br>nutrition |
| Constipation | requiring stool<br>softener or dietary<br>modification | requiring laxatives | obstipation<br>requiring manual<br>evacuation or<br>enema | obstruction or toxic<br>megacolon |

| Diarrhea | mild or transient; 3- | moderate or | >7 loose stools/day | hypotensive shock |
|---|---|---|---|---|
| | 4 loose stools/day | persistent; 5-7 | or bloody diarrhea; | or physiologic |
| | or mild diarrhea | loose stools/day or | or orthostatic | consequences |
| | last < 1 week | diarrhea lasting >1 | hypotension or | requiring |
| | COMMONIA 22 F ANDROSON NO | week | electrolyte | hospitalization |
| | | | imbalance or >2L | |
| | | | IV fluids required | |
| Oral | mild discomfort; no | some limits on | eating/talking very | unable to drink |
| Discomfort/Dysphagia | difficulty | eating/drinking | limited; unable to | fluids; requires IV |
| | swallowing | 3 | swallow solid foods | fluids |
| NEUROLOGICAL | | | | |
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Neuro-Cerebellar | slight | intention tremor, | locomotor ataxia | incapacitated |
| | incoordination | dysmetria, slurred | | |
| | dysdiadochokinesis | | | |
| Psychiatric | mild anxiety or | moderate anxiety or | | acute psychosis |
| *** | depression | depression; therapy | changes requiring | requiring |
| | | | therapy; or suicidal | hospitalization; or |
| | | normal routine | ideation; or | suicidal |
| | | | aggressive ideation | gesture/attempt or |
| | | | | hallucinations |
| Muscle Strength | subjective | mild objective | objective weakness | paralysis |
| | weakness, no | signs/symptoms no | function limited | |
| | objective | decrease in | | |
| | 77 19 19 | function | | |
| | symptoms/ signs | | 7/247 | |
| Paresthesia (burning, | mild discomfort; no | | severe discomfort; | incapacitating; or |
| tingling, etc.) | treatment required | discomfort; non- | or narcotic | not responsive to |
| | | narcotic analgesia | analgesia required | narcotic analgesia |
| | | required | with symptomatic | |
| 27 | 19.9.1 | 1 | improvement | • |
| Neuro-sensory | mild impairment in sensation | moderate | severe impairment | sensory loss |
| | | impairment (mod decreased | (decreased or loss | involves limbs and |
| | (decreased | | of sensation to | trunk; paralysis; or seizures |
| | sensation, e.g., | sensation, e.g., | knees or wrists) or | Seizures |
| | vibratory, pinprick, | | loss of sensation of at least mod degree | |
| | hot/cold in great<br>toes) in focal area | hot/cold to ankles)<br>and/or joint | in multiple | |
| | or symmetrical | position or mild | different body areas | |
| | distribution; or | impairment that is | (i.e., upper and | |
| | change in taste, | not symmetrical | lower extremities) | |
| | smell, vision and/or | not symmetrical | io wer extremities) | |
| | hearing | | | |
| MUSCULOSKELETA | | | | |
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| | Canal A | OTHER T | CING V | - I HOU I |

| Arthralgia (joint pain) Arthritis | mild pain not interfering with function mild pain with inflammation, erythema or joint swelling – but not | moderate pain,<br>analgesics and/or<br>pain interfering<br>with function but<br>not with activities<br>of daily living<br>moderate pain with<br>inflammation,<br>erythema or joint<br>swelling — | severe pain; pain and/or analgesics interfering with activities of daily living severe pain with inflammation, erythema or joint swelling —and | disabling pain permanent and/or disabling joint destruction |
|---|---|---|---|---|
| | interfering with<br>function | interfering with<br>function, but not<br>with activities of<br>daily living | interfering with<br>activities of daily<br>living | |
| Myalgia | Myalgia with no<br>limitation of<br>activity | muscle tenderness<br>(at other than<br>injection site) or<br>with moderate<br>impairment of<br>activity | severe muscle<br>tenderness with<br>marked impairment<br>of activity | frank myonecrosis |
| SKIN | | | | |
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Mucocutaneous | erythema; pruritus | diffuse, maculo<br>papular rash, dry<br>desquamation | vesiculation or<br>moist<br>desquamation or<br>ulceration | exfoliative<br>dermatitis, mucous<br>membrane<br>involvement or<br>erythema,<br>multiforme or<br>suspected Stevens-<br>Johnson or necrosis<br>requiring surgery |
| Induration | < 15mm | 15 – 30 mm | >30mm | 58 30 |
| Erythema | < 15mm | 15 – 30 mm | >30mm | |
| Edema | < 15mm | 15 - 30 mm | >30mm | 10 |
| Rash at Injection Site | < 15mm | 15 – 30 mm | >30mm | |
| Pruritus | slight itching at injection site | moderate itching at injection extremity | itching over entire<br>body | |
| SYSTEMIC | | | | T |
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Allergic Reaction | pruritus without<br>rash | localized urticaria | generalized<br>urticaria;<br>angioedema | anaphylaxis |
| SKIN | | | | |
| 18 | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Headache | mild, no treatment<br>required | transient, moderate;<br>treatment required | severe; responds to<br>initial narcotic<br>therapy | intractable; requires<br>repeated narcotic<br>therapy |

cannot work

#### Fever: oral 38.6 − 39.5 °C or 39.6 – 40.5 °C or > 40 °C or > 105 °F $37.7 - 38.5^{\circ}$ C or 101.6 – 102.9 °F 100.0 - 101.5 °F 103 − 105 °F Fatigue normal activity normal activity normal activity unable to care for reduced < 48 hours decreased 25- 50% decreased > 50% self

> 48 hours

### Appendix B: Grading of Renal Impairment

| GFR categories in CKD | | | |
|---|---|---|---|
| | Category | GFR<br>ml/min/1.73 m <sup>2</sup> | Terms |
| G1 | | ≥90 | Normal or high |
| G2 | 60 – | 89 | Mildly decreased* |
| G3a | 45 – | 59 | Mildly to moderately decreased |
| G3b | 30 – | 44 | Moderately to severely decreased |
| G4 | 15 – | 29 | Severely decreased |
| G5 | • | <15 | Kidney failure |

Abbreviations: CKD, chronic kidney disease; GFR, glomerular filtration rate.

In the absence of evidence of kidney damage, neither GFR category G1 nor G2 fulfill the criteria for CKD.

# Albuminuria categories in CKD

| Category | ACR (mg/g) | Terms |
|----------|------------|----------------------------|
| A1 | <30 | Normal to mildly increased |
| A2 | 30 - 300 | Moderately increased* |
| A3 | >300 | Severely increased** |

Abbreviations: ACR, albumin-to-creatinine ratio; CKD, chronic kidney disease.

Reference: https://www.kidney.org/professionals/explore-your-knowledge/how-to-classify-ckd

<sup>\*</sup>Relative to young adult level.

<sup>\*</sup>Relative to young adult level.

<sup>\*\*</sup>Including nephrotic syndrome (albumin excretion ACR >2220 mg/g)

### Appendix C: Child-Pugh Classification of Hepatic Impairment

The Child- Pugh classification is a means of assessing the severity of liver cirrhosis.

| Score | 1 | 2 | 3 |
|------------------------|------|---------|--------|
| bilirubin (micromol/l) | <34 | 34 - 50 | >50 |
| albumin (g/l) | >35 | 28 - 35 | <28 |
| PT (s prolonged) | <4 | 4 - 6 | >6 |
| encephalopathy | none | mild | marked |
| ascites | none | mild | marked |

If there is primary biliary cirrhosis or sclerosing cholangitis then bilirubin is classified as <68 = 1; 6 -170 = 2; >170 = 3.

The individual scores are summed and then grouped as:

- <7 = A (Mild impairment)
- 7 9 = B (Moderate impairment)
- >9 = C (Severe impairment)

A C classification forecasts a survival of less than 12 months.

From: Pugh RNH, Murray-Lyon IM, Dawson JL et al. Transection of the oesophagus for bleeding oesophageal varices. Br J Surg 1973;60:649-9.

Appendix D. SF-36<sup>TM</sup> Quality of Life Questionnaire







RAND > RAND Health > Surveys > RAND Medical Outcomes Study > 36-Item Short Form Survey (SF-36) >

# **36-Item Short Form Survey Instrument** (SF-36)

# **RAND 36-Item Health Survey 1.0 Questionnaire Items**

Choose one option for each questionnaire item.

| 1. In general, would you say your health is: |
|---|
| O 1 - Excellent |
| ○ 2 - Very good |
| ○ 3-Good |
| O 4-Fair |
| O 5 - Poor |
| 2. Compared to one year ago, how would you rate your health in general now? |
| 2. <b>Compared to one year ago</b> , how would you rate your health in general <b>now</b> ? 1 - Much better now than one year ago |
| 1 - Much better now than one year ago |
| 1 - Much better now than one year ago 2 - Somewhat better now than one year ago |
| 1 - Much better now than one year ago 2 - Somewhat better now than one year ago 3 - About the same |

The following items are about activities you might do during a typical day. Does **your health now limit you** in these activities? If so, how much?

| | Yes,<br>limited a<br>lot | Yes,<br>limited a<br>little | No, not<br>limited at<br>all |
|---|---|---|---|
| 3. <b>Vigorous activities</b> , such as running, lifting heavy objects, participating in strenuous sports | O 1 | O 2 | ○ 3 |
| 4. <b>Moderate activities</b> , such as moving a table, pushing a vacuum cleaner, bowling, or playing golf | O 1 | O 2 | O 3 |
| 5. Lifting or carrying groceries | O 1 | O 2 | ○ 3 |
| 6. Climbing <b>several</b> flights of stairs | O 1 | O 2 | ○ 3 |
| 7. Climbing <b>one</b> flight of stairs | O 1 | O 2 | ○ 3 |
| 8. Bending, kneeling, or stooping | O 1 | O 2 | ○ 3 |
| 9. Walking more than a mile | O 1 | O 2 | ○ 3 |
| 10. Walking several blocks | O 1 | O 2 | ○ 3 |
| 11. Walking one block | O 1 | O 2 | ○ 3 |
| 12. Bathing or dressing yourself | O 1 | O 2 | ○ 3 |

During the past 4 weeks, have you had any of the following problems with your work or other regular daily activities as a result of your physical health?

| <ul> <li>13. Cut down the amount of time you spent on work or other activities</li> <li>14. Accomplished less than you would like</li> <li>15. Were limited in the kind of work or other activities</li> <li>16. Had difficulty performing the work or other activities (for example, it effort)</li> </ul> | took ex | xtra | Yes 1 1 1 1 1 | No |
|---|---|---|---|---|
| During the <b>past 4 weeks</b> , have you had any of the following pro<br>other regular daily activities <b>as a result of any emotional probl</b><br>depressed or anxious)? | | | | or |
| | Yes | No | | |
| 17. Cut down the <b>amount of time</b> you spent on work or other activities | O 1 | O 2 | | |
| 18. Accomplished less than you would like | O 1 | O 2 | | |
| 19. Didn't do work or other activities as <b>carefully</b> as usual | O 1 | O 2 | | |
| 20. During the past 4 weeks, to what extent has your physical h problems interfered with your normal social activities with fam groups? 1 - Not at all 2 - Slightly 3 - Moderately 4 - Quite a bit 5 - Extremely | | | | or |

| 1 - None | |
|---|---|
| 2 - Very mild | |
| 3 - Mild | |
| 0 4 - Moderate | |
| ○ 5 - Severe | |
| 6 - Very severe | |
| 300-10-10-10-10-10-10-10-10-10-10-10-10-1 | 4 weeks, how much did pain interfere with your normal work k outside the home and housework)? |
| 300-10-10-10-10-10-10-10-10-10-10-10-10-1 | |
| (including both wor | |
| (including both wor | |
| (including both wor 1 - Not at all 2 - A little bit | |

These questions are about how you feel and how things have been with you **during the past 4 weeks**. For each question, please give the one answer that comes closest to the way you have been feeling.

How much of the time during the past 4 weeks...

| | All of<br>the<br>time | Most of the time | A good<br>bit of the<br>time | Some of the time | A little of the time | None<br>of the<br>time |
|---|---|---|---|---|---|---|
| 23. Did you feel full of pep? | $\bigcirc \ 1$ | O 2 | ○ 3 | O 4 | O 5 | O 6 |
| 24. Have you been a very nervous person? | O 1 | O 2 | O 3 | O 4 | O 5 | O 6 |
| 25. Have you felt so down in the dumps that nothing could cheer you up? | O 1 | O 2 | O 3 | O 4 | O 5 | O 6 |
| 26. Have you felt calm and peaceful? | O 1 | O 2 | ○ 3 | O 4 | O 5 | O 6 |
| 27. Did you have a lot of energy? | O 1 | O 2 | ○ 3 | O 4 | O 5 | O 6 |
| 28. Have you felt downhearted and blue? | O 1 | O 2 | ○ 3 | O 4 | O 5 | O 6 |
| 29. Did you feel worn out? | O 1 | O 2 | O 3 | O 4 | O 5 | O 6 |
| 30. Have you been a happy person? | $\bigcirc \ 1$ | O 2 | ○ 3 | O 4 | O 5 | O 6 |
| 31. Did you feel tired? | O 1 | O 2 | O 3 | O 4 | O 5 | O 6 |
| 32. During the past 4 weeks, how much of the time has your physical health or emotional problems interfered with your social activities (like visiting with friends, relatives, etc.)? 1 - All of the time 2 - Most of the time 3 - Some of the time 4 - A little of the time | | | | | | |
| 5 - None of the time | | | | | | |

Ver. 6 U.S. Only, 01 October 2019

How TRUE or FALSE is **each** of the following statements for you.

| | Definitely true | Mostly<br>true | Don't<br>know | Mostly false | Definitely<br>false |
|---|---|---|---|---|---|
| 33. I seem to get sick a little easier than other people | O 1 | O 2 | O 3 | O 4 | O 5 |
| 34. I am as healthy as anybody I know | O 1 | O 2 | ○ 3 | O 4 | O 5 |
| 35. I expect my health to get worse | O 1 | O 2 | ○ 3 | O 4 | O 5 |
| 36. My health is excellent | O 1 | O 2 | O 3 | O 4 | O 5 |

#### **ABOUT**

The RAND Corporation is a research organization that develops solutions to public policy challenges to help make communities throughout the world safer and more secure, healthier and more prosperous. RAND is nonprofit, nonpartisan, and committed to the public interest.



1776 Main Street Santa Monica, California 90401-3208

 $RAND^{\scriptsize o}$  is a registered trademark. Copyright  $\tiny \odot$  1994-2016 RAND Corporation.

Ver. 6 U.S. Only, 01 October 2019

Protocol VMT-VT-1161-CL-012

### Appendix E. EQ-5D-3L Health Status Questionnaire

### Figure 1: EQ-5D-3L (UK English sample version)

By placing a tick in one box in each group below, please indicate which statements best describe your own health state today.

| Mobility |
|----------------------------------------------------------|
| I have no problems in walking about |
| I have some problems in walking about |
| I am confined to bed |
| Self-Care |
| I have no problems with self-care |
| I have some problems washing or dressing myself |
| I am unable to wash or dress myself |
| Usual Activities (e.g. work, study, |
| housework, family or leisure activities) |
| I have no problems with performing my usual activities |
| I have some problems with performing my usual activities |
| I am unable to perform my usual activities |
| Pain/Discomfort |
| I have no pain or discomfort |
| I have moderate pain or discomfort |
| I have extreme pain or discomfort |
| Anxiety/Depression |
| I am not anxious or depressed |
| I am moderately anxious or depressed |
| I am extremely anxious or depressed |



The worst health you can imagine

Page | 8

IND 1116/5 Ver. 6 U.S. Only, 01 October 2019

# Appendix F. EQ-5D-Y Health Status Questionnaire

Figure 1: EQ-5D-Y (UK English sample version)

| Describing your health | |
|---|---|
| Under each heading, please tick the ONE box that be $TODAY$ | est describes your health |
| Mobility (walking about) | |
| I have <u>no</u> problems walking about | |
| I have <u>some</u> problems walking about | |
| I have <u>a lot</u> of problems walking about | |
| Looking after myself | |
| I have <u>no</u> problems washing or dressing myself | |
| I have <u>some</u> problems washing or dressing myself | |
| I have <u>a lot</u> of problems washing or dressing myself | |
| Doing usual activities (for example, going to school, hobbie. | <i>s,</i> |
| sports, playing, doing things with family or friends) | |
| I have <u>no</u> problems doing my usual activities | |
| I have <u>some</u> problems doing my usual activities | |
| I have <u>a lot</u> of problems doing my usual activities | |
| Having pain or discomfort | |
| I have <u>no</u> pain or discomfort | |
| I have <u>some</u> pain or discomfort | |
| I have <u>a lot</u> of pain or discomfort | |
| Feeling worried, sad or unhappy | |
| I am <u>not</u> worried, sad or unhappy | |
| I am <u>a bit</u> worried, sad or unhappy | |
| I am very worried, sad or unhappy | |

How good is your health TODAY

- We would like to know how good or bad your health is TODAY.
- This line is numbered from 0 to 100.
- 100 means the <u>best</u> health you can imagine.
   0 means the <u>worst</u> health you can imagine.
- Please mark an X on the line that shows how good or bad your health is TODAY.

The best health you can imagine



The worst health you can imagine

Appendix G. Work Productivity and Activity Impairment: Specific Health Problems Questionnaire

# Work Productivity and Activity Impairment Questionnaire: Specific Health Problem V2.0 (WPAI:SHP)

The following questions ask about the effect of vaginal yeast infections on your ability to work and perform regular activities. *Please fill in the blanks or circle a number, as indicated.* 

| reg | jular activities. Please IIII in the planks of circle a number, as indicated. |
|---|---|
| 1. | Are you currently employed (working for pay)? NO YES If NO, check "NO" and skip to question 6. |
| Th | e next questions are about the <b>past seven days</b> , not including today. |
| 2. | During the past seven days, how many hours did you miss from work because of problems associated with a vaginal yeast infection? Include hours you missed on sick days, times you went in late, left early, etc., because of a vaginal yeast infection. Do not include time you missed to participate in this study. HOURS |
| | 1100113 |
| 3. | During the past seven days, how many hours did you miss from work because of any other reason, such as vacation, holidays, time off to participate in this study? |
| | HOURS |
| 4. | During the past seven days, how many hours did you actually work? |
| | HOURS (If "0", skip to question 6.) |

Ver. 6 U.S. Only, 01 October 2019

5. During the past seven days, how much did a vaginal yeast infection affect your productivity while you were working?

Think about days you were limited in the amount or kind of work you could do, days you accomplished less than you would like, or days you could not do your work as carefully as usual. If a vaginal yeast infection affected your work only a little, choose a low number. Choose a high number if a vaginal yeast infection affected your work a great deal.

Consider only how much the vaginal yeast infection affected productivity while you were working.

| Vaginal yeast | | | | | | | | | | | | Vaginal yeast |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| infection had no | | | | | | | | | | | | infection |
| effect on my | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | completely |
| work | | | | | | | | | | | | prevented me |
| | | | | | | | | | | | | from working |

### **CIRCLE A NUMBER**

6. During the past seven days, how much did a vaginal yeast infection affect your ability to do your regular daily activities, other than work at a job?

By regular activities, we mean the usual activities you do, such as work around the house, shopping, childcare, exercising, studying, etc. Think about times you were limited in the amount or kind of activities you could do and times you accomplished less than you would like. If a vaginal yeast infection affected your activities only a little, choose a low number. Choose a high number if a vaginal yeast infection affected your activities a great deal.

Consider only how much the vaginal yeast infection affected your ability to do your regular daily activities, other than work at a job.

| Vaginal yeast<br>infection had | | | | | | | | | | | | Vaginal yeast infection |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| no effect on my daily activities | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | completely<br>prevented me<br>from doing my<br>daily activities |
| | CIRCLE A NUMBER | | | | | | | | _ | | | |

#### WPAI:SHP V2.0 (US English)

Reilly MC, Zbrozek AS, Dukes E: The validity and reproducibility of a work productivity and activity impairment measure. PharmacoEconomics 1993; 4(5):353-365.

Appendix H. Patient Health Questionnaire – 9

# PATIENT HEALTH QUESTIONNAIRE-9

| by any of the following p<br>(Use "✓" to indicate your a | ow often have you been bothered roblems? answer) | Not at a | Several<br>II days | More<br>than half<br>the days | Nearly<br>every<br>day |
|---|---|---|---|---|---|
| 1. Little interest or pleasure | e in doing things | 0 | 1 | 2 | 3 |
| 2. Feeling down, depresse | d, or hopeless | 0 | 1 | 2 | 3 |
| 3. Trouble falling or staying | g asleep, or sleeping too much | 0 | 1 | 2 | 3 |
| 4. Feeling tired or having li | ttle energy | 0 | 1 | 2 | 3 |
| 5. Poor appetite or overea | ting | 0 | 1 | 2 | 3 |
| 6. Feeling bad about yours have let yourself or you | self — or that you are a failure or<br>r family down | 0 | 1 | 2 | 3 |
| 7. Trouble concentrating o newspaper or watching | n things, such as reading the television | 0 | 1 | 2 | 3 |
| noticed? Or the opposit | slowly that other people could have<br>te — being so fidgety or restless<br>ring around a lot more than usual | 0 | 1 | 2 | 3 |
| 9. Thoughts that you would yourself in some way | d be better off dead or of hurting | 0 | 1 | 2 | 3 |
| | FOR OFFICE COD | ing <u>0</u> | + | + | |
| | | | | =Total Score | : |
| | oblems, how <u>difficult</u> have these<br>at home, or get along with other | | made it fo | r you to do | your |
| Not difficult<br>at all | Somewhat | Very<br>difficult | | Extreme<br>difficu | |

Developed by Drs. Robert L. Spitzer, Janet B.W. Williams, Kurt Kroenke and colleagues, with an educational grant from Pfizer Inc. No permission required to reproduce, translate, display or distribute.

Appendix I. RVVC History Questionnaire (Version 01) – US Only

### **RVVC History Questionnaire (Version 01)**

| 1. | How many vaginal yeast infections have you had in the last 12 months? |
|---|---|
| 2. | Of the vaginal yeast infections you have had in the <b>last 12 months</b> , how many did you receive a diagnosis from a health care provider (physician, nurse, physician's assistant, etc.)? |
| 3. | Of the vaginal yeast infections you have had in the <b>last 12 months</b> that were diagnosed by a healthcare professional, for how many did you receive a pelvic exam? |
| 4. | Of the vaginal yeast infections you have had in the <b>last 12 months</b> for which you received a pelvic exam, how many did a healthcare professional take a vaginal swab and run a test to confirm the diagnosis (either during your appointment or with a follow-up call)? |
| 5. | How many years in a row have you experienced at least 3 vaginal yeast infections per year? a) Only the last year b) More than 1 year but not more than 2 years c) More than 2 years but not more than 5 years d) More than 5 years |
| 6. | Please estimate the total number of vaginal yeast infections you have had in your <b>lifetime</b> : |
| 7. | |
| 8. | Prior to enrolling in this study, what treatment or treatments do you typically use to treat a vaginal yeast infection? <b>Select up to 3</b> a) One to three pills of fluconazole/Diflucan by prescription b) One to three pills of fluconazole/Diflucan over-the-counter (i.e., without a |
| | prescription – only available in some countries) |
| | <ul> <li>c) Fluconazole/Diflucan taken every week, by prescription</li> <li>d) Fluconazole/Diflucan taken every week, over-the-counter (i.e., without a prescription – only available in some countries)</li> </ul> |
| | e) Prescription topical cream, ointment, or suppository f) Over the counter topical gream, circument, or suppository |
| | <ul> <li>f) Over-the-counter topical cream, ointment, or suppository</li> <li>g) Homeopathic Remedies (such as probiotics, tea tree oil, coconut oil, garlic, yogurt, etc.)</li> </ul> |
| | h) Dietary or lifestyle change |
| | i) I don't know, it depends on what my doctor says |
| | j) I don't know, it depends on what my pharmacist says |
| | k) Other (please specify): |

| 9. | When you've used the treatment or treatments you previously specified, for how many <b>days</b> do your vaginal yeast infection symptoms typically last (from beginning of symptoms until symptoms are gone)? |
|---|---|
| 10. | Please estimate how much it personally cost you to diagnose, treat and prevent <b>your</b> |
| | last vaginal yeast infection (the one prior to this one), in each of the following |
| | categories of costs. Please enter "0" for any categories in which you had no out-of- |
| | pocket costs (do not leave blanks) |
| | a) Over-the counter medications: |
| | b) Prescription payments: |
| | c) Physician visit payments: |
| | d) Payments for diagnostic tests: |
| | e) Other (e.g. probiotics, homeopathic remedies, pain/itch relievers, etc.): |
| | e) other (e.g. producties, nomeopatine remedies, paintien remevers, etc.). |
| 11. | Please estimate how much it has personally cost you in total to diagnose and treat all your recurrent vaginal yeast infections over the last 12 months, in each of the following categories of costs. Please enter "0" for any categories in which you had no out-of-pocket costs (do not leave blanks). a) Over-the counter medications: b) Prescription payments: c) Physician visit payments: d) Payments for diagnostic tests: e) Other (e.g. probiotics, homeopathic remedies, pain/itch relievers, etc.): |
| 12. | How many days of work would you estimate you have missed over the past 12 |
| | months, specifically due to having or wanting to prevent a vaginal yeast |
| | infection? |

Appendix J. Extension Study – U.S. Only

IND 111675 Ver. 6 U.S. Only, 01 October 2019

# APPENDIX J. OBSERVATIONAL EXTENSION STUDY: VMT-VT-1161-CL-012

### 1.0 BACKGROUND INFORMATION AND RATIONALE

Several properties of VT-1161 suggest that it has the potential to be a best-in-class oral agent for the treatment of recurrent vulvovaginal candidiasis (RVVC), to effectively inhibit growth of causative fungal pathogens at achievable plasma levels. Its pharmacokinetic profile and extended half-life should limit recurrence of VVC. The purpose of this twelve-month Observational Extension Study is to gain additional insight into the ability of VT-1161 to prevent VVC beyond Week 48 in RVVC subjects yet to experience a recurring episode on completion of study VMT-VT-1161-CL-012. This is an observational study; there will be no active treatment. The Sponsor may choose, prior to the end of study, to extend this Extension Study for an additional period for subjects willing to continue.

### 2.0 STUDY OBJECTIVES

### 2.1 Primary Objective

The primary objective is to evaluate changes in culture-verified acute VVC episode recurrence rates through Week 96 in subjects free of a recurring VVC episode upon completion of their Week 48 visit in study VMT-VT-1161-CL-012 and who have qualified for the Extension, in an observational study.

### 3.0 STUDY DESIGN

Approximately 100 subjects in the United States who completed their Week 48 (EOS) visit and did not have a RVVC episode during the Maintenance Phase (post-randomization through Week 48 for study VMT-VT-1161-CL-012) will be offered the opportunity to enroll in an observational Extension Study. The Extension Study will monitor for recurring episodes of VVC for an additional 48 Weeks, for a total study participation of 96 weeks.

Subjects must sign the Extension Study informed consent form (ICF), or assent, at the Week 48 (EOS) visit prior to any Extension Study procedures. Subjects will be contacted approximately every 6 weeks to monitor for recurrence of VVC. Subjects experiencing a suspected recurrent episode of VVC will return to the investigational site for evaluation at an unscheduled visit.

IND 111675 Ver. 6 U.S. Only, 01 October 2019

### 3.1 Extension Duration of the Study

The observational Extension Study duration is expected to be approximately 23 months from consenting of the first subject until last visit of the last subject. The maximum Extension Study duration of individual subject participation will be 48 weeks.

### 3.2 Number of Study Sites/Total enrollment

Approximately 70 investigative sites in the United States will participate in the Extension Study. The study will seek to enroll approximately 100 subjects. Assuming a 20% discontinuation rate for the duration of the study, approximately 80 subjects are expected to complete the study.

### 4.0 STUDY POPULATION

The Investigator or other study site personnel must record in the source documents (e.g., the site's chart) and case report form (CRF) that the ICF document was signed and dated and all entry criteria were met prior to conducting any Extension Study procedures. The following criteria for enrollment must be followed explicitly; any violations of these criteria must be reported in accordance with Institutional Review Board (IRB) Policies and Procedures.

### 4.1 Inclusion Criteria

- 1. Subjects must have participated in the VMT-VT-1161-CL-012 study and completed the Week 48 visit.
- 2. Subjects must be willing and able to provide written informed consent (or assent, if applicable) and provide authorization for use of protected health information (HIPAA).
- 3. Subjects must be willing and able to comply with protocol requirements, instructions, and protocol-stated restrictions and be likely to complete the study as planned.

### 4.2 Exclusion Criteria

- 1. Subjects who, in the opinion of the Investigator, were non-compliant in the main study and / or may become non-compliant with study schedules or procedures.
- 2. Subjects who had a positive KOH and clinical signs and symptoms score of ≥3 during the Maintenance Phase (post-randomization through Week 48) of study VMT-VT-1161-CL-012.
- 3. Subjects must not plan to participate in another clinical trial.
- 4. Subjects must not be taking any prohibited medications.

IND 111675 Ver. 6 U.S. Only, 01 October 2019

### 5.0 PROHIBITED MEDICATIONS

The following prescription and over-the-counter drug products are prohibited during the study and will be considered a protocol deviation:

- 1. Topical or oral antifungal drugs, except when prescribed by the Investigator to treat a subject with a recurrent VVC episode.
- 2. Topical products applied to the vulva or vagina (e.g. antibiotic, antiviral, antitrichomonal, corticosteroids, or anti-inflammatory agents).
- 3. Oral antibacterial, antiviral, or antitrichomonal agents for the treatment of bacterial vaginosis, trichomonas, or other concomitant (urogenital) infection unless prescribed by the Investigator.
- 4. Vaginal douches, boric acid, or benzalkonium chloride disinfectant during the study.

### 6.0 STUDY ASSESSMENTS AND PROCEDURES

### 6.1 Assessments

The study subjects should be contacted within the timeframes noted in (Table 1) the Schedule of Assessments and Procedures.

IND 111675 Ver. 6 U.S. Only, 01 October 2019

Table 1: Schedule of Assessments and Procedures – Extension Study

| able 1: Schedule of Assessments and Procedures – Extension Study | | | |
|---|---|---|---|
| Activities | Week 48<br>(± 14 days) | Subject Contact<br>Every 6 Weeks <sup>b</sup><br>(± 14 days) | Unscheduled<br>Visit <sup>e</sup> |
| Sign Informed Consent or Assent Form | X | | |
| Inclusion/Exclusion Criteria | X | | |
| <b>Excluded Concomitant Medications</b> | | X | X |
| Verify if Treatment of a Suspected<br>VVC Episode Since Previous Contact | | X | X |
| Review and Record Subject Reported<br>Pregnancy Status <sup>a</sup> | | X | X |
| Vaginal Exam with Clinical Signs and<br>Symptoms of Vulvovaginitis | | | X |
| Local KOH Wet Mount | | | X |
| Central Vaginal Fungal Culture | | | X |
| PK Samples | | | X |

Abbreviations noted above - KOH: potassium hydroxide prep; PK: pharmacokinetic

- a. Subjects who became pregnant during the main study protocol or become pregnant during the Extension Study will be followed until term. Pregnancy outcome must be documented in the subject's medical record.
- b. Subject contacts should be made every 6 weeks  $\pm$  2 weeks, at Weeks 54, 60, 66, 72, 78, 84, 90 and 96. Week 96 will be the final subject contact.
- c. All procedures listed are to be completed only for unscheduled visits where a recurrent VVC episode is suspected.
#### 6.1.1 Week 48 – Clinic Visit

Once the subject has signed the IRB / Independent Ethic Committee (IEC) approved informed consent (or assent, if applicable) document, the following procedures will be performed:

- Review Inclusion and Exclusion criteria to assess the subject's eligibility.
- Remind the subject that they will be contacted approximately every 6 weeks beginning at Week 54.
- Remind the subject not to self treat or seek care from another healthcare professional for any suspected RVVC episode but instead return to the study site for evaluation (and treatment, if needed) anytime during the study.

### 6.1.2 Every 6 Weeks (±14 Days) – Subject Contact

The subjects will be contacted by investigative site personnel, every 6 weeks ( $\pm 14$  Days) at approximately Weeks 54, 60, 66, 72, 78, 84, 90, and 96 for the following evaluations:

- Review and record any excluded medications taken since the previous visit.
- Remind the subject not to self treat or seek care from another healthcare professional for any suspected RVVC episode but instead return to the study site for evaluation (and treatment, if needed) during the Extension Study.
- If applicable, review and record if the subject has become pregnant or pregnancy status if previously recorded.
- Remind subject that they will be contacted every 6 weeks and that the site will keep contacting the subject until they are available to discuss their status.

### 6.1.3 Week 96 (±14 Days) – Subject Contact

The subjects will be contacted at Week 96 for their final contact to close their participation in the study. The items below should be discussed:

- Review and record all excluded medications taken since the previous visit.
- If applicable, review and record if the subject has become pregnant or pregnancy status if previously recorded.
- Complete the "Subject Contact" and "Termination Extension" eCRF pages.

IND 1111675 Ver. 6 U.S. Only, 01 October 2019

• Thank the subject for their participation and let them know this is the last study contact.

### 6.1.4 Unscheduled Visit - Clinic Visit

Unscheduled visits are to be used if the subject suspects an RVVC episode. The following evaluations are to be performed:

- Record all excluded medications taken since the previous visit.
- Perform a vaginal exam including an assessment of clinical signs and symptoms of vulvovaginitis, as outlined in .
- Perform KOH wet mount test, performed locally ().
- Obtain vaginal swab for culture to send to the central mycology laboratory (7.1.3.1).
- Obtain PK plasma specimen.
- Remind the subject not to self treat or seek care from another healthcare professional for any suspected RVVC episode but instead return to the study site for evaluation (and treatment, if needed) during the Extension Study.
- If applicable, review and record if the subject has become pregnant or pregnancy status if previously recorded.
- Remind subject that they will be contacted every 6 weeks and that the site will keep contacting the subject until they are available to discuss their status.

### **6.2 Study Procedures**

### 6.2.1 Pregnancies

Subjects may become pregnant during the Extension Study. For any subject that became pregnant during the main study protocol or becomes pregnant during the Extension Study, the outcome of their pregnancy (birth or termination) must be documented in the subject's medical record.

### **6.2.2 KOH Wet Mount and Fungal Cultures**

A vaginal fungal culture will be obtained at the unscheduled clinic visit and sent to the central mycology laboratory for fungal identification and susceptibility testing according to approved Clinical Laboratory Standards Institute methods. Details as to the collection of samples, shipping, testing methods and analysis will be delineated in a laboratory manual. Mycology samples may

Ver. 6 U.S. Only, 01 October 2019

be retained for future analysis for a period of up to 15 years, after which time the samples will be destroyed.

A local KOH wet mount test will be performed at the unscheduled clinic visit where a recurrent VVC episode is suspected. (If the Investigator site used the Gram stain test instead of the KOH test in the main study, they may continue to use it in the Extension Study).

Subjects should not be menstruating at time of the study visits to ensure proper sample collection of the vaginal fluid.

#### **Vulvovaginal Exam and Clinical Assessment** 6.2.3

A vulvovaginal exam and clinical assessment of signs and symptoms will be evaluated at the unscheduled clinic visit. Each of the following vulvovaginal signs and symptoms will be scored and the individual scores combined for a maximum score of 18, using the following scale:

- a. Signs: erythema, edema, and excoriation
- b. Symptoms: itching, burning, and irritation

Scoring Scale: Each score should be objectively defined on a scale of 0 to 3 as follows:

0 = none (complete absence of any signs or symptoms)

1 = mild (slight)

2 = moderate (definitely present)

3 = severe (marked, intense)

### 7.0 PHARMACOKINETIC ASSESSMENTS

Assays to measure VT-1161 concentrations in plasma PK samples will be performed using a validated bioanalytical assay at a laboratory designated by Mycovia Pharmaceuticals.

The PK data may be used in a cross-population PK analysis that may be presented in a separate report. Pharmacokinetic samples may be retained for future analysis of the metabolite profile for a period of up to 15 years, after which time the samples will be destroyed.

### 8.0 STUDY TERMINATION AND SUBJECT DISCONTINUATION

### 8.1 Extension Study Screen Failures

Subjects who sign and date the Extension Study consent (or assent, if applicable) but fail to meet the inclusion and exclusion criteria are defined as entry failures. Site personnel need to maintain a screening log to document all subjects who sign a consent (or assent). A copy of the log should be retained in the Investigator's study files. Additionally, site personnel must complete the eCRF "Termination Extension" page.

## **8.2** Early Termination Conditions

If the Investigator suspects the subject is experiencing a recurrent episode, at any time during the Extension Study, the subject should be examined. The suspected RVVC episode will be documented on an 'unscheduled visit' eCRF and considered the subject's End of Extension Study (EOES) visit **ONLY if the signs and symptoms score is ≥3 and the KOH is positive**. The Investigator is to perform all unscheduled visit procedures, including submission of vaginal mycology swab to central lab for culture analysis. Upon diagnosis of a recurrent episode, the Investigator should:

- a. offer the subject standard of care treatment options.
- b. Complete the "unscheduled visit" and "Termination Extension" eCRF pages.

An unconfirmed RVVC episode is one where the subject self-treats or sees a (non-Investigator Site) health care professional and does not have documentation of the visit including the required study signs and symptoms and a positive KOH.

# 8.3 Subject Withdrawal and Premature Discontinuation from the Extension Study

Appropriate actions should be taken to ensure subjects complete each study visit within the protocol specified window and do not become lost to follow-up.

A subject may withdraw from the study at any time at her own request or may be withdrawn at any time at the discretion of the Investigator for safety, behavioral, or administrative reasons. If a subject withdraws her consent from the study participation, she may request destruction of any laboratory samples taken, and the Investigator must document this in the site study records and communicate this request to Mycovia Pharmaceuticals.

Reasons for subject discontinuation of the Extension Study at the investigative site may include, but are not limited to, the following:

- Safety reasons that are study related or serious adverse events (SAEs) that may affect the subjects' ability to continue with the required study procedures and assessments. The subject must be followed clinically until the event is resolved or deemed stable.
- Subject wishes to withdraw consent for any reason. The reason for withdrawing consent should be captured if the subject is willing to share.
- Subject non-compliance or unwillingness to comply with the procedures required by the protocol.
- Investigator discretion.
- Due to low enrollment/ continuation in the study, the Sponsor decides to stop the study.

### 8.4 Study Termination

Reasons for discontinuation of the Extension Study at the investigative site may include, but are not limited to, the following:

- Subject enrollment is unsatisfactory.
- Investigator request to withdraw from participation.
- Sponsor decision.
- Serious and/or persistent non-compliance by the Investigator with the protocol, the clinical research agreement, the Form (FDA) 1572 or applicable regulatory guidelines in conducting the study.
- Decision by the IRB/IEC to terminate or suspend approval for the investigation or the Investigator.
- Investigator fraud (altered data, omitted data, or manufactured data).

### 8.5 Subject and Study Extension Completion

A completed subject is one who has completed all Extension Study visits: Weeks 48 through Week 96 or was determined to have a positive KOH with signs and symptoms score of  $\geq$ 3 at an unscheduled clinic visit.

### 9.0 STATISTICAL ANALYSIS

### 9.1 Statistical Methods and Planned Analysis

Descriptive statistical methods will be used to summarize the data from this Extension Study. There will be no hypothesis testing. Unless otherwise stated, the term "descriptive statistics" refers to number of subjects, mean, median, standard deviation, minimum, and maximum for continuous data, confidence intervals and frequencies and percentages for categorical data.

### 9.2 Demographic and Baseline Characteristic Analyses

Subject disposition, demographics, and baseline characteristics will be summarized by treatment group.

### 9.3 Efficacy Analysis

Clinical and mycological assessments will be conducted as outlined in Table 1 of the Extension Study.

Subjects will be required to return to the study site if they suspect a recurring episode of VVC during the Extension Study. The primary objective is to measure the proportion of subjects with one or more culture-verified acute VVC episodes during the Maintenance Phase (post-randomization through Week 96) in the ITT population. An acute VVC episode during the Extension (considered a recurrent episode) is defined as a positive culture for Candida species and a clinical signs and symptoms score of ≥3.

## 9.4 Pharmacokinetic Analysis

PK samples will be collected at the unscheduled clinic visit to determine VT-1161 concentrations. Data will be presented by visit with descriptive statistics.

## 10.0 CLINICAL STUDY ADMINISTRATION/STUDY GOVERNANCE CONSIDERATIONS

## 10.1 Ethical Conduct of Study

The study will be conducted in accordance with ICH Good Clinical Practice (GCP), all applicable subject privacy requirements, the guiding principles of the current version of the Declaration of Helsinki, and applicable country-specific regulatory requirements. This includes, but is not limited to, the following:

- IRB/IEC review and favorable opinion/approval of the study protocol and amendments, as applicable, informed consent and assent (for those ages 12 to 17) documents, and investigational brochure.
- Signed informed consent form or assent (for those ages 12 to 17) to be obtained for each subject before participation in the study (and for amendments as applicable).
- Investigator reporting requirements (e.g., continuing reviews, reporting of AEs/SAEs/protocol deviations to the IRB/IEC).

If any documents are translated, an official certificate of translation must be maintained.

### **10.2 Informed Consent**

Written informed consent must be signed and dated by the subject prior to their initiation of study-related procedures or tests. The original signed informed consent for each participating subject shall be filed with records kept by the Investigator(s). A copy of the informed consent document must be provided to the subject. If applicable, it will be provided in a certified translation of the local language.

## 10.3 Quality Control (Study Monitoring)

In accordance with applicable regulations, including GCP, the representative(s) or the designated clinical study monitor of Mycovia Pharmaceuticals will contact the site staff prior to the start of the study to review the protocol, study requirements, and their responsibilities to satisfy regulatory, ethical, and Mycovia Pharmaceuticals' requirements. When reviewing the data collection procedures, the discussion will also include identification, agreement, and documentation of data items that will serve as the source document.

Mycovia Pharmaceuticals representative(s) or the designated clinical study monitor will review the study data remotely at regular intervals throughout the study and may perform on-site visits to verify the following:

- Data are Attributable, Legible, Contemporaneous, Original, Accurate and Complete (ALCOAC).
- Safety and rights of subjects are being protected.
- Study is conducted in accordance with the currently approved protocol and any other study agreements, GCP/ICH E6(R2), and all applicable regulatory requirements.

The Investigator and the head of the medical institution (where applicable) agrees to allow the clinical study monitor, direct access to all relevant documents.

Relevant documents or source documents are defined as the results of original observations and activities of a clinical investigation. Source documents may include, but are not limited to, study progress notes, e-mail correspondences, computer printouts, laboratory data, and drug accountability records.

### **10.4 Quality Assurance**

To ensure compliance with GCP/ICH E6(R2) and all applicable regulatory requirements, Mycovia Pharmaceuticals may conduct a quality assurance assessment and/or audit of the site records, and the regulatory agencies may conduct a regulatory inspection at any time during or after the completion of the study. In the event of an assessment, audit or inspection, the Investigator (and institution) must agree to grant the advisor(s), auditor(s), and inspector(s) direct access to all relevant documents and to allocate their time and the time of their staff to discuss the conduct of the study, any findings/relevant issues, and to implement any corrective and/or preventative actions to address any findings/issues identified.

### 10.5 Compliance with Standards of Medical Research/ Deviations

This protocol will be conducted in accordance with the applicable ICH E6(R2) guidelines and GCP. Any instance of non-compliance with the protocol will result in a documented deviation. If a change is deemed necessary to protect the safety, rights or welfare of a subject, Mycovia Pharmaceuticals and IRB/IEC should be notified as soon as possible and preferably prior to introducing the deviation. Major deviations are defined as, but not limited to, the following:

- Subjects who did not meet entry criteria.
- Subjects who developed withdrawal criteria during the study but were not withdrawn.

## 10.6 Data Management

Electronic case report forms (eCRFs) will be used to capture study results and data. The study coordinator or other authorized site study personnel will transcribe data from source documents into the eCRFs. The Extension eCRFs may be reviewed and source verified by the clinical study monitor to ensure data in the eCRF are correct and complete. The Medical Monitor or clinical study monitor may request redacted copies of source documents for medical review. Once the Extension Study is complete, the Investigator must sign and date all required pages, verifying the accuracy of all data contained within the eCRF.

Training will be provided for the Electronic Data Capture (EDC) system. All personnel using the EDC system must have the appropriate education, training, and experience, or any combination thereof. The Investigator will be provided with SOPs (contained in the Study Procedures Manual or a vendor-specific SOP) on the use of the EDC system. Documentation for employee education, training, and previous experience that pertains to the EDC system must be present in the Investigator files.

If electronic data systems other than those provided and maintained by Mycovia Pharmaceuticals are used for documentation and data capture, the Investigator must ensure that the systems are validated and ensure regular data back-up.

The eCRF will be signed by the Principal Investigator listed on the Food and Drug Administration (FDA) 1572 form. It is the responsibility of the Principal Investigator to ensure the eCRFs are completed and submitted to Mycovia Pharmaceuticals (or designee) in an accurate and timely manner. The processing of eCRFs will include an audit trail (to include changes made, reason for change, date of change, and person making change). At the completion of the Extension study, eCRFs (including queries and audit trails) will be retained by the Mycovia Pharmaceuticals and copies will be sent to the Investigator to maintain as the Investigator copy.

Management of clinical data will be performed in accordance with applicable Mycovia Pharmaceuticals standards and data cleaning procedures to ensure the integrity of the data (e.g., removing errors and inconsistencies in the data). Concomitant medications will be coded using WHO-DD.

## 10.7 Study and Site Closure

Upon completion or premature discontinuation of the study, the representative (or designated clinical study monitor) of Mycovia Pharmaceuticals will conduct site closure activities with the Investigator or site staff, as appropriate, in accordance with applicable regulations including GCP. Mycovia Pharmaceuticals reserves the right to suspend or prematurely discontinue this study at any time for reasons including, but not limited to, safety or ethical issues or severe non-compliance. For multicenter studies, this can occur at 1 or more or at all sites. If the Sponsor determines such action is needed, Mycovia Pharmaceuticals will discuss the reasons for taking such action with the Investigator or head of the medical institution (where applicable). When feasible, Mycovia Pharmaceuticals will provide advance notification to the Investigator or head of the medical institution (where applicable) of the impending action. If the study is suspended or prematurely discontinued for safety reasons, Mycovia Pharmaceuticals will promptly inform all Investigators, heads of medical institutions (where applicable), and/or institutions conducting the study.

Mycovia Pharmaceuticals will also promptly inform the relevant regulatory authorities of the suspension or premature discontinuation of the study and the reason(s) for the action. If required by applicable regulations, the Investigator must inform the IRB/IEC promptly and provide the reason(s) for the suspension or premature discontinuation.

Mycovia Pharmaceuticals requires the following data and materials before a study can be considered complete or terminated:

- 1. Clinical data and all test results from Extension Study Week 48 through Week 96.
- 2. Electronic CRFs properly completed by appropriate study personnel and signed and dated by the Investigator.
- 3. All outstanding queries and site issues resolved.
- 4. Copies of protocol amendments and IRB approval/notification if appropriate.
- 5. A close-out summary for the site, prepared by the Principal Investigator (an IRB summary letter is acceptable).

### 10.8 Record Retention

Following closure of the study, the Investigator must maintain all site study records (except for those required by local regulations to be maintained elsewhere), in a safe and secure location. The records must be maintained to allow easy and timely retrieval when needed (e.g., for a Mycovia Pharmaceuticals audit or regulatory inspection) and must be available for review in conjunction with the assessment of the facility, supporting systems, and relevant site staff. When permitted by local laws/regulations or institutional policy, some or all records can be maintained in a format other than hard copy (e.g., microfiche, scanned, electronic); however, caution needs to be exercised before such action is taken. The Investigator must ensure that all reproductions are legible and are a true and accurate copy of the original and meet accessibility and retrieval standards, including regenerating a hard copy, if required. Furthermore, the Investigator must ensure there is an acceptable back-up of these reproductions and that an acceptable quality control process exists for making these reproductions.

Investigators are required to retain essential documents pertaining to the conduct of this study for at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product, per ICH guidelines. The minimum retention time will meet the strictest standard applicable to that site for the study, as dictated by any institutional requirements, local laws or regulations, or

Protocol VMT-VT-1161-CL-012

Mycovia Pharmaceuticals' standards/procedures. The Investigator must notify Mycovia Pharmaceuticals of any changes to the archival arrangements, including, but not limited to, archival at an off-site facility or transfer of ownership of the records in the event the Investigator is no longer associated with the site.

### 10.9 Disclosure of Data

The Investigator agrees by his/her participation that the results of this study may be used for submission to national and/or international registration and supervising authorities. If required, these authorities will be provided with the names of Investigators, their addresses, qualifications, and extent of involvement. It is understood that the Investigator is required to provide Mycovia Pharmaceuticals with all study data, complete reports, and access to all study records.

Data generated by this study must be available for inspection by the United States FDA and other regulatory authorities, by Mycovia Pharmaceuticals, and the IRB/IEC as appropriate. At a subject's request, medical information may be given to his or her personal physician or other appropriate medical personnel responsible for his or her welfare. Subject medical information obtained during this study is confidential and disclosure to third parties other than those noted above is prohibited.

### 10.10 Financial Disclosure

The United States FDA Financial Disclosure by Clinical Investigators (21 Code of Federal Regulations 54) regulations require Sponsors to obtain certain financial information from Investigators participating in covered clinical studies; each Principal Investigator and Sub-Investigator is required to provide the required financial information and to promptly update Mycovia Pharmaceuticals with any relevant changes to their financial information throughout the course of the clinical study and for up to 1 year after its completion. This rule applies to all Investigators and Sub-Investigators participating in covered clinical studies to be submitted to the FDA in support of an application for market approval.

## **10.11 Publication Policy**

The publication policy is outlined in the Clinical Trial Agreement.

## 10.12 Confidentiality

Confidentiality is outlined in the Clinical Trial Agreement.

### 10.12.1 Data

All information about the nature of the proposed investigation provided by Mycovia Pharmaceuticals or the designated clinical study monitor to the Investigator (except for information required by law or regulations to be disclosed to the IRB/IEC, the subject, or the appropriate regulatory authority) must be kept in confidence by the Investigator.

### 10.12.2 Subject Anonymity

The anonymity of participating subjects must be maintained. Subjects will be identified by an assigned subject number on CRFs and other documents retrieved from the site or sent to the designated clinical study monitor, Sponsor, regulatory agencies, or central laboratories/reviewers. Documents that identify the subject (e.g., the signed informed consent document, subject identification record) must be maintained in strict confidence by the Investigator, except to the extent necessary to allow auditing by the appropriate regulatory authority, the clinical study monitor, or Mycovia Pharmaceuticals representatives.

## Appendix K. Protocol Amendment Summary of Changes

| Protocol Version 6 (Amendment 5): 01 October 2019<br>Country-Specific Amendment: U.S. Only | | | |
|---|---|---|---|
| Section | Change | Reason | Impact on<br>Human<br>Subject<br>(risk/benefit) |
| Version 5/<br>Amendment<br>4 | The Version 5/ Amendment 4 Extension Study Protocol was not implemented and should not be released or filed at the Investigator Site. | Redesign of the<br>Extension Study<br>Protocol on 01<br>October 2019. | Benefit |

| Protocol Version 5 (Amendment 4): 18 June 2019 | | | |
|---|---|---|---|
| Country-Specific Amendment: U.S. Only | | | |
| Section | Change | Reason | Impact on<br>Human<br>Subject<br>(risk/benefit) |
| Synopsis Page 15 & 16, Table 1 | Added "PK Samples should be collected before the weekly dosing of study drug (placebo/VT-1161)." | To clarify timing of PK sample | Benefit |
| 8.1<br>Table 1 | Added "PK Samples should be collected before the weekly dosing of study drug (placebo/VT-1161)." | To clarify timing of PK sample | Benefit |
| 8.1.2 #9 | Added "PK Samples should be collected before the weekly dosing of study drug (placebo/VT-1161)." | To clarify timing of PK sample | Benefit |
| 10.1 | Added "The initial PK sample must be drawn prior to the first dose of study drug (placebo/VT-1161)." | To clarify timing of PK sample | Benefit |
| Appendix J | Added Appendix J: Study Extension. | Implementing an Extension Study to the main study for U.S. only, to track long-term efficacy and safety | Benefit |

| Protocol Version 4 (Amendment 3): 25 February 2019 | | | |
|---|---|---|---|
| Section | Change | Reason | Impact on<br>Human<br>Subject<br>(risk/benefit) |
| Page 3 | Changed Medical Responsible information from J. Gordon Still to Claude Hughes | Individual serving as Medical Responsible for the study changed. | Not applicable |
| Synopsis<br>4.1 | Clarified Maintenance Phase dosing for VT-1161 or placebo, '7 daily doses followed by 11 weekly doses.' | Expanded description to prevent confusion of dosing regimen. | Benefit |
| Synopsis<br>Table 1<br>4.1<br>8.1.1<br>12.7<br>Append I | Added 'for all regions and questions regarding their RVVC history (US only)'. Added 'for all regions. At Screening, subjects will also be required to answer questions regarding their RVVC history (US only).' Added 'for all regions and RVVC History Questionnaire (US Only)'. Added 'all regions participating in' and 'For US only, questions regarding RVVC history will be administered at Screening using the RVVC History Questionnaire (see Appendix I) to collect information on the disease, diagnosis, and treatment profile for the subjects enrolled in the study.' Added Appendix I RVVC History Questionnaire. | To collect information on subjects' historical experience and impact of RVVC in the United States. | Not<br>applicable |
| Synopsis<br>Incl #1<br>4.4.1<br>5.1<br>7.1.1 | Added ', Romania, Ukraine,'. | Per Romania Ethics<br>Committee and<br>Ukraine Ministry of<br>Health, subjects < 18<br>years of age cannot be<br>enrolled in Romania<br>or Ukraine. | Benefit |
| Synopsis<br>Incl #1<br>5.1 | Added 'post-menarchal'. | To clarify patient population eligible for enrollment (post-menarchal was previously assumed). | Benefit |
| Synopsis<br>Incl #2<br>5.1 | Added ', or other approved diagnostic tests.' | To allow establishment of RVVC history based on locally-approved testing as outlined in the study design (missing from inclusion criterion language). | Benefit |
| Synopsis<br>Incl #5<br>5.1 | Added 'timeline per' and minor grammatical changes. | Improved clarity on timelines for Pap test requirement. | Benefit |

| Synopsis<br>Incl #9<br>5.1 | Changed 'study entry' to 'Screening' and added 'at Screening'. | Clarified<br>requirements for non-<br>childbearing potential<br>as they relate to time<br>from Screening | Benefit |
|---|---|---|---|
| Synopsis<br>Incl #10<br>5.1 | For OPTION 3 contraceptive methods, added 'In addition to OPTIONS 1 and 2, subjects of childbearing potential (includes ages 12-17) may also use 1 of the following methods of contraception after completing the Induction Phase on Study Day 1 through Week 48.' Added footnotes for: 'Sexual abstinence is defined as refraining from heterosexual intercourse during the entire study period and where this is the usual life style of the subject. Periodic abstinence (calendar, symptothermal, postovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not considered to be acceptable methods of contraception;' 'Subjects who started taking a hormonal contraceptive less than 3 months prior to the first dose of fluconazole must agree to use a double-barrier method (i.e. diaphragm plus spermicide or condom) through 3 months after starting the hormonal contraceptive;' and 'Because of the teratogenic risk associated with repeat dosing of fluconazole, OPTION 3 contraceptive methods cannot be used during Screening and the Induction Phase of the study (from Screening until Baseline (Day 1) of the study).' | Provide clarification for definition of abstinence and restrict contraceptive methods during repeat dosing of fluconazole to only highly effective methods. | Benefit |
| Synopsis 7.4.1 | Added '; refer to Section 8.1.12 on treatment options if fluconazole is ineffective.)' | Cross-reference to<br>allowed treatment<br>plan should a subject<br>fail to respond to<br>fluconazole treatment<br>for an acute VVC<br>episode. | Benefit |
| Synopsis 7.4.1 | Added '(urogenital)'. | Clarity on assumed type of other concomitant infections. | Benefit |
| Synopsis<br>Excl #5<br>5.2<br>7.4.1 | Added 'collunarium/nasal' to list of concomitant steroids permitted and to Exclusion Criterion #5. | Clarity on collunarium/nasal steroid use was missing. | Benefit |
| Synopsis<br>Excl #5<br>5.2 | Added 'nor use of topical vulvar or vaginal steroids during the study or within 7 days prior to Screening'. | Reduce potential confounding factors for efficacy assessments. | Benefit |
| Synopsis<br>Excl #6<br>5.2<br>7.4.1 | Added subjects must not use any 'vaginal douches or benzalkonium chloride disinfectant during the study.' Added 'or vaginal douches' to Exclusion Criterion #6. | Reduce potential confounding factors for efficacy assessments. | Benefit |
| Synopsis<br>Excl #14<br>5.2 | Removed 'performed by the investigative site'. | HbA1c testing will be performed by central laboratory. | Benefit |

| Table 1 | Separated central serum pregnancy test from local urine pregnancy test | Improved clarity for which testing is used at each visit | Benefit |
|---|---|---|---|
| Table 1 8.1.1 | Added '±2 days' to Screening (Day -14) Visit | Allow flexibility for scheduling Screening visit with respect to Day 1 without impact to assessments | Benefit |
| Table 1 9.1.5.3 | Added cholesterol and triglycerides testing. | Implement testing requested by PMDA under Study VMT-VT-1161-CL-012 across Phase 3 studies to evaluate across all subject populations. | Benefit |
| 1.1.1.3 | Remove '%' | Corrected erroneous unit given to pH value. | Not applicable |
| 1.2 | Replaced 'tablets' with 'capsules'. | VT-1161 is a capsule formulation for this study. | Not applicable |
| 5 | Added '(or assent for those 12-17)'. | Clarified informed consent document includes assent for subjects 12-17. | Not applicable |
| 8.1.1<br>9.1.5.6<br>9.1.5.7<br>9.1.5.8 | Clarified <i>Bacterial vaginosis</i> testing will be done locally and <i>Chlamydia trachomatis</i> and <i>Neisseria gonorrhoeae</i> testing will be done by central laboratory. Added Section 9.1.5.8 Bacterial Vaginosis, moved 'Testing for <i>Bacterial vaginosis</i> will be done locally.' from Section 9.1.5.7. | Prevent confusion on which testing is being performed locally and centrally. | Benefit |
| 8.1.1<br>9.1.5.3<br>9.1.5.4<br>9.1.5.5 | Added 'Central'. | Clarified central laboratory results are not required prior to start of fluconazole treatment. | Benefit |
| 8.1.1 | Added 'one time'. | Clarified subjects can<br>be eligible for re-<br>screening one time. | Benefit |
| 12.5 | Changed '14' to '21'. | MedDRA <sup>®</sup> dictionary<br>used for coding AEs<br>will be version 21 this<br>study | Not<br>applicable |
| 13.5 | Changed 'Subjects who were <80% or >120% compliant of all doses of IMP' to 'Subjects who were <80% IMP compliant in the Induction Phase or <50% IMP compliant in the Maintenance Phase.' | Modified protocol<br>deviation criterion for<br>consistency with<br>statistical analysis<br>population<br>definitions. | Benefit |
| Multiple,<br>see<br>below | Changes made for Protocol Version 3 (Amendment 2 – Region/Country Specific Amendment) and Protocol Version 2 (Amendment 1 – Country Specific Amendment) | Implementing changes made during EU Voluntary Harmonisation | Benefit |

Ver. 6 U.S. Only, 01 October 2019

| Procedure review as |
|---------------------|
| were beneficial to |
| subject safety and |
| data quality from a |
| global perspective. |

## Protocol Version 3 (Amendment 2): 08 October 2018 Region/Country Specific Amendment: EU/Belgium, Czech Republic, Hungary, Romania, and Ukraine

| Section | Change | Reason | Impact on<br>Human<br>Subject<br>(risk/benefit) |
|---|---|---|---|
| Synopsis | Added, '. finalized before 50% of subjects are enrolled' | Provide updated information on when SAP will be final for consistency with Section 12 in Protocol Amendment 1 | Not applicable |
| Synopsis, 7.4.1 | Added, 'carbamazepine' to concomitant/prohibited medications list of drugs with narrow therapeutic index that are metabolized by and sensitive to induction of CYP3A4' | Clarify complete list of<br>narrow therapeutic index<br>drugs metabolized by or<br>sensitive to CYP3A4 for<br>consistency with change<br>made to Exclusion<br>Criteria #7 in Protocol<br>Amendment 1 | Benefit |
| 11.2 | Added, 'Subjects who prematurely discontinue study medication, but remain in the study, may be treated according to the standard local practice.' | Additional instructions for discontinued subjects. | Benefit |
| 12.1 | Removed, 'discontinuation,' and added, 'the primary efficacy outcome measure in this study was the proportion of subjects with one or more culture-verified acute VVC episodes during the Maintenance Phase through Week 48 of the study in the ITT population (all randomized subjects). Culture-verified acute VVC was defined as a positive fungal culture for Candida species associated with a total signs and symptoms score of ≥ 3. The proportion of subjects with one or more culture-verified acute VVC episodes through Week 48 was lower in the VT-1161 dosing regimens (0-7%) compared with the placebo group (52.2%). This difference was statistically significant in all VT-1161 treatment groups compared with placebo (p<0.0001). | Provide additional explanation for how sample size was determined. | Not applicable |
| 12.4 | Added, 'The primary method of analysis is a Chisquare test for active treatment versus placebo based on the ITT population. | Provide additional information on the analysis and how missing data for the handled for the primary endpoint. | Not applicable |

Protocol VMT-VT-1161-CL-012

number and percentage of subjects with one or more culture-verified acute VVC episodes with signs and symptoms of ≥3 post randomization through Week 48 will be summarized across treatment groups including a 95% exact confidence interval and odds ratio. The percentages will also be plotted by treatment group' and 'Every effort will be made to obtain required data at each scheduled evaluation from all subjects who have been randomized, including those who discontinue the study prior to the EOS Week 48 visit. For scheduled visits where the investigator's assessment of clinical signs and symptoms or the culture result is missing, missing values will be imputed using the method of multiple imputation. For subjects who discontinue the study early and have missing assessments for all visits after discontinuation, the missing values for the expected scheduled visits will be imputed using the method of multiple imputation. The missing values will be imputed using the following auxiliary information: region, treatment, baseline BMI, baseline age, ethnicity, and visit. The procedure PROC MI in SAS will be used to generate 10 possible imputed datasets. Using these multiple imputation datasets, determination of meeting the primary endpoint of a culture-verified acute VVC episode during the Maintenance Phase will be derived. Subjects with a culture-verified acute VVC episode at any point from post randomization through Week 48 (including unscheduled visits) will be counted as having an episode when calculating the primary endpoint. The multiple datasets containing the primary endpoint will be analyzed using a Chi-square test and the results will be combined using PROC MIANALYZE to obtain an inferential result. Sensitivity analyses will be performed for the primary endpoint to assess the impact of missing/censored data on the results using different time to event and censoring calculations. Further details on the steps of these analyses are presented in the VMT VT-1161-CL-012 SAP.'

## Protocol Version 2 (Amendment 1): 07 September 2018 Country Specific Amendment: Belgium, Czech Republic, Hungary, and Romania

| Country | Country Specific Amendment: Belgium, Czech Republic, Hungary, and Romania | | |
|---|---|---|---|
| Section | Change | Reason | Impact on<br>Human<br>Subject<br>(risk/benefit) |
| Page 3 | Added 'Regulatory authorities, if required by national law, must give a favorable opinion/approval of the study protocol and amendments, informed consent and assent (for those ages 12 to 17) documents, and investigational brochure.' | Additional information regarding potential regulatory authorities' requirements. | Benefit |
| Synopsis,<br>4.4.1<br>Incl #1,<br>5.1, 7.1.1 | Added, 'In Hungary and Czech Republic only, subjects must be generally healthy, non-pregnant females 18 years of age and older as of Screening.' | Per country SOC, Hungary<br>and Czech Republic will not<br>be enrolling subjects < 18<br>years of age. | Benefit |
| Synopsis,<br>Excl #7,<br>5.2 | Added, 'carbamazepine' to list of drugs with narrow therapeutic index that are metabolized by and sensitive to induction of CYP3A4' | Clarify complete list of narrow therapeutic index drugs metabolized by or sensitive to CYP3A4 | Benefit |
| Synopsis,<br>Table 1,<br>5.2 Excl #<br>14,<br>9.1.5.3 | Removed 'only on known diabetics or subjects suspected to have diabetes' and added 'for all subjects'. | HbA1c testing will be performed on all subjects at Screening. | Benefit |
| Table 1,<br>8.1.2 –<br>8.1.12,<br>9.1.5.1 | Added local urine pregnancy testing for all visits for WOCBP. | Monitor more frequently for pregnancies throughout the study for all WOCBP. | Benefit |
| 7.3 | Removed 'Medical Monitor and' from unblinding procedures if Grade 4 AE considered related to IMP. | Clarified guidelines for consistency with unblinding guidelines outlined in Section 7.8. | Benefit |
| 7.8 | Removed 'The Investigator must contact the Medical Monitor or appropriate Mycovia Pharmaceuticals study personnel to discuss options regarding unblinding the subject's treatment assignment.' Removed "Mycovia Pharmaceuticals' Medical Monitor" and changed to 'The Investigator" for who may unblind a subject's treatment assignment only in the case of an emergency (i.e., a Grade 4 AE) OR in the event of a serious medical condition when knowledge of the study treatment is essential for the appropriate clinical management or welfare of the subject as judged by the Investigator. Added 'The Investigator must contact the Medical Monitor or appropriate Mycovia Pharmaceuticals study personnel to communicate the reasons for unblinding the subject's treatment assignment | Guidelines to allow the Investigator the ability to unblind a subject's treatment assignment in an emergency to facilitate fulfillment of Investigator responsibilities according to ICH GCP 4.3.1 and 4.7. | Benefit |

| | immediately after the unblinding occurred (ICH GCP 4.7).' | | |
|---|---|---|---|
| 8.1.12 | Added 'If the subject fails to respond to fluconazole treatment, the Investigator may employ treatment options corresponding to the site's standard of care treatment for treating the infection upon consultation with the Medical Monitor.' | Instructions for treatment of recurrent acute VVC episodes for subjects that fail to respond to fluconazole treatment during the Maintenance Phase. | Benefit |
| 11.2 | Added 'A subject may be withdrawn due to lack of tolerability or safety concerns, including study drug-related AEs or development of clinically-significant study drug-related laboratory abnormalities. If a subject is withdrawn from treatment, the subject must be followed clinically until the event is resolved or deemed stable. A subject must be discontinued from the study drug if ALT or/and AST is > 5 × the upper limit of normal (ULN) or ALT or/and AST is > 3 × ULN and serum total bilirubin is > 2.0 ULN.' | Additional discontinuation criteria. | Benefit |
| 11.3 | Added, 'Study completion is defined as when the last subject has completed their last study visit.' | To define study completion. | Not applicable |
| 12 | Updated language to 'A formal SAP will be finalized prior to 50% of enrollment. The SAP will provide a detailed description of the proposed data analysis methods and procedures. The SAP was drafted and submitted to regulatory bodies prior to the start of the study. The SAP contains all the details for the analysis of the primary and secondary endpoints as well as the sensitivity analyses for these endpoints. The additions to the SAP since that initial submission include additional sensitivity analyses, The handling of missing data is explained in detail in the SAP. The SAP also includes the descriptions of the sensitivity analyses that will be performed for each endpoint in order to assess the impact of the handling of the missing data on the results.' Originally read 'A formal SAP will be finalized prior to enrollment of the first subject.' | To provide additional information on plans for primary and secondary analyses and handling of missing data. | Not applicable |
| 12.1 | Added 'The placebo discontinuation rate was based on data generated in the Phase 2b RVVC study. When powering this study, it was determined that a separation of at least 35% between the treatment groups would be a clinically meaningful separation. Thus, the sample size was powered to pick up at least a 35% separation between the treatment groups.' | Provide additional explanation for how sample size was determined. | Not applicable |